| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized | Version: 4.0-Master, 07 Sep |
| Controlled Study to Evaluate the Safety and | 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in | <b>Page</b> : 1 of 167 |
| unicondylar knee arthroplasty (UKA) Procedure | rage: 1 of 107 |

Sponsor Name and Address: Smith & Nephew, Inc., 1450 E. Brooks Road,

Memphis, TN 38116, United States

Investigational Product(s) REAL INTELLIGENCE™ CORI™ (referred as

"CORI" throughout this document)

Single Identification Number CORI.2019.06

of Clinical Investigation

Protocol Author(s): Manvendra Saxena, Clinical Study Manager

Babajide Olayinka, Senior Biostatistician

Summary of Revision Version 2.0 04 Sep 2020

History Version 2.1 14 Jan 2021

Version 3.0-Master 03 Mar 2021

Version 4.0-Master 07 Sep 2021

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep<br>2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in | <b>Page</b> : 2 of 167 |
| unicondylar knee arthroplasty (UKA) Procedure | Page. 2 01 107 |

## 1 SIGNATURES

### 1.1 Principal Investigator Signature Page

This page will be returned to Smith & Nephew Inc. and a copy retained at the investigational site.

□ I have read the attached protocol entitled "A Prospective, Multi-center,
Randomized Controlled Study to Evaluate the Safety and Effectiveness of REAL
INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure", version
4.0-Master, dated 07Sep2022, and agree to abide by all provisions set forth herein.
I agree to comply with the Investigator's Obligations stipulated in Section 22.6
Principal Investigator Obligations according to ISO 14155:2020 and all applicable
local legislation and regulations.
I agree to ensure that the confidential information contained in this document will
not be used for any purpose other than the conduct of the described clinical
investigation without the prior written consent of Smith & Nephew Inc.

Name, Address, Professional Position Signature and Date / DocuSign Stamp

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep<br>2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | |

#### 1.2 COORDINATING INVESTIGATOR APPROVAL

□ I have read the attached protocol entitled "A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure", version 4.0-Master, dated 07Sep2022, and agree to abide by all provisions set forth therein.

Name, Address, Professional Position Signature and Date / DocuSign Stamp

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized | Version: 4.0-Master, 07 Sep |
| Controlled Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in | |
| unicondylar knee arthroplasty (UKA) Procedure | Page. 4 01 107 |

# 1.3 SPONSOR APPROVAL

| Name and Title | Signature and Date / DocuSign Stamp |
|---|---|
| Rachael Winter, Senior Director, Global Clinical Operations | DocuSigned by: Rachael Winter Signer Name: Rachael Winter Signing Reason: I approve this document Signing Time: 25-Nov-2022 08:41:03 GMT A32F12A80F1B4490986E80ACCB7471CB |
| Julian Yang, Director,<br>China Clinical Affairs | DocuSigned by: Julian Yang Signer Name: Julian Yang Signing Reason: I approve this document Signing Time: 22-Nov-2022 01:39:38 GMT 7874D1D26E584792AFFC91EBB7CEF6D0 |
| Julie Lankiewicz,<br>Clinical Strategy Director<br>Robotics | DocuSigned by: Julie Lankiewicz Signer Name: Julie Lankiewicz Signing Reason: I approve this document Signing Time: 21-Nov-2022 14:14:22 GMT 59CD0029AA274067A40E4605966E81DA |
| Michael Robinson, Independent Statistician signing on behalf of Director Biostatistics & Data Management | DocuSigned by: Michael Petins Signer Name: Michael Robinson Signing Reason: I approve this document Signing Time: 22-Nov-2022 14:40:41 GMT 0E27C33EB43441FB820C99CBC38E7E89 |

# **Clinical Protocol**

A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure

Study Number: CORI.2019.06

**Version**: 4.0-Master, 07 Sep 2022

**Page**: 5 of 167



| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep<br>2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 6 of 167 |

## 2 SYNOPSIS

| Title of Study: | A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) procedure |
|---|---|
| Study Design: | Prospective, multi-center, randomized controlled study |
| Study Type: | Post-market study in Australia, New Zealand, South Korea & China (Hong Kong) Pre-market study in China Mainland |
| Study Product: | REAL INTELLIGENCE™ CORI™ (CORI) is a computer-assisted orthopedic surgical navigation and burring system. CORI is designed to aid surgeons in planning and executing a procedure involving bone preparation for unicondylar knee arthroplasty (UKA) and total knee arthroplasty (TKA) procedures. CORI is comprised of a console control unit, optical tracking camera, primary and secondary input displays (tablet and optional display monitor), and foot pedal. The CORI software consists of a patient and user management module, a surgical planner, and an intra-operative cutting module. |
| Comparison Groups | Conventional approach with conventional manual instrumentation will be used as the comparison group. |
| Study Purpose: | This is a prospective randomized controlled study to demonstrate the safety and effectiveness of CORI and to register CORI in China mainland. |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in | <b>Page</b> : 7 of 167 |
| unicondylar knee arthroplasty (UKA) Procedure | Page. 7 01 107 |

| Primary Objective: Secondary Objective(s): | To evaluate the use of CORI in unicondylar knee arthroplasty (UKA) procedures in achieving post-operative leg alignment as compared to procedures using conventional manual instruments. To generate safety and performance evidence supporting the use of CORI procedures. To assess the safety and performance of CORI up to 12 |
|---|---|
| | months after surgery as compared to procedures using conventional manual instruments. |
| Other Objective(s): | To collect CORI system time and cutting time of the robotic drill from the CORI Case Report. |
| Sample Size: | <ul> <li>140 in total:</li> <li>70 CORI procedure for UKA</li> <li>70 Conventional procedures for UKA</li> <li>1. The statistical justification for CORI UKA is based on data collected from the NAVIO™ Navigation System, the former generation of CORI.</li> <li>2. N=70 subjects per arm, based on post-operative alignment (±3 degrees) with expected 92.1% NAVIO™ vs. 73.4% from a historical control.</li> </ul> |
| Number of Study Sites: | Up to 8 sites |
| Targeted Global<br>Regions: | Australia, China Mainland, China (Hong Kong), South Korea, and New Zealand |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in | |
| unicondylar knee arthroplasty (UKA) Procedure | Page. 8 01 107 |

| Inclusion Criteria: | <ol> <li>Subject is a suitable candidate for a UKA procedure<br/>using CORI and a compatible Smith &amp; Nephew (S+N)<br/>Knee implant system.</li> </ol> |
|---|---|
| | <ul> <li>2. Subject requires a cemented UKA as a primary indication that meets any of the following conditions:</li> <li>a) Non-inflammatory degenerative joint disease, including osteoarthritis</li> <li>b) Avascular necrosis</li> </ul> |
| | <ul><li>c) Requires correction of functional deformity</li><li>d) Requires treatment of fractures that were unmanageable using other techniques</li></ul> |
| | <ol> <li>Subject is of legal age to consent and considered<br/>skeletally mature (≥ 18 years of age at the time of<br/>surgery).</li> </ol> |
| | <ul> <li>4. Subject agrees to consent to and to follow the study visit schedule (as defined in the study protocol and informed consent form), by signing the Ethics Committee (EC) or Institutional Review Board (IRB) approved informed consent form.</li> <li>5. Subject plans to be available through one (1) year postoperative follow-up.</li> <li>6. Applicable routine radiographic assessment is possible.</li> </ul> |
| Exclusion Criteria: | <ol> <li>Subject receives a UKA on the index joint as a revision for a previously failed surgery, or need for complex implants, or any other implant than a standard UKA (e.g., stems, augments, or custom-made devices).</li> <li>Subject has been diagnosed with post-traumatic arthritis</li> </ol> |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 9 of 167 |

- 3. Subject receives simultaneous bilateral UKA OR a unilateral UKA with contralateral TKA.
- 4. Subject has one or more of the following arthroplasties that are not fully healed and well-functioning, as determined by the investigator:
  - -Contralateral primary TKA or UKA, however, the subject can only have one knee enrolled in this study.
- 5. Subject does not understand the language used in the Informed Consent Form.
- Subject does not meet the indication or is contraindicated for UKA according to specific S+N knee system's Instructions for Use (IFU).
- 7. Subject has active infection or sepsis (treated or untreated).
- 8. Subject is morbidly obese with a body mass index (BMI) greater than 40.
- Subject is pregnant or breast feeding at the time of surgery.
- 10. Subject, in the opinion of the Investigator, has advanced osteoarthritis or joint disease at the time of surgery and was better suited for an alternate procedure.
- 11. Subject currently enrolled in another orthopedic clinical trial study.
- 12. Subject has a condition(s) that may interfere with the UKA survival or outcome (i.e., Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease, or an active, local infection).

| Clinical Protocol | Study Number: CORI.2019.06 |
|-----------------------------------------------|-----------------------------|
| A Prospective, Multi-center, Randomized | Version: 4.0-Master, 07 Sep |
| Controlled Study to Evaluate the Safety and | 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in | <b>Page</b> : 10 of 167 |
| unicondylar knee arthroplasty (UKA) Procedure | Fage: 10 01 107 |

| | <ul> <li>13. Subject in the opinion of the Investigator has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, intellectual disability, drug or alcohol abuse.</li> <li>14. Subject, in the opinion of the Investigator, has a neuromuscular disorder that prohibited control of the index joint.</li> <li>15. Subject is a prisoner or meets the definition of a Vulnerable Subject per ISO 14155:2020 Section 3.55.</li> </ul> |
|---|---|
| Study Duration: | <ul><li>Estimated timeline:</li><li>Study period: 36 months</li></ul> |
| | Start enrolment: April 2022 |
| | Last subject first visit: March 2024 |
| | Last subject last visit: April 2025 |
| Primary endpoint: | Post-operative leg alignment via radiographic assessment |
| | (the proportion of subjects achieving planned post-operative |
| | leg alignment 6 weeks after surgery, defined as ± 3° from |
| | target) |
| Secondary | Component Alignment |
| endpoint(s): | Radiographic assessment (Presence of radiolucent |
| | lines, osteolysis & implant migration) |
| | <ul><li>2011 Knee Society Score (2011 KSS)</li><li>Oxford Knee Score (OKS)</li></ul> |
| | Forgotten Joint Score (FJS-12) |
| | <ul> <li>Five-level EuroQol five-dimensional (EQ-5D-5L) Visual</li> </ul> |
| | Analogue Scale (VAS) and index scores |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 11 of 167 |

| Other exploratory | Each enrolled subject's CORI Case Report will be collected to |
|---|---|
| endpoint(s): | document the system time and cutting time of the robotic drill. |
| Safety Data | <ul> <li>All adverse events (AEs) and complications occurring from the time of subject enrollment until study termination or study completion including intraoperative adverse events and complications.</li> <li>Device related re-intervention</li> <li>Device Deficiencies</li> <li>Knee implant revision rate</li> <li>All AEs will be categorized in terms of seriousness and relatedness to the study device or to the surgical procedure (Adverse Events, Serious Adverse Events, Adverse Device Effects, Serious Adverse Device effects). All Serious Adverse Device Effects will be further categorized as Anticipated or Unanticipated. The definitions for each of these categories are based on ISO 14155:202020 and applicable local laws and regulations.</li> </ul> |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 12 of 167 |

## **STUDY SCHEDULE**

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 13 of 167 |

| | Pre- | Operative | 6 weeks | 6 months | 12 months |
|---|---|---|---|---|---|
| Schedule of events | Operative<br>Data<br>-90 to 0<br>days | Data & Discharge Day 1 (+ up to 9 days) | | 185 ± 14<br>days | 365 ± 30<br>days |
| Informed<br>Consent | х | | | | |
| Demographics/<br>Medical History | x | | | | |
| Inclusion/Exclusi on | x | | | | |
| Preoperative Examinations (e.g. ECG, Blood Routine Examination, Biochemical Examination, Coagulation Examination) | x | | | | |
| Pregnancy Test <sup>2</sup> | х | | | | |
| Concomitant<br>Medication | x | | | | |
| Concomitant<br>Medication<br>Update | | х | x | x | x |
| Operative Data<br>Collection | | х | | | |
| CORI Case<br>Report (System<br>time & cutting<br>time) | | x | | | |
| Discharge Data<br>Collection | | х | | | |
| Leg alignment<br>Long leg X-ray<br>AP <sup>3</sup> | x | (x) <sup>4</sup> | х | | (x) <sup>5</sup> |

## 

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep<br>2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | |

| Standard Lateral<br>X-ray | | (x) <sup>4</sup> | x | | х |
|---|---|---|---|---|---|
| Standard A/P X-ray | | | | | x |
| KSS | х | | х | х | x |
| OKS | x | | х | х | × |
| FJS-12 | | | х | х | × |
| EQ-5D-5L | x | | x | x | × |
| Safety<br>Assessment | | x | x | x | x |
| End of Study/Exit | | | (x) <sup>6</sup> | (x) <sup>6</sup> | х |

- Only applicable at site in China
- <sup>2</sup> Only Applicable at site in China
- Pre-operative long leg X-rays (A/P) collected 6-months prior to the date of surgery is admissible.
- Post-operative standing weight bearing long leg X-rays (A/P) and standard lateral X-rays may be taken at discharge.
- Only if standing weight bearing long leg A/P X-ray is taken as a standard of care at 12 months.
- <sup>6</sup> Exit form to be completed at the point of withdrawal if the study is not completed

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 15 of 167 |

## **3 CONTENTS**

## **Table of Contents**

| 1 S | ıgnatures | 2 |
|---|---|---|
| 1.1 | Principal Investigator Signature Page | 2 |
| 1.2 | Coordinating Investigator Approval | 3 |
| 1.3 | Sponsor Approval | 4 |
| 2 S | ynopsis | 6 |
| To ass | sess the safety and performance of CORI up to 12 months after surgery | 7 |
| 3 C | ontents | 15 |
| 3.1 | List of Tables | 17 |
| 3.2 | List of Figures | 18 |
| 3.3 | List of Abbreviations And definitions | 19 |
| 4 I | ntroduction | 22 |
| 4.1 | Background | 22 |
| 4.2 | Literature Summary | 25 |
| 4.3 | Study Purpose | 32 |
| 4.4 | Safety Considerations | 32 |
| <b>5</b> O | bjective(s) | 36 |
| 5.1 | Primary Objective | 36 |
| 5.2 | Secondary Objective(s) | 36 |
| 5.3 | Other Objective(s) | 36 |
| 5.4 | Claims | 36 |
| 6 I | nvestigational Product(s) and Comparator | 37 |
| 6.1 | Identification | 37 |
| 6.2 | Product Use | 41 |
| 6.3 | Packaging and Labelling | 42 |
| 6.4 | Product Accountability Procedures | 43 |
| 6.5 | Surgical Technique | 44 |
| 6.6 | Medical Procedure | 44 |
| 7 S | ubject Enrollment and Withdrawal | 45 |
| 7.1 | Subject Population | 45 |

#### 

# Clinical Protocol A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure Study Number: CORI.2019.06 Version: 4.0-Master, 07 Sep 2022 

| 7.2 | Inclusion Criteria | 46 |
|-------|-----------------------------------------------------|----------------|
| 7.3 | Exclusion Criteria | 46 |
| 7.4 | Screening | 49 |
| 7.5 | Informed Consent | 49 |
| 7.6 | Enrolment | 50 |
| 7.7 | Lost to Follow-Up | 50 |
| 7.8 | Withdrawal | 5 <sup>^</sup> |
| 8 St | tudy Design | 53 |
| 8.1 | Study Design | 5 |
| 8.2 | Allocation and Blinding | 55 |
| 8.3 | Data Management | 56 |
| 8.4 | Study Endpoints | 5 |
| 8.5 | Methods Used to Minimize Bias and Maximize Validity | 58 |
| 9 St | tudy Procedures | 59 |
| 9.1 | Visits and Examinations | 59 |
| 9.2 | Study Methods and Measurements | 69 |
| 9.3 | Health Economics/Quality of Life | 75 |
| 10 St | tatistical Design | 77 |
| 10.1 | General | 77 |
| 10.2 | Analysis Populations | 7 |
| 10.3 | Baseline Data | 78 |
| 10.4 | Effectiveness Analysis | 78 |
| 10.5 | Safety Analyses | 84 |
| 10.6 | Interim Analyses | 84 |
| 11 Sa | ample Size Justification | 85 |
| 12 A | dverse Events and Device Deficiencies | 86 |
| 12.1 | Definitions | 86 |
| 12.2 | AE Coding Dictionary | 92 |
| 12.3 | Reporting Procedures | 93 |
| 12.4 | Unblinding of Investigational Product | 96 |
| 12.5 | Follow-up of Subjects with Adverse Events | 96 |
| 13 Tr | vestigator Obligations | 97 |

# Clinical ProtocolStudy Number: CORI.2019.06A Prospective, Multi-center, Randomized<br/>Controlled Study to Evaluate the Safety and<br/>Effectiveness of REAL INTELLIGENCE™ CORI™ in<br/>unicondylar knee arthroplasty (UKA) ProcedureVersion: 4.0-Master, 07 Sep<br/>2022Page: 17 of 167

| 14 | S | oonsor and Monitor Responsibilities | 97 |
|---|---|---|---|
| 14 | - | Contract Research Organization | |
| 14 | .2 | Site Qualification Visit | 98 |
| 14 | .3 | Site Initiation Visit | 98 |
| 14 | .4 | Interim Monitoring Visit | 98 |
| 14 | .5 | Sponsor Audits and Regulatory Inspection | 98 |
| 14 | .6 | Close-out Visit | 99 |
| 15 | Pi | otocol Deviations | 99 |
| 16 | Pr | otocol Amendments | 99 |
| 17 | Co | onfidentiality of the Study | 100 |
| 18 | | atements of Compliance | |
| 19 | | nd of Study | |
| 20 | | ıblication Policy | |
| <b>20</b> | | Publication of Study Data | |
| 20 | | Data Sharing | |
| 21 | | eferences | |
| 22 | | pendices | |
| <b>22</b> | _ | Protocol Amendment | |
| 22 | | Sponsor Details | |
| 22 | | Instructions For Use & User Manuals | |
| 22 | _ | Equipment and Special Instructions | |
| 22 | 5 | Health Economic Outcome Measures/ Quality of Life Measures | |
| 22 | .6 | Principal Investigator Obligations | |
| 3.1 | Lis | ST OF TABLES | |
| Table | e 4.2 | 2-4-1 Demographic Information for the Navigation Knee Surgical Systems | 27 |
| Table | e 8.1 | - 8-1 Overview of Study Groups | 53 |
| Table | e 9.1 | 1-9-1 Study Procedures by Visit | 60 |
| Table | e 9.2 | 2.4-9-2 2011 Knee Society Score | 72 |
| Table | e 12 | 1-12-1 Categories of Adverse Event | 86 |
| Table | e 12 | 1.4-12-2 Potential Anticipated Serious Adverse Device Effects (ASADE) | 89 |

#### 

# Clinical Protocol A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure Study Number: CORI.2019.06 Version: 4.0-Master, 07 Sep 2022 

| Table 22.4-22-1 CORI Components | 143 |
|--------------------------------------------------------------|-----|
| Table 22.4-22-2 CORI Cart | 143 |
| Table 22.4-22-3 CORI Monitor | 143 |
| Table 22.4-22-4 CORI Tray and Instrumentation | 143 |
| Table 22.4-22-5 CORI Shipping Inserts | 144 |
| Table 22.4-22-6 CORI Lids | 144 |
| Table 22.4-22-7 CORI Instrument Reduction Modules - Kits | 145 |
| Table 22.4-22-8 CORI JOURNEY II UKA Inserts | 145 |
| Table 22.4-22-9 CORI JOURNEY II Instrument Reduction Inserts | 145 |
| Table 22.4-22-10 Total Knee Instruments | 146 |
| Table 22.4-22-11 CORI Disposables | 147 |
| Table 22.4-22-12 CORI Country Bundles | 147 |
| Table 22.4-22-13 CORI Welcome Box | 148 |
| Table 22.4-22-14 CORI Product Documents / Other | 148 |
| Table 22.4-22-15 CORI Power Cords | 149 |
| 3.2 <b>LIST OF FIGURES</b> | |
| Figure 6.1-6-1 CORI | 38 |
| Figure 6.1-6-2 CORI Reusable Instruments | 40 |
| Figure 6.1-6-3 Extramedullary rod | 4 |
| Figure 6.1-6-4 Intramedullary rod | 4 |
| Figure 8.1-8-1 Study Recruitment Timeline | 54 |
| Figure 8.1-8-2 Study Flowchart | 55 |
| Figure 9.2-9-1 Leg alignment | 69 |
| Figure 9.2.2-9-2 A/P View | 7′ |
| Figure 9.2.2-9-3 Lateral View | 72 |
| Figure 12.3-12-1 Evaluation and Reporting of AE | 95 |
| Figure 12.3-12-2 Evaluation and Reporting of DD | 96 |
| Figure 6.1-6-2 CORI Reusable Instruments | 114 |
| Figure 6.1-6-2 CORI Reusable Instruments | 114 |
| Figure 8 1-8-1 Study Recruitment Timeline | 140 |

#### 

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 19 of 167 |

## 3.3 LIST OF ABBREVIATIONS AND DEFINITIONS

| Abbreviation | Definition |
|--------------|-------------------------------------------|
| ADE | Adverse Device Effect(s) |
| AE | Adverse Event(s) |
| ACL | Anterior Cruciate Ligament |
| ANCOVA | Analysis of Covariance |
| A/P | Antero-posterior |
| ASADE | Anticipated Serious Adverse Device Effect |
| AVN | Avascular Necrosis |
| BMI | Body Mass Index |
| CAS | Computer-assisted navigation systems |
| CE | Conformité Européene |
| CI | Confidence Interval |
| CORI | REAL INTELLIGENCE™ CORI™ |
| eCRF | Electronic Case Report Form(s) |
| CRO | Contract Research Organization |
| СТА | Clinical Trial Agreement |
| CV | Curriculum Vitae |
| DD | Device Deficiency(ies) |
| DMP | Data Management Plan |
| ECG | Electrocardiogram |
| EDC | Electronic Data Capture |
| EQ-5D-5L | Five-level EuroQol five-dimensional |
| FAS | Full Analysis Set Population |
| FDA | Food and Drug Administration |
| FJS-12 | Forgotten Joint Score |
| FU | Follow-Up |

## 

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 20 of 167 |

| Abbreviation | Definition |
|--------------|---------------------------------------------------|
| GCP | Good Clinical Practice |
| GDPR | EU Global Data Protection Regulation |
| HIPAA | Health Information Portability Accountability Act |
| НКА | Hip-Knee-Ankle |
| HRQoL | Health Related Quality of Life |
| IB | Investigator's Brochure |
| ICH | International Conference on Harmonization |
| IEC | Independent Ethics Committee |
| IFU | Instructions for Use |
| IP | Investigational Product |
| IRB | Institutional Review Board |
| ISF | Investigator Site File |
| ITT | Intention to Treat population |
| 2011 KSS | Knee Society Score, 2011 |
| LCL | Lateral Collateral Ligament |
| LL | Lower Limit |
| LOCF | Last Observation Carried Forward |
| MCL | Medial Collateral Ligament |
| NA or N/A | Not Applicable |
| N (or n) | Total Sample Size (or subgroup sample size) |
| NAVIO | NAVIO™ Navigation System |
| NMPA | National Medical Products Administration |
| OA | Osteoarthritis |
| OKS | Oxford Knee Score |
| OR | Operating room |
| PCL | Posterior Cruciate Ligament |
| PI | Principal Investigator |
| PICF | Patient Informed Consent Form |

## 

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep<br>2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | |

| Abbreviation | Definition |
|---|---|
| PMA | Pre-Market Authorization |
| PP | Per-protocol Population |
| PSI | Patient specific instrumentation |
| RA | Rheumatoid Arthritis |
| RCT | Randomized Controlled Trial |
| S+N | Smith & Nephew, Inc., 1450 E. Brooks Road, Memphis, TN 38116, United States |
| SADE | Serious Adverse Device Effect(s) |
| SAE | Serious Adverse Event(s) |
| SAF | Safety population |
| SAP | Statistical Analysis Plan |
| TKA | Total Knee Arthroplasty |
| UKA | Unicondylar Knee Arthroplasty |
| UL | Upper Limit |
| USADE | Unanticipated Serious Adverse Device Effect(s) |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 22 of 167 |

## 4 INTRODUCTION

## 4.1 BACKGROUND

Arthritis is a clinical syndrome of joint pain accompanied by varying degrees of functional limitation and reduced quality of life. Two common etiologies of arthritis are degeneration of the joint, osteoarthritis (OA), and inappropriate inflammatory response, rheumatoid arthritis (RA). OA is characterized by loss of cartilage, remodeling of adjacent bone, and inflammation in the affected joint [1, 2]. RA is a progressive inflammatory disease that eventually causes systemic joint damage and disability [3]. Post-traumatic arthritis is a form of osteoarthritis following an injury to a joint. Inappropriate joint biomechanics due to deformities is the main risk factor for OA [4]. The joint biomechanics are directly affected by the malalignment of the lower extremities due to anatomical deformities [5]. Varus deformity is an excessive inward angulation of the lower leg and results in a bowlegged appearance. It may cause an overloading and cartilage wear in the medial knee compartment, which could support a degeneration of the knee joint leading to OA [5].

As of 2010, there were approximately 250 million people globally with osteoarthritis of the knee joint (3.6% of the global population) [6]. The prevalence was higher in females than in males [6]. Initial treatment of arthritis may include physical therapy, nonsteroidal anti-inflammatory drugs (NSAIDs) such as ibuprofen and corticosteroids which can be taken orally or by injection.

Avascular necrosis (AVN) has several etiologies but fundamentally results from a decrease in blood flow to the affected bone, leading to cellular death [7]. Studies have reported a 3.4% and 9.4% incidence of spontaneous osteonecrosis in persons older than 50 and 65 years of age, respectively [8]. Initial treatment of AVN may include medication, stretching and not walking on the affected leg.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 23 of 167 |

Complex epiphyseal fractures around the knee joint involve the distal femur or proximal end of the tibia. The management of these fractures especially in elderly patients is challenging [9].

When the damage to the joint is advanced or conservative treatment options are exhausted, knee arthroplasty is considered the most effective treatment for patients with any of these indications.

Total knee arthroplasty (TKA) is a highly successful and frequently performed surgical treatment to reduce disability caused by end-stage osteoarthritis and other conditions affecting articular cartilage [10, 11]. Technical outcomes for TKA are excellent, with favorable postoperative health-related quality of life [12]. Also, survivorship of primary knee replacements is excellent with reported survivorship of 82.3% at 25 years [13]. TKA has traditionally been indicated in the elderly population with relatively sedentary lifestyles, but more active, younger patients (<55) are receiving TKA due to the desire for a pain-free, active lifestyle with the demand projected to continue to increase for this group. A recent systematic review has shown that functional outcomes are similar in this population compared to elderly patients with no increase in the burden of revision [14].

Unicondylar knee arthroplasty (UKA) is a surgical treatment for patients with OA or AVN that only affects a single compartment of the knee [15, 16]. In 2018, 11% of all knee arthroplasties in the United Kingdom were compartmental knee arthroplasties (UKA) [17].

In Australia, 660,000 primary TKAs and 60000 primary UKAs have been performed in 2018. Since 2003, the number of knee replacement procedures undertaken has increased by 128% [18].

The escalating prevalence of end-stage OA places an increased burden on healthcare providers, especially on less experienced surgeons and facilities that

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 24 of 167 |

perform low numbers of arthroplasties [19, 20]. Lower volume hospitals (<25 procedures/year) report higher revision rates and more complications by 5 to 8 years compared to high volume hospitals (>200 procedures/years) [20, 21]. Therefore, technology or techniques that could improve outcomes and reduce the risk of revision are becoming increasingly important.

Surgical factors that must be considered in knee arthroplasty include lower leg alignment, soft tissue balancing, maintenance of the joint line, and component size and fixation [22]. Malalignment of components in any anatomical plane can cause major complications including aseptic loosening, instability, poor function, polyethylene wear, and pain [22-24]. Additionally, implant malposition and malalignment of the joint can result in failure of the prosthesis [25]. When not aligned within a narrow tolerance of  $\leq 3^{\circ}$  of the mechanical axis, poor functional outcomes, decreased implant survivorship, increased wear, and early failure from component loosening may occur [26].

Evidence has shown that neutral mechanical alignment provides optimal outcomes in knee arthroplasty, which is achieved with conventional alignment guides in approximately 75% of TKA cases [27]. For partial knee procedures, approximately 30-60% of UKAs have been reported to be malaligned using conventional manual instruments [28]. The importance of alignment can be demonstrated by observing higher revision rates of UKA attributed to malposition or malalignment of partial knees [28, 29] while roughly 25% of TKAs have been revised for instability or malalignment [30].

As an alternative to mechanical alignment, kinematic alignment technique for knee arthroplasty aims to restore the individual knee anatomy and ligament tension, to restore native knee kinematics [31]. Kinematic alignment restores the obliquity and level of the joint line anatomically so the femoral component is slightly more valgus

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | |

(1° to 2°) and the tibial component is slightly more varus (1° to 2°) than mechanically aligned components.

A significant innovation in knee arthroplasty has been the introduction of computer navigation and robotic-assisted surgery. One such technology is CORI. This system is a semi-autonomous image-free system. During the surgery, the surgeon maps the condylar landmarks and determines alignment indices to define the volume and orientation of bone to be removed. The tools to remove the bone and place the implants are controlled and manipulated by the surgeon with the guidance of a 3-dimensional digital map of the surgical surface.

Comparisons of navigation systems to conventional instruments have demonstrated that robotic platforms produce fewer positioning errors in both UKA and TKA [32-34]. When used in medial or lateral UKA procedures, robotics reported short learning curves, increased accuracy in posterior tibial slope, and coronal tibial alignment in comparison to other alignment methods [35-37].

For China, CORI is an investigational device - for details of the full literature review, pre-clinical, clinical, safety data and a risk analysis refer to the Investigator's Brochure (IB).

#### 4.2 LITERATURE SUMMARY

A thorough analysis of the literature was performed, and publications were identified that contained clinical outcomes, accuracy measurements, or safety information pertaining to the Navigation Knee Surgical Systems.

Use of the Navigation Knee Surgical Systems was reported in 7 publications with 1 being a prospective study and the remaining 6 being retrospective studies shown in Table 4.2-4-1. Three (3) of the studies solely reported on outcomes of the Navigation Knee Surgical Systems, three (3) compared the Navigation Knee Surgical

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 26 of 167 |

Systems to conventional instruments, and one (1) study compared the Navigation Knee Surgical Systems to conventional instruments, patient specific instrumentation (PSI), and computer-assisted navigation (CAS) systems. All of the studies were for the NAVIO $^{\text{TM}}$  Navigation System (NAVIO) and reported outcomes for UKA. The data provided in these publications is also applicable to the equivalent CORI.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 27 of 167 |

Table 4.2-4-1 Demographic Information for the Navigation Knee Surgical Systems

| Primary<br>Author | Year | Navigation<br>System | Indication | Joints<br>(n) | Male<br>(%) | Age,<br>mean±SD<br>(range) | Follow-up,<br>mean±SD |
|---|---|---|---|---|---|---|---|
| Batailler<br>[38] | 2019 | NAVIO <sup>1</sup> | UKA | 80 | 33.8 | 69 ± 9.6<br>(49-87) | 1.64 ±<br>0.75<br>years |
| Battenberg<br>[39] | 2019 | NAVIO <sup>1</sup> | UKA | 128 | 57.8 | 64.7 ± 9.6<br>(45-92) | 2.3 years |
| Canetti [40] | 2018 | NAVIO <sup>1</sup> | UKA | 11 | 18.0 | 66.5 ± 6.8<br>(57-79) | 2.87 ±<br>0.88<br>years |
| Gregori<br>[41] | 2016 | NAVIO <sup>1</sup> | UKA | 92 | - | - | Periop |
| Herry [42] | 2017 | NAVIO <sup>1</sup> | UKA | 40 | 32.5 | 69 ± 9.6<br>(49-87) | Periop |
| Vega Parra<br>[43] | 2017 | NAVIO <sup>1</sup> | UKA | 47 | 51.0 | 67<br>(45-77) | 1 year |
| Sephton<br>[44] | 2019 | NAVIO <sup>1</sup> | UKA | 67 | 49.0 | 68 ± 10 | Periop |
| | | | Total | 414 | 49.0%A<br>(33.8-<br>57.8) | 66.8A<br>(45-92) | 1.14<br>years<br>(Periop-<br>2.87) |

<sup>&</sup>lt;sup>1</sup> NAVIO<sup>™</sup> Surgical System

### 4.2.1 Demographic Information

A total of 414 joints were reported in the reviewed literature. Herry et al.[42] and Canetti et al.[40] likely shared the same patient population as Batailler et al.[38] Therefore, these joints were not included in the total, but these publications were not excluded due to different outcomes being reported among the studies. The Navigation Knee Surgical Systems are used intraoperatively to assist with implantation of knee prostheses, and studies report on a combination of intraoperative alignment parameters, clinical outcomes, and safety information. Three (3) studies provided early postoperative follow-up between the perioperative period and one year post-operative time point. Four (4) additional studies reported follow-up of one year or longer, two of which reported outcomes after 2 years of

| <b>Clinical Protocol</b> | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 28 of 167 |

follow-up. The gender of the patients was almost evenly distributed, as men comprised 49% of the total population from all 7 publications. The age of patients undergoing UKA with the NAVIO ranged from 45 to 92 years with an average age of 66.8 years for the total patient population from all 7 publications.

### 4.2.2 Clinical Outcome

Outcome measures were evaluated in three publications with Knee Society Score (KSS), satisfaction rate, return to sport, Lysholm scale, Forgotten Joint score (FJS-12), University of California, Los Angeles (UCLA) activity scale, Knee injury and Osteoarthritis Outcome Score (KOOS) and Knee Society Function Score (KSFS) being reported.

KSS, KSFS, and satisfaction rates were the most commonly employed outcome measures, being reported by both Batailler et al.[38] and Canetti et al.[40]. These studies reported KSS and KSFS scores ranging from 92.6 to 96.4 and 90 to 97.2, respectively, indicating excellent functional outcomes. Satisfaction was scored on a scale from 1-5 with values corresponding with feeling disappointed to very satisfied. The percentages reported are the number of patients that indicated they were very satisfied with their procedure; this does not include patients that indicated they were just satisfied. Other outcome scores were reported in a single study, and none of these outcomes evidenced reduced function.

Batailler et al.[38] and Canetti et al. compared patients operated on with NAVIO to patients who were operated on using conventional instruments. For KSFS and satisfaction rate, no statistically significant differences were observed between the two groups. However, Canetti et al. observed a statistically significant increase in KSS and quicker return to sport for NAVIO. As the KSS difference was not observed in the larger cohort of Batailler et al.[38], the observed difference may be due to the smaller sample size. The percentage of patients returning to sports, UCLA,

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 29 of 167 |

Lysholm scale, and FJS-12 were not statistically significant between the two cohorts.

Overall, patients undergoing knee procedures with NAVIO showed improved KSS, KSFS, KOOS, and UCLA scores compared to pre-operative values.

# 4.2.3 Mechanical Alignment Accuracy

The Navigation Knee Surgical Systems are intended to assist in planning and executing a procedure involving bone preparation for UKA procedures. Publications have provided accuracy measurements for the Navigation Knee Surgical Systems themselves and compared to conventional instruments. Three (3) publications investigated alignment accuracy in various planes, the incidence of outliers, and restitution of the joint line [38, 41, 42].

The reviewed publications indicate that the Navigation Knee Surgical Systems can produce the desired mechanical axis, hip knee ankle angle, coronal femoral angle, coronal tibial angle, tibial slope, and joint line deviation in the majority of cases. Outliers were reported for most of the angular alignment parameters, and only one study indicated a rate higher than 15% [38]. This increased outlier rate is likely due to the decreased tolerance imposed by the authors as outliers were defined as being within 2° of the desired value compared to the standard 3°.

Batailler et al.[38] and Herry et al.[42] compared alignment with NAVIO to conventional instrumentation. Statistically significant differences were not observed between the hip knee ankle angle or tibial slope for medial or lateral UKAs. However, there were statistically fewer outliers for NAVIO in the hip knee ankle angle for medial and lateral UKA, the tibial slope for medial UKA, and the coronal tibial angle. In addition, the joint line was significantly less distalized when NAVIO was used.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 30 of 167 |

Using the Navigation Knee Surgical Systems results in a knee prosthesis that is well aligned and implanted according to the surgical plan. This is supported by satisfactory angular outcomes in the mean mechanical axis, hip knee ankle angle, coronal femoral angle, coronal tibial angle, and tibial slope. In addition, the joint line was less distal compared to when conventional instrumentation was utilized.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 31 of 167 |

# 4.2.4 Adverse Events & Complications

Complications related to the surgery, revision of the implant, and general complications were reported in the 7 included publications. Overall, the revision rate for prostheses implanted using the Navigation Knee Surgical Systems was 1.2% (5/414 procedures). Revisions were due to aseptic loosening without implant malpositioning (3, 0.7%) and unexplained pain (2, 0.5%). Additional reoperations included three (3) arthroscopic partial lateral meniscectomies, two (2) arthroscopic arthrolyses, and one (1) arthrotomy and lavage. Batailler et al.[38] noted that complications that affect robotic-assisted techniques (e.g., pin-site infections, broken pins, or fractures at the pin site) did not occur in their cohort.

#### 4.2.5 Conclusion

Using the Navigation knee surgical systems results in a knee prosthesis that is implanted according to the patient specific surgical plan. This is evidenced by satisfactory angular outcomes and restitution of the joint line. In addition, patients undergoing these procedures with the Navigation knee surgical systems showed improved outcomes scores compared to pre-operative values. The clinical outcomes, alignment accuracy, and adverse events for the Navigation Knee Surgical Systems reported in the literature are similar to those reported for comparable devices.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 32 of 167 |

## 4.3 STUDY PURPOSE

This is a prospective, multi-center, randomized controlled study to demonstrate the safety and effectiveness of CORI to support the regulatory approval by the National Medical Products Administration (NMPA) in China. Data collected in this study may also be used to maintain product registration in global markets including, but not limited to, Australia (Therapeutic Goods Administration (TGA)) and Europe (Conformité Européene (CE)).

#### 4.4 SAFETY CONSIDERATIONS

CORI's intended use, indications and contraindications can be found in the User's Manual & Instructions for Use (IFU) for Australia, China (Hong Kong), South Korea, and New Zealand or the Investigator's Brochure for China Mainland.

#### 4.4.1 Intended Use

CORI is intended to assist the surgeon in providing software-defined spatial boundaries for orientation and reference information to anatomical structures during orthopedic procedures.

#### 4.4.2 Indications

CORI is indicated for use in surgical knee procedures, in which the use of stereotactic surgery may be appropriate, and where reference to rigid anatomical bony structures can be determined. These procedures include unicondylar knee replacement (UKR) and total knee arthroplasty (TKA).

CORI is indicated for use with cemented implants only.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 33 of 167 |

## 4.4.3 Contraindications

CORI is not intended to be used on children, pregnant women, patients who have mental or neuromuscular disorders that do not allow control of the knee joint, or any other patients contraindicated for knee replacement.

#### 4.4.4 Environments of Use

CORI is intended to be used by trained medical professionals in a hospital or clinical setting equivalent to an orthopedic surgery suite. The CORI Instruments will be used in a sterile environment and must be sterilized prior to use.

#### **4.4.5 Potential Adverse Effects**

As with any surgical procedure, there is risk involved. Potential complications accompanying surgery may occur, including allergic reaction (anaphylactic and minor), infection, mild to serious physical injury, localized static shock, delay in the operation, surgical site nerve injury, vascular injuries of the lower extremity, soft tissue damage, major bone gouging at the surgical site, bone fracture, immature implant failure, unstable knee joint, limited or restricted knee range of motion, major blunt impact injury, unintended laceration/puncture wound, and osteonecrosis.

The CORI User's Manual (Document ID: 500230, REAL INTELLIGENCE™ CORI™ for Knee Arthroplasty) states the following warnings and cautions:

CORI is a surgical tool designed to provide assistance to the surgeon; it is not
a substitute for the surgeon's experience and skill. The surgeon is responsible
for implant planning and the conduct of the surgery during which CORI is being
used.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 34 of 167 |

- CORI and accessories should be used only by, or under the supervision of, a qualified surgeon or qualified member of his or her staff who is familiar with this document and has received training from S+N.
- Use of equipment not specifically designated in this manual as compatible with CORI may result in the system not functioning properly, leading to patient or user injury.
- Refer servicing only to trained service personnel. Equipment damage, personal injury, or death may result if CORI is not serviced properly.
- To avoid risk of electrical shock, only connect the CORI Cart to a supply main with protective earth.
- Modification of CORI can cause the system to malfunction and could result in user and/or patient injury.
- Connecting electrical equipment to the multiple socket output effectively leads to creating a Medical Equipment System and could result in a reduced level of safety.
- The transformer outlet is only to be used for CORI components. Do not connect
  any other device or improper extension cord to the transformer (max. load 600
  VA) outlet. Failure to comply with this warning may result in shock hazard or
  product damage.
- Additional equipment connected to medical electrical equipment must comply with the respective IEC or ISO standards. All configurations shall comply with the requirements for medical electrical systems (see IEC 60601-1). Anyone connecting additional equipment to medical electrical equipment configures a medical system and is therefore responsible that the system complies with the requirements for medical electrical systems. Attention is drawn to the fact that local laws take priority over the above-mentioned requirements. If in doubt, contact a qualified Biomedical technician or your local Smith & Nephew representative.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 35 of 167 |

- Any person who connects external equipment to signal input and signal output ports or other connectors has formed a system and is therefore responsible for the system to comply with the requirements of IEC 60601-1. If in doubt, contact a qualified Biomedical technician or your local Smith & Nephew representative.
- Only USB-powered devices, such as USB flash drives, should be connected to CORI USB ports. Any person that connects a self-powered USB device has formed a medical system and is therefore responsible for the system to comply with the requirements of IEC 60601-1. If in doubt, contact a qualified Biomedical technician or your local Smith & Nephew representative.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 36 of 167 |

# 5 OBJECTIVE(S)

### **5.1** PRIMARY OBJECTIVE

The primary objective of this study is to evaluate the use of CORI in UKA procedures in achieving post-operative leg alignment as compared to procedures using conventional manual instruments.

# **5.2 Secondary Objective(s)**

The secondary objective of this study is to generate safety and performance evidence supporting the use of CORI procedures. To assess the safety and performance of CORI up to 12 months after surgery as compared to procedures using conventional manual instruments.

# 5.3 OTHER OBJECTIVE(S)

Other objectives are to collect the system time and cutting time of the robotic drill from the CORI Case Report.

## 5.4 CLAIMS

No claims to be confirmed by this investigation.
| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 37 of 167 |

# **6 INVESTIGATIONAL PRODUCT(S) AND COMPARATOR**

#### **6.1 IDENTIFICATION**

## 6.1.1 Investigational Product

CORI is a computer-assisted orthopedic surgical navigation and burring system. It is designed to aid surgeons in planning and executing a procedure involving bone preparation for unicondylar knee arthroplasty (UKA) and total knee arthroplasty (TKA) procedures.

CORI is currently available for the use of the following S+N UKA implant Systems, the implant system will be selected according to the registration status in each country.

Table 6.1-6-1 S+N Implant Systems available with CORI

| Implant System | Manufacturer |
|------------------------------------------|----------------------|
| Journey II Unicompartamental Knee System | Smith & Nephew, Inc. |
| Journey Uni | Smith & Nephew, Inc. |

CORI is comprised of a console control unit, optical tracking camera, primary and secondary input displays (tablet and optional display monitor), instrument trays and foot pedal (Figure 6.1-6-1). CORI software consists of a patient and user management module, a surgical planner, and an intra-operative cutting module. The system uses the tracked position of the surgical bur to control its cutting engagement to the bone that is intended to be removed. This cutting control is based on the bur's proximity to the planned target surface of the bone.

CORI incorporates a detailed user interface that provides procedure setup, tracking status, visual indicators, and real-time cutting progress during the procedure. The system uses the tracked position of the surgical bur to control its cutting engagement to the bone that is intended to be removed. The cutting control is based on the bur's proximity to the planned target surface of the bone. CORI

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 38 of 167 |

software controls the cutting engagement of the surgical bur based on its proximity to the planned target surface. The cutting control is achieved with two modes:

- Exposure control adjusts the bur's exposure with respect to a guard. If the surgeon encroaches on a portion of bone that is not to be cut, CORI retracts the bur inside the guard, disabling cutting.
- Speed control regulates the signal going to the drill motor controller itself and limits the speed of the drill if the target surface is approached. This mode of operation is useful in shaping surfaces of the condyle as well as placing post holes and fixation features for femoral and tibial cut guides.

The surgeon can disable both controls and operate CORI robotic drill as a standard navigated surgical drill.



Figure 6.1-6-1 CORI





• **Console:** It houses the robotic drill tool control, power management, video and audio distribution, central processing unit, and irrigation pump/control.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 39 of 167 |

- Optical Tracking Camera: It is used to determine the position of the surgical bur tip and point probe relative to the position of the tibia and femur tracker frames. The position is determined using reflective markers affixed to the robotic drill, point probe, and tibia and femur frames.
- **Foot Pedal:** The left foot pedal allows variable input for robotic drill speed control and provides navigation or confirmation action in certain situations. The right pedal and small circular buttons are used to navigate forward and backward in the workflow and dismiss error messages.
- Tablet: The wired display monitor provides a touchscreen interface for the user to interact with the system.
- Display Monitor: It provides duplicate display and control of the system user interface.
- **Cart:** It provides a location for the system console, mounting for the optical tracking camera and display monitor, and storage for the foot pedal, tablet, and power cords.
- CORI Instrument Trays UKA & TKA: There are two instrument trays, one
  for unicondylar knee arthroplasty (UKA) and for total knee arthroplasty (TKA)
  procedures. Both CORI instrument trays contain reusable, re-sterilizable tools
  to assist in surgical site preparation, implant placement planning, and bone
  removal. The tray is comprised of two levels.
  - \*Only UKA related components will be used for the study.

CORI also includes specific reusable instruments as shown in Figure 6.1-6-2.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 40 of 167 |

Figure 6.1-6-2 CORI Reusable Instruments



**CORI Robotic Drill** 

Checkpoint Pins Bone Screw

- **CORI Robotic Drill:** Controls the position and speed of the bur. It is intended for 75 uses and is able to be autoclaved, auto washed, and disinfected.
- **Point Probe:** Tracked instrument used in robotic drill calibration, and bone registration, checkpoint verification.
- Femur & Tibia Trackers: Rigid arrays placed on the femur and tibia to track
  the relative position of bones to point probe and robotic drill tools using
  reflective markers.
- **Checkpoint Pins:** placed in femur and tibia and checked periodically with the point probe to verify that the tibia and femur tracking arrays have not moved during the procedure.

Details on single use instruments of CORI can be found in Section 22.3.

CORI, as well as the single use components, are manufactured by Smith+Nephew, Blue Belt Technologies, 2905 Northwest Blvd. Suite 40, Plymouth, MN 55441, USA

### **6.1.2 Comparator Treatment**

CORI will be compared to conventional manual instrumentation currently available in Australia, China (Hong Kong), New Zealand, South Korea, and China Mainland.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep<br>2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 41 of 167 |

Arthroplasty has traditionally used conventional manual instruments to guide placement of the implant and determine bone resection in reference to anatomical landmarks. Manual instruments include intramedullary or extramedullary rods that centralize and align the components according to the surgical plan as shown in Figure 6.1-6-3 & Figure 6.1-6-4.

Figure 6.1-6-3 Extramedullary rod Figure 6.1-6-4 Intramedullary rod





6.1.3 Ancillary Product(s)

Not applicable.

#### 6.2 PRODUCT USE

CORI has a user's manual (Document ID: 500230, REAL INTELLIGENCE™ CORI™ for Knee Arthroplasty). The purpose of this user's manual is to serve as the master reference document for properly trained users in the function and operation of CORI and its accessories.

In addition, the following devices are packaged with an IFU to ensure that the device is used properly and for the intended purposes:

#### 

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 42 of 167 |

- IFU REAL INTELLIGENCE™ CORI™ Burs (Document ID: 500172)
- IFU REAL INTELLIGENCE™ CORI™ Flat Markers (Document ID: 500198)
- IFU REAL INTELLIGENCE™ CORI™ Irrigation (Document ID: 500173)
- IFU REAL INTELLIGENCE™ CORI™ Instrumentation Tray (Document ID: 500229)

For Australia, Hong Kong, South Korea, and New Zealand the list of reference documents can be found in Appendix Section 22.3Instruction For Use & User Manual.

For China mainland, details of the use of CORI can be found in the Investigator's Brochure.

### 6.3 PACKAGING AND LABELLING

Packaging and labeling are prepared to meet regulatory requirements. Package integrity and labelling should be verified prior to use of the product and confirmed in the eCRF.

## 6.3.1 Labelling of Investigational Product

All product components of the CORI System are commercial products in the Australia, China(Hong Kong), South Korea, and New Zealand and are being used as approved. Labeling is done as per the standard commercial packaging.

In China mailand, CORI is a an investigational product. The standard commercial packaging as marketed in the US is used. However, additional labels will be included on the commercial packaging to meet the regulatory requirements for investigational devices in countries where the devices are not approved for marketing.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 43 of 167 |

Compatible S+N Knee Implant Systems are commercial products in Australia, China (Hong Kong), New Zealand, and China mainland and are being used as approved.

## **6.3.2 Comparator Product**

Conventional approach with conventional manual instrumentation will be used as the comparison group and there will be no packaging involved with the conventional approach.

S+N Knee Implant Systems are commercial products in Australia, Hong Kong, New Zealand, South Korea, and China mainland and are being used as approved.

#### **6.4 Product Accountability Procedures**

This study is a post-market study in Australia, Hong Kong, South Korea, and New Zealand. However, the sponsor provides the study sites with CORI System (Console, Optical Tracking Camera, Foot Pedal, Tablet, Display Monitor, Cart, CORI Instrument Trays UKA) as well as with reusable instrumentation (CORI robotic Drill, Point Probe, Femur & Tibia Trackers, Checkpoint Pins). Therefore, the following product accountability procedures will be applied for CORI at all study sites.

The investigational site will maintain an inventory of the investigational product. The Sponsor or its designee will provide a log(s) to facilitate IP inventory control. The log will contain details of receipt, use, returns etc. of IP. All IP accountability logs must be retained in the Investigator Site File (ISF). These records must be available for inspection by the Sponsor, its designees, or by regulatory agencies at any time.

The Study Monitor will ensure that the procedures and records are in place for the appropriate reconciliation of all IP. As part of monitoring, the Study Monitor will check that site personnel are following the proper procedures for accountability and completing all necessary documentation.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 44 of 167 |

No product accountability procedures will be applied for the S+N Knee Implant Systems as these are commercially available products.

For details on CORI and reusable instrumetation please refer to Section 6.1.1 Investigational Product.

## **6.5** Surgical Technique

All study related procedures with CORI must be performed according to the user's manual (Document ID: 500230 CORI Robotics for Knee Arthroplasty for Australia, Hong Kong, South Korea, and New Zealand, as well as Investigator's Brochure for China) and according to the according to the surgical technique and IFU of the specific S+N Implant System.

Surgeons selected to participate in this study will be familiar with CORI and have written evidence of training and expertise in the study procedure. The Surgeon will conduct Pre-study in order to establish the expertise of the individual surgeons. The exact number of pre-study cases may be adjusted depending on the level of the individual experience of the surgeon.

CORI Case Reports Forms of the non-randomized cases will be collected as proof of surgeons' experience and for inclusion in the safety analysis set (applicable only at sites in China).

#### **6.6 Medical Procedure**

There are 3 basic steps in unicondylar knee arthroplasty. The first step is preparing the bone and removing the cartridge from the damaged knee compartment. This will be completed using either the CORI robotic drill or an oscillating saw. The surgeon will then position the metal implants on the damaged side of the femur and tibia using several orthopaedic tools. Finally, a spacer will be inserted between the metal implants to reduce friction when the knee flexes and extends. At various times during

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 45 of 167 |

the procedure, the hip-knee-ankle angle (HKA) will be checked using the CORI advanced tracking system or via the use of intramedullary and / or extramedullary rods. How the angle is measured will depend on which treatment arm the subject is randomized to receive. All unicondylar knee arthroplasty is completed using general anaesthetic by a surgical team trained in both the CORI system and the use of standard manual instrumentation.

### 7 SUBJECT ENROLLMENT AND WITHDRAWAL

#### 7.1 SUBJECT POPULATION

At least 145 subjects will be enrolled into the study. At least 5 of these subjects will be treated with CORI directly to fulfil the learning needs of the surgeons prior to enrolling, a further 140 subjects who will be enrolled in the randomized stage of the study in up to 8 sites in Australia, Hong Kong, New Zealand, South Korea, and China mainland. Seventy (70) subjects will be enrolled for UKA with the use of the CORI and 70 subjects will be enrolled for UKA with the use of conventional manual instrumentation. Vulnerable subjects will not be enrolled in this study.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 46 of 167 |

### 7.2 INCLUSION CRITERIA

Subjects will be considered qualified for enrollment if they meet the following criteria:

- Subject is a suitable candidate for a UKA procedure using CORI and a compatible S+N Knee Implant System.
- 2 Subject requires a cemented UKA as a primary indication that meets any of the following conditions:
  - a) Non-inflammatory degenerative joint disease, including osteoarthritis
  - b) Avascular necrosis
  - c) Requires correction of functional deformity
  - d) Requires treatment of fractures that were unmanageable using other techniques
- 3 Subject is of legal age to consent and considered skeletally mature (≥ 18 years of age at the time of surgery)
- Subject agrees to consent to and to follow the study visit schedule (as defined in the study protocol and informed consent form), by signing the Ethics Committee (EC) or Institutional Review Board (IRB) approved informed consent form.
- 5 Subject plans to be available through one (1) year postoperative follow-up.
- 6 Applicable routine radiographic assessment is possible.

#### 7.3 EXCLUSION CRITERIA

Any one (1) of the following criteria will disqualify a potential subject from participation in the study:

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 47 of 167 |

- Subject receives a UKA on the index joint as a revision for a previously failed surgery, or need for complex implants, or any other implant than a standard UKA (e.g. stems, augments, or custom made devices).
- 2 Subject has been diagnosed with post-traumatic arthritis
- 3 Subject receives simultaneous bilateral UKA OR a unilateral UKA with contralateral TKA.
- 4 Subject has one or more of the following arthroplasties that are not fully healed and well-functioning, as determined by the investigator:
  - -Contralateral primary TKA or UKA, however, the subject can only have one knee enrolled in the study.
- 5 Subject does not understand the language used in the Informed Consent Form.
- 6 Subject does not meet the indication or is contraindicated for UKA according to specific S+N knee system's Instructions for Use (IFU).
- 7 Subject has active infection or sepsis (treated or untreated).
- 8 Subject is morbidly obese with a body mass index (BMI) greater than 40.
- 9 Subject is pregnant or breast feeding at the time of surgery.
- 10 Subject, in the opinion of the Investigator, has advanced osteoarthritis or joint disease at the time of surgery and was better suited for an alternate procedure.
- 11 Subject currently enrolled in another orthopedic clinical trial study.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 48 of 167 |

- Subject has a condition(s) that may interfere with the UKA survival or outcome (i.e., Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease, or an active, local infection).
- Subject in the opinion of the Investigator, has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, intellectual disability, drug or alcohol abuse.
- 14 Subject, in the opinion of the Investigator, has a neuromuscular disorder that prohibited control of the index joint.
- 15 Subject is a prisoner or meets the definition of a Vulnerable Subject per ISO 14155:2020 Section 3.55.<sup>1</sup>

<sup>&</sup>lt;sup>1</sup> ISO 14155:2020 Section 3.55 States: Vulnerable subject – Individuals who are unable to fully understand all aspects of the investigation that are relevant to the decision to participate, or who could be manipulated or unduly influenced as a result of a compromised position, expectation of benefits or fear of retaliatory response

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 49 of 167 |

## 7.4 SCREENING

Investigators should consecutively screen all subjects presenting with degenerative joint disease of the knee, requiring correction of functional deformity, or treatment of fractures that were unmanageable using other techniques to determine whether they meet all inclusion and none of the exclusion criteria.

Participating study sites are required to document all screened subjects considered for inclusion in this study. If a subject is excluded from the study, the reasons for exclusion will be documented in the subject's source documents and noted on the Screening and Enrollment Log. All screening activities that occur prior to consent shall be referred to as pre-screening.

In China sites, part of the screening process will include documentation of women's childbearing potential. If the woman is not of childbearing potential this should be documented in the medical history (e.g., surgically postmenopausal, postmenopausal [i.e., at least one year without menses]). For women of childbearing potential, their method of birth control should be documented in the source.

#### 7.5 INFORMED CONSENT

Before conducting any study procedures or examinations, the purpose and nature of the study should be explained to the subject in their native language.

The subject, or their legally authorized representative (if applicable), will then **read**, **sign**, and **personally date** the IRB/IEC-approved informed consent document(s) (see below for difficulties with reading and writing). Additionally, the individual who obtains consent from the subject will sign and date the informed consent document.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep<br>2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 50 of 167 |

A copy of the signed informed consent document will be provided to the subject, a copy will be placed in the subject's medical record, with the original filed in the ISF.

If the subject is unable to read, the informed consent document and associated study information may be read aloud to the subject in the presence of an impartial witness. If possible, the subject shall sign and personally date the Informed Consent Form (ICF). Where this is not possible, due to difficulties in writing, the subject shall provide verbal consent to participate in the study. The witness shall then personally sign and date the informed consent form, attesting that the information was accurately explained and that the informed consent was freely given.

ICFs will comply with applicable laws and regulations in Australia (Privacy Act 1988), China, South Korea, and New Zealand (Privacy Act 1993). If new information becomes available during the course of the study that can significantly affect a subject's future health and medical care, Smith + Nephew will ensure that information shall be provided to the subject(s) affected in written form and if relevant, all affected subjects shall be asked to confirm their continuing consent in writing.

#### 7.6 ENROLMENT

Subjects for whom the consent process has been completed and have been treated with the study product are considered enrolled.

Subjects that provided informed consent but do not receive the study treatment for any reason will be considered as screen failure.

### 7.7 LOST TO FOLLOW-UP

A subject will be considered lost to follow-up if he/she does not appear for the scheduled study visit for two (2) consecutive visits, and study personnel is unable to contact the subject.

#### 

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 51 of 167 |

Some actively enrolled subjects will not return for follow-up exams on time. Study personnel must make a reasonable effort to contact the subject and document the following contact attempts before declaring a subject to be lost to follow-up: the subject has been contacted according to the site's policies, but no fewer than two documented phone contacts and one certified letter without response. Copies of all attempts to reach the subjects by mail or email and/or the attempts to contact the subject via other means should be documented, and that documentation should be kept with the subject's source documents.

#### 7.8 WITHDRAWAL

#### 7.8.1 Withdrawal from Treatment

Subjects may be withdrawn early from having the study treatment at a date close to surgery or during surgery for the following reasons:

- At the discretion of the Investigator due to:
  - A change in treatment is clinically warranted
  - An adverse event
  - o Any other significant reason identified by the Investigator

### 7.8.2 Withdrawal from Study

The Investigator may withdraw subjects from the study for many reasons, including but not limited to the following:

- Subject noncompliance (e.g., did not follow instructions, took disallowed medications)
- Subject is lost to follow-up
- The Investigator or the Sponsor terminates the study for any reason
- Concurrent illness
- Adverse Events/Adverse Device Effects

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 52 of 167 |

Any other significant reason identified by the Investigator

For each case, the information will be recorded in the subject's source document and the electronic Case Report Form (eCRF), detailing circumstances leading to the withdrawal.

Subjects who withdraw or are withdrawn by the investigator cannot be re-enrolled in the study. Withdrawn subjects will not be replaced.

If at any point during the study, the unicondylar prosthesis needs to be revised for any reason the following will apply: Subjects shall continue to have follow-up visits in order to monitor the subject's health status. Potential data following the revision surgery will not be included as study data but presented separately as safety data.

For minor revisions, where not the whole knee implant system is replaced (e.g. replacement of inserts) the subject shall continue with the study specific schedule and data will be presented.

# 7.8.3 Subject's Withdrawal of Consent to Participate in the Study

Study participation is voluntary, and subjects may withdraw from the study at any time. Where subjects withdraw consent, the Investigator should make a reasonable effort to ascertain the reason(s), while fully respecting the subject's right to privacy. The reason for withdrawal will be recorded in the eCRF and source documents.

### 7.8.4 Use of Data Following Withdrawal

In cases where the subject withdraws consent, the data collected up to the point of withdrawal may be used, but no additional data for that subject may be collected.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 53 of 167 |

#### 8 STUDY DESIGN

#### 8.1 STUDY DESIGN

This study is a prospective, multi-center, randomized controlled, non-blinded follow-up study to evaluate the use of CORI in UKA procedure in achieving post-operative leg alignment. Up to 8 sites will participate within Australia, China (Hong Kong), New Zealand, South Korea, and China Mainland.

The pre-randomized stage of the study will comprise of at least 5 subjects enrolled and treated with CORI directly in order to fulfil the learning needs of the surgeons. Subjects who will comprise the randomized stage of the study will be enrolled and randomized into one of two (2) groups, as shown in Table 8.1-8-1.

All groups are treated with knee arthroplasty with a S+N Knee Implant System. (The implant system will be selected according to the registration status in each country).

**Table 8.1- 8-1 Overview of Study Groups** 

| Surgery | Knee Implant system | Surgical Technique (Groups) | Number of Subjects |
|---|---|---|---|
| D : 111/A | S+N UKA Implant | CORI | 70 |
| Primary UKA | System (Journey II | CON | , 3 |
| | Unicompartamental Knee | Conventional manual | 70 |
| | System, Journey Uni) | instrumentation | 70 |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 54 of 167 |

Figure 8.1-8-1 Study Recruitment Timeline

| August | March | April | March | April |
|---------|------------|-------------------------|---------|----------|
| 2020 | 2022 | 2022 | 2024 | 2025 |
| USA Mar | KEL ACCESS | ining &<br>-study Cases | rolment | ollow-up |

The study is expected to enroll all subjects within a 12-month timeframe. Subjects will be followed-up for a time period of 12 months after surgery. Figure 8.1-8-1 details the Study Recruitment timeline.

This study is being conducted in parallel to a global cohort study titled: "A Prospective, Multi-center Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) and total knee arthroplasty (TKA) Procedures" (Protocol ID: CORI.2019.07). The study data may be combined for analysis. Further details are described in Section 10 Statistical Design and the Statistical Analysis Plan (SAP).

Figure 8.1-8-2 details the different steps of study conduct from screening to enrollment and follow-up.

Subjects may be assigned a subject ID, but then not enrolled in the study (e.g. did not receive the study device or decided not to participate in the study).

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 55 of 167 |

Figure 8.1-8-2 Study Flowchart



## **8.2 ALLOCATION AND BLINDING**

### **8.2.1 Treatment Allocation**

Subjects will be randomly assigned to the CORI navigational or conventional manual instrumentation groups according to a balanced randomization procedure using a 1:1 allocation ratio. To ensure balanced group assignment within each investigational site, a block (by investigational site) randomization schedule will be generated. Only sites will be included that are willing to perform both, CORI Navigated and conventional instrumentation UKA procedures. Subjects who satisfy all inclusion and exclusion criteria will be randomized in a 1:1 randomization allocation ratio. The block size should be sufficiently small to allow approximately equal allocation of subjects in each group should the study be terminated prematurely whilst also being large enough so as the next treatment cannot be guessed.

#### 

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 56 of 167 |

## 8.2.2 Blinding

The study is non-blinded.

#### 8.3 DATA MANAGEMENT

This study utilizes a validated, encrypted electronic data capture system that is 21 CFR Part 11 compliant. Access to the electronic data capture system is restricted by study role in accordance with Smith and Nephew procedures.

A Data Management Plan (DMP) is written according to Smith and Nephew procedures containing details of the data management process. The following is a brief description of the key points detailed in this plan.

## 8.3.1 Data Review and Quality Assurance

Data will be transcribed from the data source to an electronic Case Report Form (eCRF). All data requested on the eCRFs are considered required. Data points not collected and/or recorded will be considered deviations unless otherwise specified.

Data collection is the responsibility of the clinical trial staff at the site under the supervision of the Principal Investigator. The Principal Investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported. The Principal Investigator must provide his/her electronic signature on the appropriate eCRFs to be documented in compliance with local regulations. Changes to data previously submitted to the sponsor will require a new signature by the Investigator to acknowledge/approve the changes.

Visual and computer data review will be performed in line with Smith and Nephew procedures to identify possible data discrepancies. Manual and automatic queries will be created within the electronic data capture system, and will be issued by Smith and Nephew to the site for appropriate response. Site staff are responsible for resolving all queries in the electronic data capture system.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 57 of 167 |

#### 8.3.2 Retention Period

All eCRFs will be archived once the study is completed and will kept for a period of no less than five years after the later of the following dates: the date of which the study is terminated or completed or; the date that the records are no longer required supporting marketing applications.

#### **8.4 STUDY ENDPOINTS**

## 8.4.1 Primary Endpoint

The primary endpoint of this study is defined as the evaluation of the proportion of subjects achieving planned post-operative leg alignment. Achieved leg alignment is defined as  $\pm$  3° from the subject's specific target in comparison with conventional manual instrumentation.

## 8.4.2 Secondary Endpoints

The following secondary endpoints have been defined for this study in order to evaluate the safety and performance of CORI in comparison with conventional manual instrumentation up to 12 months post-operatively:

- Component Alignment
- Radiographic assessment (Presence of radiolucent lines, osteolysis & implant migration)
- 2011 Knee Society Score (2011 KSS)
- Oxford Knee Score (OKS)
- Forgotten Joint Score (FJS-12)
- Five-level EuroQol five-dimensional (EQ-5D-5L) VAS & index scores

### 8.4.3 Other Endpoints

The following additional endpoints have been defined for this study:

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 58 of 167 |

- Leg alignment pre- and post-cementation for CORI UKA
- Navigations System time as extracted from the Subject's CORI Case Report generated by the CORI Software.
- Cutting time of the robotic drills extracted from the Subject's CORI Case Report, generated by the CORI Software.

## 8.4.4 Safety Endpoints

Safety endpoints include the collection of the following events:

- All adverse events (AEs) and complications occurring from the time of subject enrollment until study termination or study completion including intraoperative adverse events and complications.
- Device related re-intervention
- Device Deficiencies
- Knee implant revision rate

#### 8.5 METHODS USED TO MINIMIZE BIAS AND MAXIMIZE VALIDITY

### 8.5.1 Multiple sites

After fulfillment of all eligibility criteria (including informed consent), subjects will be enrolled and randomized at multiple sites, utilizing up to 8 sites in total for the study. Subject enrollment will continue until the completion of recruitment of a minimum of 140 subjects. File records and enrollment registration forms for screening work must be retained and submitted to the Sponsor as needed.

## **8.5.2 Prospective Consecutive Enrolment**

Subjects meeting all inclusion/exclusion criteria will be randomly allocated to one of two treatment groups (CORI Navigational versus conventional manual instrumentation) in a 1:1 allocation ratio. Blocked randomization to balance this allocation ratio by investigational site and overall will be implemented through a

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep<br>2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 59 of 167 |

network-based randomization system. A randomization number is allocated only when subjects have signed the Informed Consent Form and satisfy all study eligibility criteria.

## **8.5.3 Subject Attrition**

Subject attrition for the sample size has been accounted for in the sample size estimation.

## 8.5.4 Pre-specification of Statistical Analysis

The primary outcome measure has been pre-specified as well as the type of statistical analysis to be performed in order to evaluate this outcome. The details of all analyses to be performed will further be pre-specified in the Statistical Analysis Plan (SAP) so as to minimize any threats to external validity and yield clinically relevant estimates of effects and precision.

#### 9 STUDY PROCEDURES

#### 9.1 VISITS AND EXAMINATIONS

### **9.1.1 Summary**

For a summary of the required procedures by visit, refer to the Study Schematic Table 9.1.1-9-1 Study Procedures by Visit.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | |

Table 9.1.1-9-1 Study Procedures by Visit

| Schedule of events | Pre-<br>Operative<br>Data<br>-90 to 0<br>days | Operative Data & Discharge Day 1 (+ up to 9 days) | 42 ± 14 | 6 months<br>185 ± 14<br>days | 12<br>months<br>365 ± 30<br>days |
|---|---|---|---|---|---|
| Informed Consent | x | | | | |
| Demographics/<br>Medical History | x | | | | |
| Inclusion/Exclusion | x | | | | |
| Preoperative Examinations (eg. ECG, Blood Routine Examination, Biochemical Examination, Coagulation Examination) <sup>1</sup> | x | | | | |
| Pregnancy Test <sup>2</sup> | х | | | | |
| Concomitant<br>Medication | х | | | | |
| Concomitant<br>Medication Update | | x | x | X | x |
| Operative Data<br>Collection | | x | | | |
| CORI Case Report (System time & cutting time) | | x | | | |
| Discharge Data<br>Collection | | x | | | |
| Leg alignment Long<br>leg X-ray AP <sup>3</sup> | x | (x) <sup>4</sup> | х | | (x) <sup>5</sup> |
| Standard Lateral X-ray | | (x) <sup>4</sup> | х | | х |
| Standard A/P X-ray | | | | | х |

#### 

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 61 of 167 |

| KSS | х | | х | х | х |
|-------------------|---|---|------------------|------------------|---|
| OKS | х | | х | х | х |
| FJS-12 | | | х | х | х |
| EQ-5D-5L | х | | х | х | х |
| Safety Assessment | | х | х | х | х |
| End of Study/Exit | | | (x) <sup>6</sup> | (x) <sup>6</sup> | х |

- Only applicable at sites in China
- <sup>2</sup> Only Applicable at site in China
- Pre-operative long leg X-rays (A/P) collected 6-months prior to the date of surgery is admissible
- Post-operative standing weight bearing long leg X-rays (A/P) and standard lateral X-rays may be taken at discharge.
- Only if standing weight bearing long leg A/P X-ray is taken as a standard of care at 12 months.
- <sup>6</sup> Exit form to be completed at the point of withdrawal if the study is not completed.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 62 of 167 |

## 9.1.2 Screening/Pre-operative Visit

1. Obtain written informed consent from the subject as detailed in Section 7.5.

## ---- Do not proceed until the consent has been obtained -----

- 2. Obtain demographic information and medical history, including information on all concomitant medications/therapies.
- 3. Screen the subject for protocol inclusion/exclusion criteria.
- 4. The eCRF will assign the subject a study number. The subject identification log shall be completed accordingly.
- 5. Instruct the subject on treatment procedures.
- Collect radiographic images of the affected knee for evaluation of leg alignment (Standing weight bearing A/P long leg X-ray).
- 7. Collect the 2011 KSS score objective measures (joint alignment, instability, motions & symptoms).
- 8. Have the subject complete the 2011 KSS score subject questions.
- 9. Have the subject complete the OKS patient-reported outcome measure.
- 10. Have the subject complete the EQ-5D-5L patient-reported outcome measure.
- 11. The subject will be randomized to treatment group (CORI or Manual conventional instrumentation).
- 12. Subjects will be instructed to return for the Operation Visit on a scheduled date.

### 9.1.3 Operation Visit & Discharge (Day 1+up to 9 days)

1. Prior to surgery, check if there is any change in eligibility of the subject since the pre-operative visit. If the subject is no longer eligible, document as screening failure.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 63 of 167 |

- 2. Query subject regarding any changes in general health and the use of concomitant medications/therapies.
- 3. Collect data on the surgical plan: Target Leg alignment.
- 4. Perform surgery and collect intra-operative data on the appropriate eCRF.

  This includes but is not limited to the following information:
  - Knee Implant Data
  - Surgical data (e.g. duration, blood loss, surgical approach)
  - Collect pre- (with the trial implant in place) and post cementation alignment with the use of CORI.
  - Collect the Subject's CORI Case Report, generated CORI Software (System time, cutting time) for CORI group.
- 5. Complete discharge eCRF.
- 6. If any adverse device effects or device deficiencies are observed or reported, they must be recorded as instructed in Section 12 Adverse Events and Device Deficiencies.
- 7. Instruct the subject on proper postoperative care/procedures.
- 8. Instruct the subject returning to the site for the next follow up visit 6 weeks  $(42 \pm 14 \text{ days})$  after the surgery date.

# 9.1.4 Follow-up visits at 6 weeks (42 $\pm$ 14 days)

- 1. Query subject regarding any changes in general health and the use of concomitant medications/therapies.
- If any adverse device effects or device deficiencies are observed or reported, they must be recorded as instructed in Section 12 - Adverse Events and Device Deficiencies.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 64 of 167 |

- 3. Verify with the subject if any revision has occurred since the last visit. If any revision is observed or reported, it must be recorded as instructed in Section 12 Adverse Events and Device Deficiencies.
- 4. Collect the 2011 KSS score objective measures (joint alignment, instability, motions & symptoms).
- 5. Have the subject complete the 2011 KSS score subject questions.
- 6. Have the subject complete the OKS patient-reported outcome measure
- 7. Have the subject complete the EQ-5D-5L patient-reported outcome measure.
- 8. Have the subject complete the FJS-12 patient-reported outcome measure.
- 9. Collect the standing weight bearing long leg (A/P) and standard lateral (non-weight bearing) radiographic images of the affected knee. Review the images to complete the appropriate eCRF for leg alignment and component alignment.
- 10. Instruct the subject on follow-up procedures, including returning to the site for the next follow-up visit in 6 months (185  $\pm$  14 days) after the surgery date.

### 9.1.5 6 months (185 $\pm$ 14 days) after surgery

- 1. Query subject regarding any changes in general health and the use of concomitant medications/therapies.
- 2. If any adverse device effects or device deficiencies are observed or reported, they must be recorded as instructed in Section 12 Adverse Events and Device Deficiencies.
- 3. Verify with the subject if any revision has occurred since the last visit. If any revision is observed or reported, it must be recorded as instructed in Section 12 Adverse Events and Device Deficiencies.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 65 of 167 |

- 4. Collect the 2011 KSS score objective measures (joint alignment, instability, motions & symptoms).
- 5. Have the subject complete the 2011 KSS score subject questions.
- 6. Have the subject complete the OKS patient-reported outcome measure
- 7. Have the subject complete the EQ-5D-5L patient-reported outcome measure.
- 8. Have the subject complete the FJS-12 patient-reported outcome measure.
- 9. Instruct the subject on follow-up procedures, including returning to the site for the next follow-up visit 12 months (365  $\pm$  30 days) after the surgery date.

## 9.1.6 Exit visit 12 months (365 $\pm$ 30 days) after surgery

- 1. Query subject regarding any changes in general health and the use of concomitant medications/therapies.
- 2. If any adverse device effects or device deficiencies are observed or reported, they must be recorded as instructed in Section 12 Adverse Events and Device Deficiencies.
- 3. Verify with the subject if any revision has occurred since the last visit. If any revision is observed or reported, it must be recorded as instructed in Section 12 Adverse Events and Device Deficiencies.
- 4. Collect standard A/P and lateral radiographic images of the affected knee. Review the images to complete the appropriate eCRF for standard radiographic evaluation (presence of radiolucent lines, osteolysis and implant migration).
- 5. In case a standing long leg X-ray is taken as a standard of care, please complete the respective leg alignment eCRF (optional).

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 66 of 167 |

- Collect the 2011 KSS score objective measures (joint alignment, instability, motions & symptoms).
- 7. Have the subject complete the 2011 KSS score subject questions.
- 8. Have the subject complete the OKS patient-reported outcome measure
- 9. Have the subject complete the EQ-5D-5L patient-reported outcome measure.
- 10. Have the subject complete the FJS-12 patient-reported outcome measure.
- 11. Complete Exit Visit eCRF.

### 9.1.7 Unscheduled Visits

Unscheduled examinations may be conducted at the discretion of the Investigator with all obtained information recorded in the source documents and on the appropriate eCRF. The subject should be scheduled to return for the next scheduled study visit within the acceptable time window.

### 9.1.8 Concomitant Medications and Therapies

Concomitant medications and concomitant therapies (e.g., physical therapy, pain medication) are recorded at any time from enrollment into the study through the subject's last study visit.

#### **Concomitant Medications**

### **Excluded Concomitant Medications**

There are no restrictions on concomitant medications for this study.

### Recording Concomitant Medications in the eCRF

Only medications related to the study treatment and medications used to treat an adverse event related to the study device and device deficiency will be recorded in

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 67 of 167 |

the eCRF. Reference the eCRF Completion Guidelines for how medications are recorded.

## **Concomitant Therapies**

Therapies Prohibited During the Study

There are no restrictions on concomitant therapies for this study.

### Recording Concomitant Therapies in the eCRF

Only therapies related to the study treatment and therapies used to treat an adverse event related to the study device and device deficiency will be recorded in the eCRF. Reference the eCRF Completion Guidelines for how therapies are recorded.

## 9.1.9 Discontinued Subjects

Discontinued subjects are those who voluntarily discontinue participation, who are withdrawn for reasons of safety or use of prohibited concomitant medications/therapies, who are lost to follow-up, refer to Section 7.8 for further details. Where possible, the next scheduled study visit should be completed for all subjects who discontinue the study early. Where consent is withdrawn, the date and any reason given for discontinuation should be captured, at a minimum (see Section 7.8.3).

Finally, if appropriate, the Investigator will also advise the subject of subsequent therapy and/or procedures necessary for their medical condition.

#### 9.1.10 Subject Pregnancy

Women of child-bearing potential are not excluded from the study. However, if a woman becomes pregnant during the study, S+N must be contacted immediately

| <b>Clinical Protocol</b> | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 68 of 167 |

once the investigator is made aware of the pregnancy. All study procedures that are contraindicated during pregnancy and/or lactation (e.g., x-rays) will not be required. A decision will be made regarding the continuation in the study of the pregnant woman. Pregnancy is not an adverse event; however, complications related to the pregnancy may be reportable as determined on a case-by-case basis. Pregnancy-related information will be collected until the end of the pregnancy.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 69 of 167 |

#### 9.2 STUDY METHODS AND MEASUREMENTS

## 9.2.1 Leg alignment

The leg alignment should be measured from an antero-posterior (A/P) view standing weight bearing full leg ('long leg') x-ray. The following axes shall be identified:

- Mechanical Axis of the femur: Axis from the center of the femoral head to the center of the distal femur.
- Mechanical Axis of the tibia: Axis from the center of the proximal to the center of the distal tibia.

The angular deviation from the neutral position (180°) shall be measured as shown as "E" in Figure 9.2-9-1. The angular deviation from the neutral position shall be recorded in the eCRF.

Figure 9.2-9-1 Leg alignment



Red: Mechanical Axis of Femur: Axis from the center of the femoral head to the center of the distal femur

Yellow: Mechanical Axis of Tibia: Axis from the center of the proximal to the center of the distal center of the tibia.

Blue: Neutral position axis (180°).

E: Deviation angle from the neutral position.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep<br>2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 70 of 167 |

### Pre-Operative Leg alignment

The pre-operative leg alignment evaluated from a standing weight bearing long leg standing A/P shall be recorded.

## Target Leg alignment (Surgical Plan)

The operative plan for leg alignment as entered in CORI shall be recorded in the eCRF for each subject. The planned leg alignment serves as the target for post-operative leg alignment. This may not be a neutral position.

## Pre- & Post-Cementation Leg alignment (for CORI UKA only)

The pre-cementation leg alignment shall be recorded with the use of CORI (manual screenshot to be taken) with the trials implant is placed.

Once the final implant has been cemented the post-cementation leg alignment shall be recorded with CORI (manual screenshot to be taken).

## Post-Operative Leg alignment

The leg alignment shall be assessed post-operatively and 6 weeks after surgery on standing weight bearing long leg A/P X-ray and lateral X-ray. Optionally, leg alignment can be assessed optionally at 12 months, in case a standing weight bearing long leg A/P X-ray is taken at 12 months.

Post-operative leg alignment is achieved when the deviation from the subject specific target does not exceed ±3 degrees.

All leg alignment measures will be added to the eCRF.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 71 of 167 |

## 9.2.2 Component Alignment

Component alignment will be assessed on long leg standing A/P X-rays and standard non-weight bearing lateral X-rays taken 6 weeks after surgery (or at discharge). The following angles will be evaluated on the X-rays and recorded in the eCRF:

#### A/P View

- Femoral A/P Angle: From the A/P radiograph, the femoral flexion angle is to be obtained using standard radiographic tools. Femoral flexion angle is defined as the angle formed between a line across the base of the femoral condyles and a line that is centered along the femoral canal
- Tibial A/P Angle: From the A/P radiograph, the tibial angle denotes the angle formed on the medial side of the knee from intersecting lines parallel to the tibial base plate and a line drawn parallel to the tibial canal (Figure 9.2-9-2).
- Total Valgus Angle: Is the sum of the femoral flexion angle and the tibial angle.

#### Lateral View

 Femoral Flexion Angle: The lateral view femoral flexion angle is obtained from the intersection of a line from the center of the femoral implant to the top of the femur with a

Figure 9.2.2-9-2 A/P View



A: Femoral A/P Angle B: Tibial A/P Angle A+B: Total Valgus Angle

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 72 of 167 |

line through the femoral canal. The angle is measured on the proximal side of the intersection

 Tibial Lateral Angle: The lateral view tibial angle is the angle obtained from the intersection of a line drawn parallel to the bottom of the tibial base insert and a line through the center of the tibial base and the tibial canal.

Figure 9.2.2-9-3 Lateral View



X: Femoral Flexion Angle Y: Tibial Lateral Angle

## 9.2.3 Standard Radiographic Evaluation

Standard radiographic evaluation on antero-posterior (A/P) and lateral views shall be performed 12 months after surgery in order to identify any radiographic observations such as radiolucent lines around the implant components. The presence of radiolucent lines, osteolysis & implant migration shall be recorded in the eCRF.

# 9.2.4 2011 Knee Society Score (2011 KSS)

The 2011 Knee Society Score will be collected at the pre-operative visit and 6 weeks, 6- and 12-months after surgery.

The 2011 KSS is a validated tool that combines an objective physician-derived component with a subjective subject-derived component [45, 46]. The 2011 KSS consists of 34 questions and provides sub-scores across 4 dimensions as shown in Table 9.2.4-9-2.

Table 9.2.4-9-2 2011 Knee Society Score

| # | Sub-Score | # Questions | Completion by |
|---|----------------------|-------------|---------------|
| 1 | Objective Knee Score | 4 | Surgeon |
| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 73 of 167 |

| 2 | Symptoms | 3 | Subject |
|---|-----------------------|----|---------|
| 2 | Subject Satisfaction | 5 | Subject |
| _ | Score | | Jubject |
| 3 | Subject Expectation | 3 | Subject |
| 4 | Functional Knee Score | 19 | Subject |

The Objective Knee Score is rated by the clinician and assesses a range of clinical outcomes: UKA alignment, stability, ROM and symptoms. The Subject Satisfaction Score assesses the satisfaction with 5 daily activities (sitting, lying in bed, getting out of bed, light household duties, and leisure activities). The Subject Expectation Score evaluates the subject's expectations prior to surgery. The post-operative questions differ from the pre-operative questions and ask if the subject's pre-operative expectations have been met. As the pre- and post-operative scores are based on different questions, they cannot be directly compared. The Functional Knee Score is derived from assessments of walking and standing, standard activities, advanced activities, and discretionary activities.

A paper questionnaire will be provided by the Sponsor to be completed by the subject. Responses for the 2011 KSS will then be recorded in the eCRF.

# 9.2.5 Oxford Knee Score (OKS)

The OKS will be collected at the pre-operative visit and 6 weeks, 6- and 12-months after surgery.

The OKS is a Patient Reported Outcome questionnaire that was developed to specifically assess the patient's perspective of outcome following Total Knee Arthroplasty. The OKS is a patient self-completion PRO containing 12 equally weighted questions on activities of daily living. The OKS has been developed and validated specifically to assess perceived function and pain answered on a Likert scale after TKA [47, 48]. Responses to each question ranges from 0-4 with a range of a

| <b>Clinical Protocol</b> | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 74 of 167 |

possible overall score from 0-48. A score of 0 is the worst possible outcome while a score of 48 is the best possible outcome. The benefit to this questionnaire is that it is short, practical, reliable, valid and sensitive to clinically important changes over time.

A paper questionnaire will be provided by the Sponsor to be completed by the subject. Responses for the OKS will then be recorded in the eCRF.

# 9.2.6 Forgotten Joint Score (FJS-12)

The FJS-12will be collected at 6 weeks, 6- and 12-months after surgery. A paper questionnaire will be provided by the Sponsor to be completed by the subject.

The FJS-12 comprises measures for the assessment of joint-specific patient reported outcomes. This questionnaire focuses on the study subject's awareness of the partially or fully replaced knee joint in everyday life. Joint awareness can be simply defined as any unintended perception of a joint [49]. Subjects are asked to rate their awareness of their knee arthroplasty in 12 questions with a five point Likert response format: "Never", "almost never", "seldom", "sometimes" and "mostly". The item scores are summed and linearly transformed in a 0 to 100 scale with a high value reflecting the ability of the subject to forget about the replaced knee joint during the activities of daily living.

A paper questionnaire will be provided by the Sponsor to be completed by the subject. Responses for the FJS-12 will then be recorded in the eCRF.

# 9.2.7 CORI System Time & Cutting Time

CORI System Time and the Cutting Time of the robotic drill shall be collected postoperatively.

CORI Case Report, including case logs, will be extracted from CORI via USB and time data will be extracted for CORI System Time and the Cutting Time

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 75 of 167 |

In the case logs, the following time stamps will be recorded in the log file of the CORI Case Report:

- 1. State-Machine transition: [ Adjust Camera ] --> [ Checkpoint Definition ]
- 2. State-Machine transition: [ Checkpoint Verification ] --> [ Remove Bone ]
- 3. State-Machine transition: [ Remove Bone ] --> [ Baseline Stress ROM Collection ]

# **CORI System Time**

CORI System starts with the checkpoint definition until the bone is removed. This is calculated by the time difference between #3 and #1.

# **Cutting Time**

The Cutting Time of the robotic drill is the time from the start until the end of bone removal and is calculated by the time difference between #3 and #2.

The CORI System time and the cutting time of the robotic drill will not be recorded in the eCRF as they will be extracted directly from the CORI Case Report.

# 9.3 HEALTH ECONOMICS/QUALITY OF LIFE

# 9.3.1 EQ-5D-5L

The EQ-5D-5L questionnaire will be collected at the pre-operative visit as well as 6 weeks, 6- and 12-months after surgery. A paper questionnaire will be provided by the Sponsor to be completed by the subject.

The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 76 of 167 |

The descriptive system is used to describe the subject's health state and consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels to choose the most appropriate answer: no problems, slight problems, moderate problems, severe problems, and extreme problems. The subject is asked to indicate his/her health state by marking the most appropriate statement in each of the five areas [50].

The EQ VAS records the subject's self-rated health on a vertical visual analogue scale. The endpoints on the scale are labelled "The best health you can imagine" and "The worst health you can imagine". The VAS can be used as a quantitative measure of health outcome as judged by the individual respondents.

A paper questionnaire will be provided by the Sponsor to be completed by the subject. Responses for the EQ-5D-5L Score will then be recorded in the eCRF.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 77 of 167 |

# **10 STATISTICAL DESIGN**

A Statistical Analysis Plan (SAP) will be written and finalized prior to database lock. The following is a brief description of the analyses to be described in this plan.

## 10.1 GENERAL

S+N's Global Biostatistics group will conduct the statistical analysis for this study. Unless otherwise stated, all significance tests and hypothesis testing will be two-sided, performed at the 5% significance level. Resulting p-values will be quoted and 95% two-sided confidence intervals will be generated where appropriate. Where data summaries are specified, categorical and ordinal variables will be summarized with frequencies and percentages. Continuous variables will be summarized with the following summary statistics: the number of observations, mean, median, standard deviation, minimum and maximum values.

All statistical comparisons of data will describe the test statistic used as well as its distributional assumptions. For continuous variables, in an event of marked deviation from normality assumption, a commensurate non-parametric test would be used as an alternative thereby eliminating the possibility of violation of normality assumptions. All analyses will be performed using SAS version 9.3 (or a later version).

### **10.2 Analysis Populations**

The following are the analysis populations:

- Enrolled Population: This is defined as subjects enrolled and/or randomized to either CORI or Conventional manual instrumentation groups. A total of 140 patients will be competitively enrolled and or/randomized in the study across all the sites including the sites in China.
- Safety Population (SAF): This is defined as all subjects who were treated for UKA (include non-randomized subjects in China as CORI is a pre-market

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 78 of 167 |

product in China) with the use of CORI or conventional manual instrumentation.

- Intent-to-Treat Population (ITT): The ITT population is a subset of the randomized population which is defined as subjects randomized to either CORI or conventional manual instrumentation groups who have at least one post-operative assessment on any of the effectiveness endpoints or health-related quality of life (HRQoL) endpoints. Data summarized on the ITT population will be based on the intervention the subject was randomized to receive which may be different from the intervention the subject actually received.
- Per-Protocol Population (PP): The PP population is a subset of subjects in the FAS population who do not have major protocol deviations and who satisfied all enrollment eligibility criteria. Major protocol deviations will include but not only restricted to subjects enrolled who do not satisfy the study entry eligibility criteria. All other criteria that will be categorized as major deviations will be formally classified on a case-by-case basis prior to the final study database lock.

#### 10.3 BASELINE DATA

All observations available prior to the operative date will be defined as baseline (or preoperative) data. All demographic and pre-operative characteristics data will be summarized at baseline. All demographic and baseline characteristics will be summarized using the enrolled SAF, ITT and PP analysis populations.

### 10.4 EFFECTIVENESS ANALYSIS

# 10.4.1 Analysis of Primary Endpoint

Leg alignment

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 79 of 167 |

The primary endpoint, the proportion of knees achieving post-operative leg alignment, defined as  $\pm 3^{\circ}$  from the target (pre-operative planned leg alignment) assessed at the 6 weeks study visit in CORI UKA ( $\Pi_1$ ) and conventional manual instrumentation UKA ( $\Pi_0$ ) groups.

The hypotheses are as follows:

- $H_0(\text{null})$ :  $\Pi_1 <= \Pi_0 \text{ versus}$
- $H_1$  (alternate):  $\Pi_1 > \Pi_0$ .

The proportions as described above will be supported with the use of a two-sided 95% confidence intervals (CI), estimated using exact binomial methods.

Superiority of  $\Pi_1$  over  $\Pi_0$  will be inferred if and only if the lower limit of the 95% CI for  $\Pi_1$  is greater than the upper limit of the 95% CI for  $\Pi_0$ .

As supportive analysis on the primary endpoint, the difference between the target and actual leg alignment achieved postoperatively will be summarized for each group (i.e. CORI UKA and the Conventional manual instrumentation UKA) using summary statistics for continuous variables. Ninety-five (95) % CIs based on the Student's t-distribution will be calculated for the means.

The primary endpoint and the supportive analysis will be summarized using the FAS analysis population as primary and then PP analysis population for sensitivity.

For missing primary endpoint data, the Missing Value Treated as Failure (MVTF) missing value imputation method will be used. This is considered a conservative imputation method as all missing data on the primary endpoint will be considered as a failure, i.e. not attaining the pre-specified target alignment. More specific details of this imputation method will be included in the SAP.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 80 of 167 |

# 10.4.2 Analysis of Secondary Endpoints

# Component Alignment

Femoral components (internal rotation, valgus and anterior tilt) and tibial components (internal rotation, valgus, and posterior slope) will be summarized using descriptive summary characteristics for continuous variables. These would additionally be stratified by surgical technique within each group (CORI Navigational versus Conventional Manual Instrumentation).

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 81 of 167 |

# Standard Radiographic Assessment

The presence of radiographic observations: implant loosening, implant migration, and osteolysis and other pertinent radiographic findings will be summarized as counts (n) and percentages (%) by visit. These would additionally be stratified by surgical technique within each group (CORI Navigational versus Conventional Manual Instrumentation).

Radiolucent lines (mm) by zone and visit will be summarized using descriptive statistics for continuous variables. These would additionally be stratified by surgical technique within each group (CORI Navigational versus Conventional Manual Instrumentation).

# 2011 Knee Society Score (KSS)

The 2011 KSS objective, function and satisfaction scores will be summarized at the pre-operative and postoperative visits using continuous summary characteristics. For each of these 3 KSS scores, independent repeated measures Analysis of Covariance (ANCOVA) models (to account for the correlation between subjects with bilateral knees) will be used to model the change from preoperative to postoperative KSS scores as the dependent variable. As a minimum, each model will contain a group (pre-operative and postoperative) and the investigational site as a fixed term with a repeated specification for the knee. Pre-operative prognostic and demographic variables not only restricted to age, BMI and sex, but that can also be ascertained to have an impact on the KSS scores will be introduced as covariates in the final model. These covariates will be added to the model using a stepwise approach and a covariate is retained in the final model if and only if its associated p-value ≤ 0.1. Model based means (adjusted means or Least Square Means, LSMeans) and corresponding standard errors associated with each change from preoperative to postoperative KSS score will be presented by group. Model based

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 82 of 167 |

differences (and corresponding standard errors) between the CORI Navigational and Conventional manual instrumentation groups and their corresponding 95% CIs will additionally be summarized. If the p-value associated with the group term in the model is significant (i.e. p < 0.05), then the 95% CIs corresponding to the model based differences between the CORI Navigational and Conventional manual instrumentation groups will additionally be presented.

The 2011 KSS subject expectation score will be summarized at the pre-operative and postoperative follow-up visits using descriptive characteristics for continuous variables.

## Oxford Knee Score (OKS)

The OKS (0-48) will be summarized at the preoperative and postoperative visits using continuous summary characteristics. Change from preoperative to postoperative visits will also be summarized. The repeated measures ANCOVA model to account for the correlation between subjects in case of bilateral knees analogous to that specified for the 2011 KSS will be used.

# Forgotten Joint Score (FJS-12)

The transformed FJS-12 score (0-100) will be summarized at the postoperative visits using continuous summary characteristics. Change from preoperative to postoperative visits will also be summarized. The repeated measures ANCOVA model to account for the correlation between subjects in case of bilateral knees analogous to that specified for the 2011 KSS will be used.

## EQ-5D-5L Score

The HRQoL Index score and VAS score will be summarized using summary statistics for continuous variables pre-operatively and at all postoperative visits. Change from

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | |

preoperative to postoperative visits will also be summarized. In the case of bilateral knees, repeated measures ANCOVA models will account for correlation between subjects with bilateral knees each for the index score and VAS analogous to that specified for the 2011 KSS will be used.

The 2011 KSS, transformed FJS-12 and EQ-5D-5L scores will additionally be summarized by group (i.e. the CORI Navigational and Conventional manual instrumentation groups) and visit using descriptive statistics for continuous variables.

The Multiple Imputation (MI) missing value imputation method will be used as the imputation method for missing 2011 KSS, FJS-12, OKS, and EQ-5D-5L endpoints. Details of the MI method will be included in the SAP.

All secondary endpoints will be summarized using the FAS analysis population.

# 10.4.3 Analysis of Other Endpoint(s)

The analyses for other endpoints (will be summarized separately in the CORI Navigational and Conventional manual instrumentation groups).

Leg alignment pre- and post-cementation (CORI UKA only)

Leg alignment is classified as normal, varus deformity and valgus deformity. Shift tables to summarize the changes from pre- to post-cementation will be created.

# **CORI System Time & Cutting Time**

CORI System and cutting times will be summarized using summary statistics for continuous variables. The average operating and cutting times summarized using summary statistics for continuous variables. Additionally, 95% CIs based on the t-statistic will be presented.

## 

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep<br>2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | |

All other endpoints will be summarized using the FAS analysis population.

### 10.5 SAFETY ANALYSES

All safety analyses will be summarized separately for each of the groups (i.e. CORI Navigational and Conventional manual instrumentation groups) as follows:

- The number of adverse events will be reported by seriousness, relationship to study device and anticipation.
- The number of subjects experiencing adverse events will be summarised by seriousness, relationship to study device and anticipation.
- An overall AE summary table that will summarize as number (n) and percentages (%), the overall incidence according to subjects with at least one AE; subjects with at least one AE by worst severity (mild, moderate, or severe); subjects with at least one AE by worst outcome (resolved, ongoing/unresolved, or death); subjects with an AE that led to study discontinuation) and; subjects with at least one AE by worse relatedness to device. Other events such as SAEs, ADEs, SADEs or UADEs will also be similarly summarized using the number (n) and percentages (%).
- Incidence of device-related re-interventions that occur on-study will be summarized as number (n) and percentages as well as by type.
- A listing of device deficiencies that occur on-study will be provided.
- Knee implant revision rate will be summarized as proportions with 95% CIs estimated using exact binomial methods.

All safety endpoints will be summarized using the SAF analysis population.

## **10.6 INTERIM ANALYSES**

A first interim analysis is planned for after completion of the 6 weeks visit in order to support the China NMPA registration. More specific details on the interim analyses will be included in the SAP.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 85 of 167 |

# 11 SAMPLE SIZE JUSTIFICATION

Parratte et al.[51] looked at the effects of postoperative mechanical axis alignment on the survival of TKAs. They found that of the 398 TKAs reviewed in the paper there were 292 (73.4%) which post-operatively were defined as mechanically aligned (i.e. with a mechanical axis of  $0^{\circ} \pm 3^{\circ}$ ).

This study is designed to demonstrate superiority in the proportion of knees achieving post-operative leg alignment in the CORI Navigational group over the Conventional manual instrumentation group.

The proportion of mechanically aligned TKAs using NAVIO from a recent analysis was estimated to be 92.1% [52]. This proportion is expected to be equivalent if NAVIO was used to determine the proportion of mechanically aligned UKAs. Using these assumptions, enrollment of 63 UKAs per group will provide 80% power to show that the lower limit of the two-sided 95% confidence interval for the proportion of mechanically aligned UKAs is greater than that obtained from literature. To account for up to a 10% attrition rate in knees enrolled, 70 knees in each group (140 knees combined) will be enrolled into the randomized stage of the study. A minimum of an additional 5 subjects who will be treated with CORI directly to fulfil the learning needs of the surgeons will be enrolled at the pre-randomized study stage, thus leading to a minimum total study enrollment of 145 subjects.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep<br>2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in | |
| unicondylar knee arthroplasty (UKA) Procedure | 1 age: 00 of 107 |

# 12 ADVERSE EVENTS AND DEVICE DEFICIENCIES

# **12.1 DEFINITIONS**

The categories of adverse events are shown in Table 12.1-12-1. The definitions for each of these categories are given in the subsequent sections.

Table 12.1-12-1 Categories of Adverse Event

| | NOT DEVICE-<br>RELATED | DEVICE- OR PROC | EDURE-RELATED |
|---|---|---|---|
| NON-<br>SERIOUS | Adverse Event (AE) | Adverse Device Effect (ADE) | |
| | CERTOLIC ADVERGE | Serious Adverse<br>(SADE) (se | |
| SERIOUS | SERIOUS ADVERSE EVENT (SAE) | ANTICIPATED ANTICIPATED SERIOUS ADVERSE DEVICE EFFECT | UNANTICIPATED UNANTICIPATED SERIOUS ADVERSE DEVICE EFFECT |
| | | (ASADE) | (USADE) |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 87 of 167 |

#### 12.1.1 Adverse Event

An <u>Adverse Event (AE)</u> is any untoward medical occurrence, unintended disease or injury or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device and whether anticipated or unanticipated.

- Note 1: This definition includes events related to the investigational medical device or the comparator.
- Note 2: This definition includes events related to the procedures involved.
- Note 3: For users or other persons, this definition is restricted to events related to the use of investigational medical devices.

AE is used both to refer to AE which do not meet the definitions of Adverse Device Effects or Serious Adverse Events and as an umbrella term referring to adverse events of all classifications.

An AE can be any unfavorable and unintended sign (for example, an abnormal laboratory finding), symptom, or disease. For reporting purposes, emphasis is placed first and foremost on whether or not the event constitutes an <u>untoward medical occurrence</u>.

## 12.1.2 Adverse Device Effect

An <u>Adverse Device Effect (ADE)</u> is an adverse event related to the use of an investigational medical device.

- Note 1: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation or operation, or any malfunction of the investigational medical device.
- Note 2: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device.
- Note 3: This includes "comparator" if the comparator is a medical device.

**Not Related** - An AE is considered to be not related to the use of an IP or the procedure when the effect is DEFINITELY UNRELATED to have any relationship to the use of the IP or the procedure.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 88 of 167 |

**Related** – An AE is considered to be related to the use of an IP or the procedure when there is a POSSIBLE, or DEFINITE relationship between the AE and the use of the IP or the procedure.

An ADE is further categorized depending on whether the criteria in section 12.1.3 and 12.1.4 are met.

# **12.1.3** Related Serious Adverse Events and Serious Adverse Device Effects

An AE or ADE is considered a **Serious** Adverse Event (SAE) or **Serious** Adverse Device Effects (SADE) if, it led to any of the following:

- a) Death,
- b) Serious deterioration in the health of the subject, users or other persons as defined by one or more of the following:
  - 1) Alife-threatening illness or injury, or
  - 2) A permanent impairment of a body structure or a body function including chronic diseases, or
  - 3) In-patient or prolonged hospitalization, or
  - 4) -Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function,
- c) Fetal distress, fetal death or a congenital abnormality or birth defect including physical or mental impairment

Note 1: Planned hospitalization for a pre-existing condition, or a procedure required by the study protocol, without serious deterioration in health, is not considered a serious adverse event.

# 12.1.4 Anticipated/Unanticipated Serious Adverse Device Effect

An Unanticipated Serious Adverse Device Effect (USADE) is a serious ADE which by its nature, incidence, severity or outcome has not been identified in the current version of the risk assessment.

Note 1: Anticipated serious adverse device effect (ASADE) is an effect which by its nature, incidence, severity or outcome has been identified in the risk assessment.

A list of potential ASADE for CORI is provided in Table 12.1.4-12-2. Please also refer to Section 4.4.5 Potential Adverse Effects.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep<br>2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 89 of 167 |

**Table 12.1.4-12-2 Potential Anticipated Serious Adverse Device Effects (ASADE)** 

| # | Potential Harm | Description |
|---|---|---|
| 1 | Allergic Reaction<br>to Materials | Hypersensitivity caused by exposure to material constituents of the product that leads to local inflammatory reaction and tissue damage. Contact with an allergen may cause swelling and redness of the skin in minor cases. A severe anaphylactic reaction may occur. |
| 2 | Bone Fracture | Any break or fracture to any bone. (Applicable to displaced and non-displaced fractures) The bone break could be reduced (set) and immobilized during the same surgery during which it occurred if it is detected. If the fracture occurs after the surgery, additional medical attention would be required. Subsequent healing returns normal body function for the subject. |
| 3 | Burn | 3 <sup>rd</sup> degree burn extending through the dermis which requires excision. 4 <sup>th</sup> degree burn extending into the subcutaneous tissue, muscle and bone with eschar formation. Burns may be caused by thermal or chemical burns. |
| 4 | Cardiac<br>Arrhythmia -<br>symptomatic | Variation from the normal heart rhythm symptomatic. |
| 5 | Cement Leakage | Cement can end up in an unintended location in the joint. Cement leakage may cause early wear of poly or pain to the subject and may require revision surgery. |
| 6 | Unstable knee<br>joint | The implant components are placed in such a way that there is too much laxity in the ligaments. The subject experiences instability throughout the range of motion, There is an increased risk of early loosening/ wear of the implant. This may impact the stability and wear of implant components. Implants loosening could lead to early revision surgery. |
| 7 | Restricted Range<br>of Motion | The implants are placed in such a way that excessive forces are placed on the ligaments (ACL, PCL, MCL, and LCL). This leads to an unintended reduction in the range of motion or progression of disease in a non- operative compartment. This may be serious, if the subject's range of motion has been worsened compared to the range of motion prior to surgery, or it has been restored suboptimally. |

#### 

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 90 of 167 |

| # | Potential Harm | Description |
|---|---|---|
| # | Fotential narm | Description |
| | Infection | Invasion and multiplication of microorganisms in body tissues, especially microorganisms causing local cellular injury due to competitive metabolism, toxins, intracellular replication, or antigen-antibody response. The infection may lead to a diseased state in the receiving host if the host has inadequate resistance and/or lacks immunity to overcome the invasion by the pathogen. |
| 8 | | Most typically, the resultant disease state can be treated through the use of antibiotics. When the pathogen is particularly virulent, or when the host has low resistance, the disease state may lead to a permanent impairment of some aspect of bodily function or, in extreme cases, to death. Infections caused by a transfer of body fluids during orthopedic surgery can in most cases be treated by a course of antibiotics. Severe infections that can occur by the transfer of body fluids during the procedure include HIV and hepatitis. |
| 9 | Delay | A delay in the operation time exceeding 60 minutes of intra-<br>operative case time. A wound being open longer would more likely<br>result in soft tissue edema, increased blood loss, muscle necrosis<br>as a result of extended tourniquet time and a higher chance of<br>infection. |
| 10 | Immature implant failure | Implant components wear before their intended service life resulting in early revision surgery. |
| 11 | Neurological<br>Injury | Damage to the nerve systems of the subject's leg. A neurological injury could result in temporary or permanent paralysis. |
| 12 | Physical Injury -<br>Serious | A physical injury that necessitates medical intervention. |
| 13 | Soft Tissue<br>Damage | Damage to ligaments or tendons leading to loss of stability in the knee joint. In severe cases of ligament damage, additional surgery may be required. |
| 14 | Surgeon Operates<br>on Wrong Part of<br>Anatomy | The clinical impacts of operating on the wrong subject anatomy relate to the resultant function of the skeletal element that was treated and the need to repeat treatment for the desired skeletal element. The impact on the subject may be additional surgery under full anesthesia. |
| 15 | Vascular Injury -<br>Main Low-<br>extremity vessels | Damage to the vascular systems of the subject's leg. In severe cases, dis-vascularization occurs that is, the subject loses blood flow to the leg when a clot forms in significant arteries of the leg. Additional surgery would be required to correct blood |

## 

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 91 of 167 |

| # | Potential Harm | Description |
|---|---|---|
| | | flow. If blood flow to the leg is not restored, the patient's leg may |
| | | need to be amputated. |

# 12.1.5 Guidance Regarding the Determination of Unanticipated Events:

During causality assessment activity, clinical judgement shall be used and the relevant documents, such as the Investigator's Brochure, the Clinical Protocol or the Risk Analysis Report shall be consulted, as all the foreseeable serious adverse events and the potential risks are listed and assessed there. The presence of confounding factors, such as concomitant medication/treatment, the natural history of the underlying disease, other concurrent illness or risk factors shall also be considered [MEDDEV 2.7/3 Rev 3 Sec 8].

# 12.1.6 Severity

The severity of every AE will be assessed by the PI or medically qualified site staff to whom the responsibility has been delegated and documented on the delegation of authority log. AE should be classified as mild, moderate, or severe, regardless of whether or not the AE are considered to be serious or non-serious. The classification should be based on the following definitions:

- **Mild** An event is mild if the subject is aware of, but can easily tolerate the sign or symptom.
- **Moderate** An event is moderate if the sign or symptom results in discomfort significant enough to cause interference with the subject's usual activities.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 92 of 167 |

**Severe** - An event is severe if the sign or symptom is incapacitating and results in the subject's inability to work or engage in their usual activities.

# **12.1.7** Device Deficiency

A Device Deficiency (DD) is an inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance. DD includes malfunctions, use errors and inadequate labeling.

Note 1: DD includes malfunctions, use errors and inadequacy in the information supplied by the manufacturer including labelling.

Note 2: This definition includes device deficiencies related to the investigational medical device or the comparator.

Device deficiencies that did not lead to an adverse event but could have led to a medical occurrence

- a) if either suitable action had not been taken,
- b) if intervention had not been made, or
- c) if circumstances had been less fortunate,

are considered Device Deficiencies with potential to cause SADE and shall be reported as specified in section 12.3.

## 12.2 AE CODING DICTIONARY

Coding for this study will be done per International Medical Device Regulators

Forum (IMDRF) AE Terminology Annex E – Clinical signs, symptoms, and conditions.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 93 of 167 |

# 12.3 REPORTING PROCEDURES

AE of any kind and DD will be recorded in the applicable CRF and source notes to include the date of occurrence, treatment and the details resolution. The Investigator will evaluate all AE for relationship to the device and procedure, seriousness, and severity (if applicable). DD will be evaluated for potential to cause SADE. The following timescales should be followed for the AE/DD information to be submitted/entered into the CRF and reported to the Sponsor or designee (see figure 12.2-1):

- ADE and DD without unreasonable delay
- SAE, SADE and DD with potential to cause SADE immediately (i.e. within 24 hours of the investigator being informed about the event)
- All other events according to usual timescales

In addition to inputting SAE and SADE information within 24 hours of being aware of the event, the investigator should email <u>Clinical.safety@Smith-nephew.com</u> to alert the safety representative of the events existence and to clarify details if necessary.

For ADE and DD, date of occurrence, and details of the product/procedure related to the event will be included and where applicable, pictures taken of the device. The deficient product should be retained for return to S+N unless it is contaminated (e.g., used dressings must not be retained). Updates to submitted information will be recorded in the CRF according to the timescales above.

All adverse events will be reviewed by a medically qualified person appointed by the Sponsor to determine which, if any, meet criteria for expedited reporting to the regulatory authorities.

The investigator will inform the regulatory agency and IRB/IEC of adverse events as per the requirements listed below: -

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 94 of 167 |

The investigator should inform the regulatory agency and IRB/IEC of adverse events as per the requirements of each site. The detailed information is described in Safety Monitoring Plan.

All other events will be reported on a periodic/annual basis.

Depending on the nature of the adverse event, S+N may request copies of the subject's medical records, Imaging, Operative notes, as well as results of any relevant laboratory tests performed or other documentation related to the AE. If the subject was hospitalized, a copy of the discharge summary may be requested by S+N and should be forwarded as soon as it becomes available. In certain cases, S+N also may request a letter from the Investigator that summarizes the events related to the case. Refer to the ISF Sponsor Contact Information Sheet to report SAE, unanticipated SADE, anticipated SADE, and DD.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 95 of 167 |

Figure 12.3-12-1 Evaluation and Reporting of AE



| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 96 of 167 |

Figure 12.3-12-2 Evaluation and Reporting of DD



## 12.4 Unblinding of Investigational Product

Not applicable.

# 12.5 FOLLOW-UP OF SUBJECTS WITH ADVERSE EVENTS

For subjects who are experiencing ongoing unresolved AE at the time of their study completion or early discontinuation from the study, it is recommended that the Investigator schedule an appropriate follow-up visit to determine the outcome of the event.

Any additional data must be documented and available to the Sponsor who will determine whether the data need to be documented in the eCRF or the Clinical Study Report.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 97 of 167 |

# 12.5.1 Ongoing Adverse Events at Study Discontinuation

Adverse events which are **related** to a study procedure or S+N IP and are ongoing at the end of subject's participation: The event should be followed until it is either resolved or until the event has become chronic and is not expected to further improve based on Investigator's review of the event.

Adverse events that are **not related** to a study procedure or S+N IP and are ongoing at the end of subject's participation should be followed for 30 days after discontinuation or if the AE is resolved, whichever is sooner.

At the time of data analysis (e.g., interim or final), an evaluation of ongoing events should take place and be listed as ongoing in the safety table.

### 13 INVESTIGATOR OBLIGATIONS

The Principal Investigator will comply with the commitments outlined in the in the Statement of Investigator, provided by the Sponsor, and with Good Clinical Practice (GCP), and all applicable regulatory requirements as outlined in Appendix-Principal Investigator Obligations as well as all applicable local laws and regulations.

In addition, the PI will ensure that the Financial Disclosure Statements will be completed by the PI and the Sub-Investigator upon entry into the study and any changes that affect their financial disclosure status occur during the course of the study and up to one year after study completion.

# 14 SPONSOR AND MONITOR RESPONSIBILITIES

The Sponsor will designate a monitor to conduct the appropriate site visits at the appropriate intervals. The clinical investigation will be monitored to ensure that: the rights and wellbeing of the subjects are protected; the reported data are accurate, complete, and verifiable from the source documents; and the study is conducted in

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 98 of 167 |

compliance with the currently approved protocol and amendment(s), if applicable, with GCP regulations, and with applicable regulatory requirements.

Detailed monitoring requirements will be documented in the Clinical Monitoring Plan for this study.

### 14.1 CONTRACT RESEARCH ORGANIZATION

The Sponsor has engaged Contract Research Organization (CRO) to assist in conducting this study. When appropriate, the CRO is referred to in study documents as "Sponsor's agent."

# 14.2 SITE QUALIFICATION VISIT

A site qualification visit may be performed by the Sponsor prior to the execution of a clinical agreement to ensure that all Investigators have the appropriate training, staff, facilities, and resources to adequately conduct the study.

## 14.3 SITE INITIATION VISIT

A site initiation visit to provide training on the specifics of the study, site obligations and expectations of study conduct will be performed by the Sponsor or qualified person designated by the Sponsor following the execution of the Clinical Trial Agreement (CTA) and documented IRB/IEC approval.

## 14.4 Interim Monitoring Visit

Regular interim monitoring visits will be performed by the Sponsor or qualified person designated by the Sponsor.

#### 14.5 Sponsor Audits and Regulatory Inspection

Quality Assurance auditors, whether an employee of the Sponsor or its designee, may evaluate study conduct at the study sites. These parties must have access to

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 99 of 167 |

any and all study reports and source documentation, regardless of location and format.

### 14.6 CLOSE-OUT VISIT

A study close-out visit will be performed by the Sponsor or designee to retrieve and account for all remaining clinical data and to resolve outstanding queries. During study close-out, the monitor will review investigator files to ensure required documents and records are on file, confirm the disposition of any other ancillary items used for the study, and review regulatory requirements regarding records retention and IRB or IEC reporting requirements. When no subjects have been included, a remote close-out visit may be conducted.

## 15 PROTOCOL DEVIATIONS

An Investigator must not make any changes or deviate from this protocol, except to protect the life and physical well-being of a subject in an emergency. Protocol deviations reported by the Investigator or discovered during monitoring visits will be compiled in a Protocol / GCP Deviation Log (TMP-CD-31-02 Protocol/GCP Deviation Log). Significant and/or recurrent protocol/GCP deviations will be documented on a protocol deviation form (TMP-CD-31-01 Protocol/GCP Deviation) including identified root cause and, as necessary, appropriate corrective and preventive actions will be put in place and and signed off by the study personnel.

# 16 PROTOCOL AMENDMENTS

Amendments should be made only in necessary cases once the study has started. Protocol amendments must be approved by the protocol signatories prior to submission to the IRB or IEC. Protocol amendments need to be approved by the IRB or IEC, according to the applicable requirements prior to implementation at the site.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 100 of 167 |

## 17 CONFIDENTIALITY OF THE STUDY

The confidentiality of this study and associated documents is governed by the terms of the Clinical Trial Agreement (CTA).

## 18 STATEMENTS OF COMPLIANCE

This clinical study will be performed in compliance with the ethical principles of the Declaration of Helsinki; and ISO 14155: Clinical investigation of medical devices – Good Clinical Practice.

This clinical study will not commence until the required approval/favorable opinion from the IRB/IEC or regulatory authority has been obtained. Any additional requirements imposed by the IRB/IEC or regulatory authority will be followed.

Public/Products Liability Insurance has been purchased by Smith & Nephew plc. Worldwide and incorporates coverage for personal injury in respect of clinical studies. The Sponsor agrees to operate in good faith and in accordance with the local guidelines regarding compensation for injury resulting from participation in an industry-sponsored clinical trial.

#### 19 END OF STUDY

The end of this study is defined by the last follow-up visit that occurs in the whole study population. Due to defined visit windows, the last follow-up visit must not necessarily be of the last subject treated.

Should circumstances arise which require the termination of the entire study prior to its planned completion (e.g., safety concerns) or circumstances arise which mean the end of the participation of an individual site (e.g., departure of Investigator, non-compliance), then this will be undertaken according to the SOPs of the Sponsor. The requirement for subject follow up in these instances will be considered as part

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 101 of 167 |

of these processes. The sponsor may decide to discontinue a specific study site under the following conditions:

- Non-compliance to GCP or study protocol
- Failure to enroll in subjects
- Unsafe or unethical practices

# 20 PUBLICATION POLICY

# 20.1 Publication of Study Data

The preparation and submission for publication of manuscripts containing the study results shall be in accordance with a process determined by the Clinical Trial Agreements between the study Sponsor and participating institutions. The publication or presentation of any study results shall comply with all applicable privacy laws.

## 20.2 DATA SHARING

Smith+Nephew is committed to upholding the highest ethical and legal standards involved in conducting clinical trials. Smith & Nephew, therefore, supports the data sharing requirements of The International Committee of Medical Journal Editors (ICMJE) published on the 6th June 2017. In accordance, Smith+Nephew will consider requests to share individual (de-identified) participant data that underlie the results of any interventional clinical trial, as presented from the 1st July 2018 within an ICMJE associated journal. Requests made by researchers who provide a methodologically sound proposal will be considered. Requests may include data that underlie results presented in text, tables, figures, and appendices, together with data dictionaries. The availability of these data will begin nine months and end 36 months after article publication. Data supplied may only be used by the researcher(s) named in the approved research proposal for the purposes of achieving the aims of the analyses specified therein. All proposals should be

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 102 of 167 |

directed to <a href="mailto:datasharing.gcs@smith-nephew.com">datasharing.gcs@smith-nephew.com</a>. To gain access, data requestors will need to sign a data access agreement.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 103 of 167 |

## 21 REFERENCES

- 1. Ferreira de Meneses, S., F. Rannou, and D.J. Hunter, *Osteoarthritis guidelines:* Barriers to implementation and solutions. Ann Phys Rehabil Med, 2016. **59**(3): p. 170-173.
- 2. Cutolo, M., et al., *Commentary on recent therapeutic guidelines for osteoarthritis.* Semin Arthritis Rheum, 2015. **44**(6): p. 611-7.
- 3. Arora, S., A. Rafiq, and M. Jolly, *Management of rheumatoid arthritis: Review of current guidelines*. Journal of Arthroscopy and Joint Surgery, 2016. **3**(2): p. 45-50.
- 4. Saxby, D.J. and D.G. Lloyd, *Osteoarthritis year in review 2016: mechanics.* Osteoarthritis Cartilage, 2017. **25**(2): p. 190-198.
- 5. Xie, K., et al., The effect of varus knee deformities on the ankle alignment in patients with knee osteoarthritis. J Orthop Surg Res, 2019. **14**(1): p. 134.
- 6. Cross, M., et al., *The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study.* Ann Rheum Dis, 2014. **73**(7): p. 1323-30.
- 7. Karim, A.R., et al., *Osteonecrosis of the knee*. Annals of translational medicine, 2015. **3**(1).
- 8. Pape, D., et al., *Prevalence of spontaneous osteonecrosis of the medial femoral condyle in elderly patients.* Knee Surg Sports Traumatol Arthrosc, 2002. **10**(4): p. 233-40.
- 9. Parratte, S., et al., *Primary total knee arthroplasty in the management of epiphyseal fracture around the knee.* Orthop Traumatol Surg Res, 2011. **97**(6 Suppl): p. S87-94.
- 10. Tang, X.B., et al., A Meta-Analysis of Patellar Replacement in Total Knee Arthroplasty for Patients With Knee Osteoarthritis. J Arthroplasty, 2018. **33**(3): p. 960-967.
- 11. Winter, A.R., J.E. Collins, and J.N. Katz, *The likelihood of total knee arthroplasty following arthroscopic surgery for osteoarthritis: a systematic review.* BMC Musculoskelet Disord, 2017. **18**(1): p. 408.
- 12. Hofstede, S.N., et al., Mobile bearing vs fixed bearing prostheses for posterior cruciate retaining total knee arthroplasty for postoperative functional status in patients with osteoarthritis and rheumatoid arthritis. Cochrane Database Syst Rev, 2015(2): p. Cd003130.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 104 of 167 |

- 13. Evans, J.T., et al., How long does a knee replacement last? A systematic review and meta-analysis of case series and national registry reports with more than 15 years of follow-up. The Lancet, 2019. **393**(10172): p. 655-663.
- 14. Aujla, R.S. and C.N. Esler, *Total Knee Arthroplasty for Osteoarthritis in Patients Less Than Fifty-Five Years of Age: A Systematic Review.* J Arthroplasty, 2017. **32**(8): p. 2598-2603.e1.
- 15. Yoon, C., et al., Does unicompartmental knee arthroplasty have worse outcomes in spontaneous osteonecrosis of the knee than in medial compartment osteoarthritis? A systematic review and meta-analysis. Arch Orthop Trauma Surg, 2019. **139**(3): p. 393-403.
- 16. Yue, J., L. Zhang, and C. Yang, *The impact of patellofemoral arthritis on unicompartmental knee arthroplasty*. Acta Orthop Belg, 2015. **81**(4): p. 587-93.
- 17. Registry, N.J., *Types of primary knee replacements undertaken*, 2018: England, Wales, Northern Ireland.
- 18. (AOANJRR), A.O.A.N.J.R.R., *Hip, Knee & Shoulder Arthroplasty: 2019 Annual Report.* . Adelaide: AOA, 2019, 2019.
- 19. Camarda, L., et al., *Patient-specific instrumentation for total knee arthroplasty: a literature review.* Musculoskelet Surg, 2015. **99**(1): p. 11-8.
- 20. Confalonieri, N., et al., *Navigated "small implants" in knee reconstruction.* Knee Surg Sports Traumatol Arthrosc, 2016. **24**(11): p. 3507-3516.
- 21. Burnett, R.S. and R.L. Barrack, *Computer-assisted total knee arthroplasty is currently of no proven clinical benefit: a systematic review.* Clin Orthop Relat Res, 2013. **471**(1): p. 264-76.
- 22. van der List, J.P., et al., *Current state of computer navigation and robotics in unicompartmental and total knee arthroplasty: a systematic review with meta-analysis.* Knee Surg Sports Traumatol Arthrosc, 2016. **24**(11): p. 3482-3495.
- 23. Roche, M., L. Elson, and C. Anderson, *Dynamic soft tissue balancing in total knee arthroplasty*. Orthopedic Clinics of North America, 2014. **45**(2): p. 157-165.
- 24. Mayman, D., *Handheld navigation in total knee arthroplasty.* Orthop Clin North Am, 2014. **45**(2): p. 185-90.
- van der List, J.P., H. Chawla, and A.D. Pearle, *Robotic-Assisted Knee Arthroplasty: An Overview.* Am J Orthop (Belle Mead NJ), 2016. **45**(4): p. 202-11.

#### 

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 105 of 167 |

- 26. Clayton, A.W., et al., *Does the use of navigation in total knee arthroplasty affect outcomes?* J Knee Surg, 2014. **27**(3): p. 171-5.
- 27. Abdel, M.P., et al., Coronal alignment in total knee replacement: historical review, contemporary analysis, and future direction. Bone Joint J, 2014. **96-b**(7): p. 857-62.
- 28. Nair, R., G. Tripathy, and G.R. Deysine, *Computer navigation systems in unicompartmental knee arthroplasty: a systematic review.* Am J Orthop (Belle Mead NJ), 2014. **43**(6): p. 256-61.
- 29. Banerjee, S., et al., *Robotic-assisted knee arthroplasty*. Expert Review of Medical Devices, 2015. **12**(6): p. 727-735.
- 30. Nodzo, S.R., K.M. Carroll, and D.J. Mayman, *Disposable Navigation for Total Knee Arthroplasty*. Am J Orthop (Belle Mead NJ), 2016. **45**(4): p. 240-5.
- 31. Blakeney, W., et al., *Kinematic alignment in total knee arthroplasty better reproduces normal gait than mechanical alignment.* Knee Surg Sports Traumatol Arthrosc, 2019. **27**(5): p. 1410-1417.
- 32. Lonner, J.H. and V.M. Moretti, *The Evolution of Image-Free Robotic Assistance in Unicompartmental Knee Arthroplasty.* Am J Orthop (Belle Mead NJ), 2016. **45**(4): p. 249-54.
- 33. Khlopas, A., et al., *Robotic Arm-Assisted Total Knee Arthroplasty*. J Arthroplasty, 2018. **33**(7): p. 2002-2006.
- 34. Robinson, P.G., et al., A systematic review of robotic-assisted unicompartmental knee arthroplasty: prosthesis design and type should be reported. Bone Joint J, 2019. **101-b**(7): p. 838-847.
- 35. Jacofsky, D.J. and M. Allen, *Robotics in Arthroplasty: A Comprehensive Review.* J Arthroplasty, 2016. **31**(10): p. 2353-63.
- 36. Thein, R., et al., *Lateral Robotic Unicompartmental Knee Arthroplasty*. Sports Medicine and Arthroscopy Review, 2014. **22**(4): p. 223-228.
- 37. Roche, M., Robotic-assisted unicompartmental knee arthroplasty: the MAKO experience. Orthop Clin North Am, 2015. **46**(1): p. 125-31.
- 38. Batailler, C., et al., *Improved implant position and lower revision rate with robotic-assisted unicompartmental knee arthroplasty.* Knee surgery, sports traumatology, arthroscopy: official journal of the ESSKA, 2019. **27**(4): p. 1232-1240.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 106 of 167 |

- 39. Battenberg, A.K., N.A. Netravali, and J.H. Lonner, *A novel handheld robotic-assisted system for unicompartmental knee arthroplasty: surgical technique and early survivorship.* J Robot Surg, 2019.
- 40. Canetti, R., et al., Faster return to sport after robotic-assisted lateral unicompartmental knee arthroplasty: a comparative study. Archives of orthopaedic and trauma surgery, 2018. **138**(12): p. 1765-1771.
- 41. Gregori, A., F. Picard, and J. Lonner, *ACCURACY OF IMAGELESS ROBOTICALLY ASSISTED UNICONDYLAR KNEE ARTHROPLASTY.* Bone Joint J, 2016. **98**(SUPP 5): p. 33-33.
- 42. Herry, Y., et al., *Improved joint-line restitution in unicompartmental knee arthroplasty using a robotic-assisted surgical technique.* International Orthopaedics, 2017. **41**(11): p. 2265-2271.
- 43. Vega Parra, P.D., et al., Robotic-assisted unicompartmental knee replacement with navio surgical system: Outcome Evaluation using the Knee Injury Osteoarthritis Outcome Score. Revista Chilena de Ortopedia y Traumatologia, 2017. **58**(1): p. 7-12.
- 44. Sephton, B.M., et al., *Predictors of extended length of stay after unicompartmental knee arthroplasty.* Journal of Clinical Orthopaedics and Trauma, 2019.
- 45. Asif, S. and D.S. Choon, *Midterm results of cemented Press Fit Condylar Sigma total knee arthroplasty system.* J Orthop Surg (Hong Kong), 2005. **13**(3): p. 280-4.
- 46. Insall, J.N., et al., *Rationale of the Knee Society clinical rating system.* Clin Orthop Relat Res, 1989(248): p. 13-4.
- 47. Dawson, J., et al., *Questionnaire on the perceptions of patients about total knee replacement.* J Bone Joint Surg Br, 1998. **80**(1): p. 63-9.
- 48. Murray, D.W., et al., *The use of the Oxford hip and knee scores.* J Bone Joint Surg Br, 2007. **89**(8): p. 1010-4.
- 49. Behrend, H., et al., *The "forgotten joint" as the ultimate goal in joint arthroplasty:* validation of a new patient-reported outcome measure. J Arthroplasty, 2012. **27**(3): p. 430-436.e1.
- 50. Janssen, M.F., et al., *Measurement properties of the EQ-5D-5L compared to the EQ-5D-3L across eight patient groups: a multi-country study.* Qual Life Res, 2013. **22**(7): p. 1717-27.
- 51. Parratte, S., et al., Effect of postoperative mechanical axis alignment on the fifteenyear survival of modern, cemented total knee replacements. J Bone Joint Surg Am, 2010. **92**(12): p. 2143-9.

#### 

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 107 of 167 |

52. Nephew, S., Clinical Study Report 6-month Follow-up: "Clinical, Radiographic and Patient-reported Outcomes Associated with the Use of the NAVIO™ Robotic-assisted Surgical System in Total Knee Arthroplasty", 2019.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 108 of 167 |

## 22 APPENDICES

## 22.1 PROTOCOL AMENDMENT

# 22.1.1 General Purpose

The purpose of the protocol amendment is to meet the requirements of the Hongkong site during the EC approval session. The protocol amendment for version 2.1 is minor.

The purpose to have the 2nd protocol amendment into version 3.0-Master is to update the protocol from Template B into Template D and also update the information within the protocol.

The purpose of amending version 3.0 to version 4.0-Master is to expand the presurgery visit window from -28 to -90 days. South Korea has also been added as a location for where the study will be conducted and staged bilateral subjects can now be enrolled. Subject has one or more of the following arthroplasties that are not fully healed and well-functioning, as determined by the investigator: Contralateral primary TKA or UKA, however, the subject can only have one knee enrolled in this study.

. An additional exclusion was added to restrict the enrolment of subjects who currently enrolled in another study orthopaedic clinical trial study at least 1 year prior to screening. Some of the changes in this version are being made to maintain alignment with the changes required by the regulatory authorities in China.

# 22.1.2 Rationale

The rationale to 1<sup>st</sup> time updates the protocol is due to the protocol title inconsistency with other documents. Since the amendment is change that do not materially affect the study which is simply update the protocol title from "procedures" into "Procedure".

The rationale to 2<sup>nd</sup> time updates the protocol is due to the protocol template updated from version B to version D. And also, the information inside of the protocol need to be further updated.
| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 109 of 167 |

The rationale to 3<sup>rd</sup> time update is to allow more patient to enrol in the study and update the information based on ISO14155 2020 and to maintain alignment with the changes required by the regulatory authorities in China.

# 22.1.3 Effect on Study Status

Not applicable. The amendment in version 2.0, 2.1 and 3.0-Master was in effect and implemented prior to subject enrolment.

The amendment in Version 4.0-Master will not impact the status of study, however, patient enrolment may improve.

22.1.4 Details

1st Update from Version 2.0 to Version 2.1

| Section | Current Text | Revised Text |
|---|---|---|
| | Version 2.0 (04SEP2020) | Version 2.1 (14JAN2021) |
| | A Prospective, Multi-center, | A Prospective, Multi-center, |
| | Randomized Controlled Study to | Randomized Controlled Study to |
| | Evaluate the Safety and I | Evaluate the Safety and |
| la a a d'a u | Effectiveness of REAL I | Effectiveness of REAL |
| header | INTELLIGENCE™ CORI™ in | INTELLIGENCE™ CORI™ in |
| | unicondylar knee arthroplasty i | unicondylar knee arthroplasty (UKA) |
| | (UKA) procedures | Procedure |
| | Version: 2.0, 04SEP2020 | Version: 2.1, 14JAN2021 |
| | A Prospective, Multi-center, | A Prospective, Multi-center, |
| Section | Randomized Controlled Study to | Randomized Controlled Study to |
| 1.2.1&1.2.2 | Evaluate the Safety and I | Evaluate the Safety and |
| | Effectiveness of REAL I | Effectiveness of REAL |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 110 of 167 |

| | INTELLIGENCE™ CORI™ in | INTELLIGENCE™ CORI™ in |
|---|---|---|
| | unicondylar knee arthroplasty | unicondylar knee arthroplasty (UKA) |
| | (UKA) procedures", version 2.0, | Procedure", version 2.1, dated |
| | dated 04SEP2020 | 14JAN2021 |
| | A Prospective, Multi-center, | A Prospective, Multi-center, |
| | Randomized Controlled Study to | Randomized Controlled Study to |
| | Evaluate the Safety and | Evaluate the Safety and |
| Synopsis | Effectiveness of REAL | Effectiveness of REAL |
| | INTELLIGENCE™ CORI™ in | INTELLIGENCE™ CORI™ in |
| | unicondylar knee arthroplasty | unicondylar knee arthroplasty |
| | (UKA) procedures | (UKA) Procedure |

# 2nd Update from Version 2.1 to Version 3.0-Master

| Section | Current Text<br>Version 2.1 (14JAN2021) | Revised Text<br>Version 3.0-Master (03MAR2021) |
|---|---|---|
| | Original Text | Added "Single Identification Number |
| Cover | | of Clinical Investigation: |
| Page | | CORI.2019.06" |
| | Protocol Author(s): | Protocol Author(s): |
| | Rahel Meister, Senior Clinical | Michelle Li, Associate Clinical Study |
| | Study Manager | Manager |
| Cover | Babajide Olayinka, Senior | Rahel Meister, Senior Clinical Study |
| Page | Biostatistician | Manager |
| | | Babajide Olayinka, Senior |
| | | Biostatistician |
| | Version: 2.1, Date: 14JAN2021 | Version: 3.0-Master, Date: |
| Header | | 03MAR2021 |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 111 of 167 |

| | TMP-CD-05-01 - Clinical | TMP-CD-05-01 - Clinical Protocol- |
|---|---|---|
| Footer | Protocol-Device – Revision B; | Device – Revision D; SOP-CD-05 |
| | SOP-CD-05 Clinical Protocols | Clinical Protocols |
| | Protocol Version: 2.1, Date: | Protocol Version: 3.0-Master, Date: |
| Section | 14JAN2021 | 03MAR2021 |
| 1.1 &1.2 | | Merge the Signature and Date into |
| | | same column |
| | I agree to comply with the | I agree to comply with the |
| | Investigator's Obligations | Investigator's Obligations stipulated |
| | stipulated in Section 22.5 | in Section 6 Principal Investigator |
| C4: 1 1 | Principal Investigator Obligations | Obligations according to ISO |
| Section 1.1 | according to ISO 14155:2011. | 14155:2011 and all applicable local |
| | and applicable laws and | legislation and regulations |
| | regulation in China (NMPA) of | |
| | the protocol. | |
| | Refer to version 2.0 for full | Full stakeholders signature list |
| | sponsor approval. Approval of | |
| | the head of China clinical | |
| | operations indicates approval | |
| | both of the changes to the | |
| | protocol and of the changes | |
| Section 1.2 | being processed and approved | |
| | as a minor amendment. | |
| | Astrid Yung | |
| | Associate Director, Clinical | |
| | Strategy and Operations | |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep<br>2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | |

| | 11. Subject in the opinion of the | 11. Subject in the opinion of the |
|---|---|---|
| Sections 2 | Investigator has an emotional or | Investigator has an emotional or |
| | neurological condition that would | neurological condition that would pre- |
| | pre-empt their ability or | empt their ability or willingness to |
| and 7.3 | willingness to participate in the | participate in the study including |
| | study including mental illness, | mental illness, intellectual disability, |
| | mental retardation, drug or | or drug or alcohol abuse. |
| | alcohol abuse. | |
| | Study Duration: | Study Duration: |
| | Estimated timeline: | Estimated timeline: |
| | •Study period: 25 months (12 | •Study period: 25 months (12 months |
| | months enrolment) | enrolment) |
| | •Start enrolment: December | •Start enrolment: March 2021 |
| Section 2 | 2020 | •Last subject first visit: March 2022 |
| | •Last subject first visit: February | •Last subject last visit: May 2023 |
| | 2022 | |
| | •Last subject last visit: April | |
| | 2020 | |
| | Safety Data: | Safety Data: |
| | All AEs will be categorized in | All AEs will be categorized in terms of |
| | terms of seriousness and | seriousness and relatedness to the |
| | relatedness to the study device | study device or to the surgical |
| | or to the surgical procedure | procedure (Adverse Events, Serious |
| Section 2 | (Adverse Events, Serious | Adverse Events, Adverse Device |
| | Adverse Events, Adverse Device | Effects, Serious Adverse Device |
| | Effects, Serious Adverse Device | effects). All Serious Adverse Device |
| | , | Effects will be further categorized as |
| | Device Effects will be further | Anticipated or Unanticipated. The |
| | categorized as Anticipated or | definitions for each of these |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 113 of 167 |

| | Unanticipated. The definitions for | categories are based on ISO |
|---|---|---|
| | each of these categories are | 14155:2011 and applicable local laws |
| | based on ISO 14155:2011 and | and regulations. |
| | applicable local laws and | |
| | regulations. in China. | |
| | (Including hardware and | |
| | instrumentation), complications, | |
| | and revisions. | |
| | Original Table of Content, List of | Updated Table of Content, List of |
| Section 3.1 | Tables & List of Figures | Tables & List of Figures |
| 83.2 & 3.3 | | Numbering updated for all tables and |
| | | figures throughout the protocol |
| | KSS - Knee Society Score | 2011 KSS - Knee Society Score, 2011 |
| Section 3.4 | | HKA – Hip-Knee-Ankle |
| | The primary objective of this | The primary objective of this study is |
| | study is to evaluate the use of | to evaluate the use of CORI in UKA |
| | CORI in UKA procedures in | procedures in achieving post- |
| Section 5.1 | achieving post-operative leg | operative leg alignment as compared |
| | alignment as compared to | to procedures using conventional |
| | procedures using standard | manual instruments. |
| | instruments. | |
| | The secondary objective of this | The secondary objective of this study |
| | study is to assess the safety and | is to generate safety and performance |
| | performance of CORI up to 12 | evidence supporting the use of CORI |
| | months after surgery as | procedures. To assess the safety and |
| Section 5.2 | compared to procedures using | performance of CORI up to 12 months |
| | conventional manual | after surgery as compared to |
| | instruments. | procedures using conventional |
| | | manual instruments. |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 114 of 167 |

| | Other objectives are to | Other objectives are to collect the |
|---|---|---|
| Section<br>5.3 | determine the system time and | system time and cutting time of the |
| | cutting time of the robotic drill of | robotic drill from the CORI Case |
| | UKA procedures with CORI. | Report. |
| G 6 | Title: NVESTIGATIONAL | Title: NVESTIGATIONAL PRODUCT(S) |
| Section 6 | PRODUCT(S) | AND COMPARATOR |
| | Figure 6.1-6-1 CORI | Figure 6.1-6-2 CORI Reusable |
| | Reusable Instruments | Instruments |
| Section | CORI Robotic Drill: Controls | CORI Robotic Drill: Controls the |
| 6.1.1 | the position and speed of the | position and speed of the bur. It is |
| | bur. It is intended for 5 uses and | intended for 75 uses and is able to be |
| | is able to be autoclaved, auto | autoclaved, auto washed, and |
| | washed, and disinfected. | disinfected. |
| Section | Not Exist | Added new section "Ancillary |
| 6.1.3 | | Product(s)->Not applicable. |
| | For Australia, Hong Kong and | For Australia, Hong Kong and New |
| | New Zealand the list of reference | Zealand the list of reference |
| Section | documents can be found in | |
| 6.2 | Appendix Section 22.2 | Section 22.3 Instruction For Use & |
| | Instruction For Use & User | User Manual. |
| | Manual. | |
| | | The standard commercial packaging |
| Section<br>6.3.1 | pacaing as marketed in the US is | as marketed in the US is used. |
| | used. However, additional labels | However, additional labels will be |
| | will be included on the | included on the commercial |
| | commercial packaing to meet the | packaging to meet the regulatory |
| | regulatory requirements for | requirements for investigational |
| | investational devices in countries | devices in countries where the |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep<br>2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 115 of 167 |

| | where the devices are not | devices are not approved for |
|---|---|---|
| | approved for marketing. | marketing. |
| | Not Exist | New added section "Medical |
| | | Procedure-> There are 3 basic steps |
| | | in unicondylar knee arthroplasty. The |
| | | first step is preparing the bone and |
| | | removing the cartridge from the |
| | | damaged knee compartment. This will |
| | | be completed using either the CORI |
| | | robotic drill or an oscillating saw. The |
| | | surgeon will then position the metal |
| | | implants on the damaged side of the |
| | | femur and tibia using several |
| | | orthopaedic tools. Finally, a spacer |
| | | will be inserted between the metal |
| Section<br>6.6 | | implants to reduce friction when the |
| 0.0 | | knee flexes and extends. At various |
| | | times during the procedure, the hip- |
| | | knee-ankle angle (HKA) will be |
| | | checked using the CORI advanced |
| | | tracking system or via the use of |
| | | intramedullary and / or |
| | | extramedullary rods. How the angle is |
| | | measured will depend on which |
| | | treatment arm the subject is |
| | | randomized to receive. All |
| | | unicondylar knee arthroplasty is |
| | | completed using general anaesthetic |
| | | by a surgical team trained in both the |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized | Version: 4.0-Master, 07 Sep |
| Controlled Study to Evaluate the Safety and | 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | |

| | | CORI system and the use of standard |
|---|---|---|
| | | manual instrumentation. |
| Section 7.3 | Exclusion Criteria No. 1-7 | Exclusion Criteria No. 7-13 |
| | The subject, or their legally | The subject, or their legally |
| Section 7.5 | authorized representative | authorized representative (if |
| 7.5 | | applicable) |
| | • Subject noncompliance (e.g., | Subject noncompliance (e.g., did |
| | did not follow instructions, | not follow instructions, took |
| | took disallowed medications) | disallowed medications) |
| | Subject lost to follow-up | Subject is lost to follow-up |
| | • The Investigator or the | • The Investigator or the Sponsor |
| | Sponsor stops the study for | terminates the study for any |
| | any reason and decides to | reason |
| | withdraw subject(s) from the | Concurrent illness |
| Section | study | Adverse Events/Adverse Device |
| 7.8.2 | Concurrent illness | Effects |
| | Adverse Events/Adverse | • Any other significant reason |
| | Device Effects | identified by the Investigator. |
| | Any other significant reason | |
| | identified by the Investigator | Subjects who withdraw or are |
| | | withdrawn by the Investigator cannot |
| | Subjects who drop out or are | be-re-enrolled in the study. |
| | withdrawn will not be-re-entered | |
| | into the study at a later date. | |
| | Study participation is voluntary, | Study participation is voluntary, and |
| Section<br>7.8.3 | and subjects may withdraw at | subjects may withdraw from the |
| | any point during the study | study at any time. Where subjects |
| | without giving their reason for | withdraw consent, the Investigator |

unicondylar knee arthroplasty (UKA) Procedure

# Clinical Protocol A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in  Study Number: CORI.2019.06 Version: 4.0-Master, 07 Sep 2022 

| | daine an Mhaire airbianta | should made a management offert to |
|---|---|---|
| | doing so. Where subjects | |
| | withdraw consent, the | ascertain the reason(s), while fully |
| | Investigator should make a | respecting the subject's right to |
| | reasonable effort to ascertain the | privacy. The reason for withdrawal |
| | reason(s), while fully respecting | will be recorded in the eCRF and |
| | the subject's privacy. The reason | source documents. |
| | for withdrawal will be recorded in | |
| | the eCRF and source documents. | |
| Section<br>8.1-Figure<br>8-1 | August November December 2020 2020 2020 UKA Market Access Principles UKA Cohort Enrolment UKA Cohort Enrolment | August November March March May 2020 2020 2021 2022 2023 UKA Market Access Training & Pre-Study Cases Enrolment Follow-up |
| | Within the Primary UKA segment | Subjects will be randomly assigned to |
| | of the study, subjects will be | the CORI navigational or conventional |
| | randomly assigned to the CORI | manual instrumentation groups |
| Section | Navigational or Conventional | according to a balanced |
| 8.2.1 | manual instrumentation groups | randomization procedure using a 1:1 |
| | according to a balanced | allocation ratio. |
| | randomization procedure using a | |
| | 1:1 allocation ratio. | |
| | Not Exist | New added section "DATA |
| | | MANAGEMENT" |
| Section<br>8.3 | | This study utilizes a validated, |
| | | encrypted electronic data capture |
| | | system that is 21 CFR Part 11 |
| | | compliant. Access to the electronic |
| | | data capture system is restricted by |
| | | study role in accordance with Smith |
| | | and Nephew procedures. |
| | | and Nephew procedures. |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 118 of 167 |

A Data Management Plan (DMP) is written according to Smith and Nephew procedures containing details of the data management process. The following is a brief description of the key points detailed in this plan.

8.3.1 Data Review and Quality Assurance

Data will be transcribed from the data source to an electronic Case Report Form (eCRF). All data requested on the eCRFs are considered required. Data points not collected and/or recorded will be considered deviations unless otherwise specified.

Data collection is the responsibility of the clinical trial staff at the site under the supervision of the Principal Investigator. The Principal Investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported. The Principal Investigator provide his/her electronic signature on the appropriate eCRFs to be documented in compliance with local regulations. Changes to data

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 119 of 167 |

| | | proviously submitted to the special |
|---|---|---|
| | | previously submitted to the sponsor |
| | | will require a new signature by the |
| | | Investigator to acknowledge/approve |
| | | the changes. |
| | | Visual and computer data review will |
| | | be performed in line with Smith and |
| | | Nephew procedures to identify |
| | | possible data discrepancies. Manual |
| | | and automatic queries will be created |
| | | within the electronic data capture |
| | | system, and will be issued by Smith |
| | | and Nephew to the site for |
| | | appropriate response. Site staff are |
| | | responsible for resolving all queries in |
| | | the electronic data capture system. |
| | | 8.3.2 Retention Period |
| | | All eCRFs will be archived once the |
| | | study is completed and will kept for a |
| | | period of no less than five years after |
| | | the later of the following dates: the |
| | | date of which the study is terminated |
| | | or completed or; the date that the |
| | | records are no longer required |
| | | supporting marketing applications. |
| Section<br>8.4.3 | robotic drills | robotic drills |
| Section | In order to eliminate selection | Original Sentence deleted |
| 8.5.1 | bias, investigators will | |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep<br>2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in | |
| unicondylar knee arthroplasty (UKA) Procedure | raye. 120 01 10/ |

| | continuously screen eligible | |
|---|---|---|
| | subjects. | |
| | Subjects meeting all | Subjects meeting all |
| | inclusion/exclusion criteria will | inclusion/exclusion criteria will be |
| | be randomly allocated into any of | randomly allocated to one of two |
| Section<br>8.5.2 | two study groups (CORI | treatment groups (CORI Navigational |
| 0.3.2 | Navigational versus conventional | versus conventional manual |
| | manual instrumentation groups) | instrumentation) in a 1:1 allocation |
| | in a 1:1 allocation ratio. | ratio. |
| | The details of the analyses will | The details of all analysis to be |
| | further be pre-specified in the | performed will further be pre- |
| | Statistical Analysis Plan (SAP) so | specified in the Statistical Analysis |
| Section<br>8.5.4 | as minimize any threats to | Plan (SAP) so as to minimize any |
| 0.5.4 | external validity and yield | threats to external validity and yield |
| | clinically relevant estimates of | clinically relevant estimates of effects |
| | effects and precision. | and precision. |
| | 1.Obtain written informed | 1.Obtain written informed consent |
| | consent from the subject as | from the subject as detailed in |
| | detailed in Section 7.5. Any | Section 7.5. |
| | subject who signs an informed | |
| Section<br>9.1.2 | consent but fails to meet the | |
| | entry criteria is considered to be | |
| | a Screen Failure. Their | |
| | demographic information must | |
| | be captured in the appropriate | |
| | electronic Case Report Form | |
| | (eCRF) with the reason for | |
| | screen failure specified. | |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 121 of 167 |

| | Original text | Add" No. 11- The subject will be |
|---|---|---|
| Section<br>9.1.2 | | randomized to treatment group |
| | | (CORI or Manual conventional |
| | | instrumentation)." |
| | 1. Check if there is any change in | 1. Prior to surgery, check if there is |
| | eligibility of the subject since the | any change in eligibility of the subject |
| | pre-operative visit. If the subject | since the pre-operative visit. If the |
| | is no longer eligible, document | subject is no longer eligible, |
| | as screening failure | document as screening failure. |
| Section<br>9.1.3 | 7. Instruct the subject on proper | 7. Instruct the subject on proper |
| 9.1.3 | postoperative care/procedures, | postoperative care/procedures. |
| | including any contraindicated | |
| | treatments/medication(s). | Remove Randomization procedure |
| | | into Pre-op, which is mentioned |
| | | above. |
| | Where possible, a full Exit Visit | Where possible, the next scheduled |
| Section | should be completed for all | study visit should be completed for all |
| 9.1.9 | subjects who discontinue the | subjects who discontinue the study |
| | study early. | early. |
| Section | radiolucent lines, osteolysis & | radiolucent lines, osteolysis & implant |
| 9.2.3 | implant migration) | migration |
| | All statistical comparisons of | All statistical comparisons of data will |
| Section | data would describe the test | describe the test statistic used as well |
| 10.1 | statistic used as well as its | as its distributional assumptions. |
| | distributional assumptions. | |
| | Original Text | Newly Added "Randomized |
| Section<br>10.2 | | Population: This is defined as subjects |
| 10.2 | | randomized to either CORI or |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 122 of 167 |

| | | Conventional manual instrumentation |
|---|---|---|
| | | groups." |
| The ITT population | n is defined as | The ITT population is a subset of the |
| subjects randomiz | zed to either | randomized population which is |
| CORI or convent | tional manual | defined as subjects randomized to |
| instrumentation | groups who | either CORI or conventional manual |
| have at least one p | post-operative | instrumentation groups who have at |
| assessment on | any of the | least one post-operative assessment |
| | ndpoints or | on any of the effectiveness endpoints |
| Section health-related qu | uality of life | or health-related quality of life |
| (HRQoL) endpo | oints. Data | (HRQoL) endpoints. Data summarized |
| summarized on | the ITT | on the ITT population will be based on |
| population will be | based on the | the intervention the subject was |
| implant the s | subject was | randomized to receive which may be |
| randomized to r | eceive which | different from the intervention the |
| may be different fr | om device the | subject actually received. |
| subject actually re- | ceived. | |
| Original Text | | New Added "For missing primary |
| | | endpoint data, the Missing Value |
| | | Treated as Failure (MVTF) missing |
| | | value imputation method will be used. |
| | | This is considered a conservative |
| Section | | imputation method as all missing data |
| 10.4.1 | | on the primary endpoint will be |
| | | considered as a failure, i.e. not |
| | | attaining the pre-specified target |
| | | alignment. More specific details of this |
| | | imputation method will be included in |
| | | • |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep<br>2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 123 of 167 |

| | The transformed FJS-12 score | The transformed FJS-12 score (0- |
|---|---|---|
| Section | (0-100) will be summarized at | 100) will be summarized at the |
| | the preoperative and | postoperative visits using continuous |
| 10.4.2 | postoperative visits using | summary characteristics. |
| | continuous summary | |
| | characteristics. | |
| Section | Original Text | Text Updated according to Protocol |
| 12.1.1<br>&12.1.2 | | Template Rev D. |
| &12.1.3 | | |
| &12.1.4<br>&12.1.7 & | | |
| 12.3 | The Driverine Investigates will | The Drive sized Toylooki sake will save play |
| | The Principal Investigator will | The Principal Investigator will comply |
| | comply with the commitments | with the commitments outlined in the |
| | outlined in the in the Statement | in the Statement of Investigator, |
| | of Investigator, provided by the | provided by the Sponsor, and with |
| | Sponsor, and with Good Clinical | Good Clinical Practice (GCP), and all |
| Section 13 | Practice (GCP), and all applicable | applicable regulatory requirements as |
| | regulatory requirements as | outlined in Appendix-Principal |
| | outlined in Appendix-Principal | Investigator Obligations as well as all |
| | Investigator Obligations as well | applicable local laws and regulations. |
| | as applicable laws and | |
| | regulations in China of this | |
| | protocol. | |
| | Not Exist | New added section "Interim |
| Castina | | Monitoring Visit-> Regular interim |
| Section<br>14.4 | | monitoring visits will be performed by |
| | | the Sponsor or qualified person |
| | | designated by the Sponsor." |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 124 of 167 |

| | Public/Products Liability | Public/Products Liability Insurance |
|---|---|---|
| | Insurance has been purchased | has been purchased by Smith & |
| | by Smith & Nephew plc. | Nephew plc. Worldwide and |
| | Worldwide and incorporates | incorporates coverage for personal |
| | coverage for personal injury in | injury in respect of clinical studies. |
| | respect of clinical studies. The | The Sponsor agrees to operate in |
| Section 18 | Sponsor agrees to operate in | good faith and in accordance with the |
| | good faith and in accordance | local guidelines regarding |
| | with ABHI (Association of British | compensation for injury resulting |
| | Healthcare Industries) guidelines | from participation in an industry- |
| | regarding compensation for | sponsored clinical trial. |
| | injury arising in the course of | |
| | clinical studies. | |
| | Should circumstances arise | Should circumstances arise which |
| | which require the termination of | require the termination of the entire |
| | the entire study prior to its | study prior to its planned completion |
| | planned completion (e.g., safety | (e.g., safety concerns) or |
| | concerns) or circumstances arise | circumstances arise which mean the |
| | which mean the end of the | end of the participation of an |
| Section 19 | participation of an individual site | individual site (e.g., departure of |
| | (e.g., departure of Investigator, | Investigator, non-compliance), then |
| | non-compliance), then this will | this will be undertaken according to |
| | be undertaken according to the | the SOPs of the Sponsor. The |
| | SOPs of the Sponsor. | requirement for subject follow up in |
| | | these instances will be considered as |
| | | part of these processes. |
| Section<br>20.2 | S+N | Smith+Nephew |
| 20.2 | | |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 125 of 167 |

| | The accompany to be a larger than a contract | The |
|---|---|---|
| | I ne purpose to nave the protocol | The purpose to have the 1 <sup>ST</sup> protocol |
| | amendment is to meet the | amendment is to meet the |
| | requirements of the Hongkong | requirements of the Hong Kong site |
| | site during the EC approval | during the EC approval session. The |
| | session. The protocol | protocol amendment for version 2.1 is |
| Section | amendment for version 2.1 is | minor. |
| 22.1.1 | minor. | The purpose to have the 2nd protocol |
| | | amendment into version 3.0-Master is |
| | | to update the protocol from Template |
| | | B into Template D and also update the |
| | | information within the protocol. |
| | The rationale to update the | The rationale to 1 <sup>ST</sup> time protocol |
| | protocol is due to the protocol | update is due to the protocol title |
| | title inconsistency with other | inconsistency with other documents. |
| | documents. Since the | Since the amendment is change that |
| | amendment is change that do | do not materially affect the study |
| | not materially affect the study | which is simply update the protocol |
| | which is simply update the | title from "procedures" into |
| | protocol title from "procedures" | "Procedure". Therefore, the |
| Section | into "Procedure". Therefore, the | amendment for version 2.1 is |
| 22.1.2 | amendment for version 2.1 is | considered as minor. |
| | considered as minor. | |
| | | The rationale to 2nd time update the |
| | | protocol is due to the protocol |
| | | template updated from version B to |
| | | version D. And also the information |
| | | inside of the protocol need to be |
| | | · |
| | | further updated. |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 126 of 167 |

| | $1^{\text{ST}}$ Update from Version 2.0 to | 2 <sup>nd</sup> Update from Version 2.1 to |
|---|---|---|
| Section<br>22.1.4 | Version 2.1 | Version 3.0-Master. |
| | | This table added |
| | Not Exist | New section added "Sponsor |
| Section | | Details"-> Smith & Nephew, Inc., |
| 22.2 | | 1450 E. Brooks Road, Memphis, TN |
| | | 38116, United States |
| Section | Not applicable | Refer to Section 9.2 & 9.3 for Quality- |
| 22.4 | | of-Life measures. |

# 3rd Update from Version 3.0-Master to Version 4.0-Master

| | Current Text | Revised Text |
|---|---|---|
| Section | Version 3.0-Master (03<br>MAR2021) | Version 4.0-Master (07 Sep 2022) |
| Throughout<br>as<br>applicable | acronym vs full term. | I at first use and tidying up use of the n+Nephew, and Smith&Nephew more |
| ISO 14155<br>reference | ISO reference changed from ISO 14155:2011 to ISO14155:2020 throughout the study. | |
| Header | Version: 3.0-Master, 03<br>MAR2021 | Version: 4.0-Master, Date 07 Sep 2022 |
| Section<br>1.1&1.2 | Protocol version and date: 3.0-Master, 03 MAR2021 | Version: 4.0-Master, Date 07 Sep 2022 |
| Cover Page | Protocol Author(s): Michelle Li, Associate Clinical Study Manager | Protocol Author(s): Michelle Li, Associate Clinical Study Manager |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 127 of 167 |

| | Pahal Maistar Sanjar Clinical | Rahel Meister, Senior Clinical Study |
|---|---|---|
| | • | |
| | Study Manager | Manager |
| | Babajide Olayinka, Senior | Manvendra Saxena, Clinical Study |
| | Biostatistician | Manager |
| | | Babajide Olayinka, Senior |
| | Sponsor Approval | Biostatistician |
| | Kelli C. Armstrong, | |
| | Clinical Strategy Director | Sponsor Approval |
| | Robotics | Julie Lankiewicz, |
| | | Clinical Strategy Director Robotics |
| | Alan Rossington, Director | |
| | Biostatistics & Data | Michael Robinson |
| | Management | Independent Statistician |
| | Original Text- Coordinating | Update the section into Clinical |
| Section 1.2 Investigator Approval | | Institution Approval page |
| Section 1.3 | Full internal sponsor approval | Only China operation head approval |
| | | a. Added "Targeted Global |
| | | Region- Added South Korea |
| | | b. Exclusion Criteria: Changed |
| | | "point 3: Subject receives |
| | | simultaneous bilateral UKA |
| Synopsis- | | OR a unilateral UKA with |
| Exclusion Criteria & | Original Text | contralateral TKA. |
| Section 7.3 | | c. Added exclusion criteria |
| | | "point 4: Subject has one or |
| | | arthroplasties that are not |
| | | fully healed and well- |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep<br>2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 128 of 167 |

| functioning, as determined |
|------------------------------------|
| by the investigator: |
| -Contralateral primary TKA or |
| UKA, however, the subject |
| can only have one knee |
| enrolled in this study". And |
| "point 6: Subject currently |
| enrolled in another orthopedic |
| d. Study Duration Timeline |
| updated |
| e. Study Schedule |
| Screening |
| i. Visit Duration changed |
| from -28 to 0 day to- |
| 90 to 0 days. |
| ii. Added subsection 1- |
| pre-operative long leg |
| X-rays (A/P) collected |
| 6-months prior to the |
| date of surgery is |
| admissible. |
| Study Duration |
| Study period: 49 months |
| Start enrollment: April 2022 |
| Last subject first visit: Feb 2024 |
| Last subject last visit: May 2026 |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 129 of 167 |

| Study<br>Schedule &<br>Table 9.1.1- | ldy nedule & Original Study Schedule Table Information Consert Demographics/Medica | Schedu<br>le of<br>events | | Data<br>&<br>Disc<br>harg<br>e<br>Day | 6<br>we<br>eks<br>42<br>±<br>14<br>day<br>s | 6<br>mo<br>nth<br>s<br>180<br>±<br>14<br>day<br>s | 12<br>mo<br>nth<br>s<br>365<br>±<br>30<br>day<br>s |
|---|---|---|---|---|---|---|---|
| 9-1 | | Informe<br>d<br>Consent | x | | | | |
| | | Demogr<br>aphics/<br>Medical<br>History | х | | | | |
| | | | | Inclusio<br>n/Exclu<br>sion | х | | |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 130 of 167 |

| Preoper ative Examin ations (eg. ECG, Blood Routine Examin ation, Bioche mical Examin ation, Coagula tion Examin ation) (1) | x | | | | |
|---|---|---|---|---|---|
| Pregnan<br>cy Test | х | | | | |
| Concom<br>itant<br>Medicati<br>on | x | - | | | |
| Concom<br>itant<br>Medicati<br>on<br>Update | | x | х | x | х |
| Operati<br>ve Data<br>Collecti<br>on | | x | | | |

# Clinical Protocol A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure Study Number: CORI.2019.06 Version: 4.0-Master, 07 Sep 2022 

| CORI<br>Case | | | | | |
|---|---|---|---|---|---|
| Report<br>(Syste<br>m time<br>&<br>cutting<br>time) | | х | | | |
| Dischar<br>ge Data<br>Collecti<br>on | | x | | | |
| Leg<br>alignme<br>nt long<br>leg X-<br>ray AP <sup>3</sup> | x | (x) <sup>4</sup> | x | | (x) <sup>5</sup> |
| Standar<br>d<br>Lateral<br>X-ray:<br>Knee | | (x) <sup>4</sup> | x | | x |
| Standar<br>d A/P<br>X-ray:<br>Knee | | | | | х |
| KSS<br>2011 | | | | | |
| OKS | Х | | х | х | х |
| FJS | Х | | Х | Х | x |
| EQ-5D-<br>5L | | | x | x | х |
| Safety<br>Assess<br>ment | Х | | х | x | х |
| End of<br>Study/E<br>xit | | x | х | x | х |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 132 of 167 |

| | | <ol> <li>(x)<sup>6</sup> (x)<sup>6</sup> (x)</li> <li>Applicable, at China sites only</li> <li>Applicable, at China sites only.</li> <li>Pre-operative long leg X-rays (A/P) collected 6-months prior to the date of surgery is admissible.</li> <li>Post-operative standing weight bearing long leg X-rays (A/P) and standard lateral X-rays may be taken at discharge.</li> <li>To be performed, only if standing weight bearing long leg A/P X-ray is taken as a standard of care at 12 and 24 months.</li> <li>Exit form to be completed at the point of withdrawal if the study is not completed.</li> </ol> |
|---|---|---|
| Region<br>South Korea | Not exist | Added throughout the protocol where applicable. |
| Section 6.5<br>"Surgical<br>Technique" | Original Text | All CORI study related procedures must be performed according to the User's Manual (Document ID: 500230 CORI for Knee Arthroplasty for Australia, Hong Kong, South Korea, and New Zealand, as well as Investigator's Brochure for China) and according to the according to the surgical technique |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 133 of 167 |

and IFU of the specific Smith+Nephew Implant System.

The primary endpoint of post-operative leg alignment is defined as the proportion of subjects achieving post-operative leg alignment 6 weeks after surgery within ± 3° from target. Because this assessment is comparing the target alignment vs measured alignment from 6 weeks postoperative imaging, the defined method of preoperatively planning alignment is left up to the individual investigator's discretion. Each investigator is to plan according to their own techniques.

For the analysis of the primary endpoint, X-ray or CT may be utilized.

The recommended CORI bone removal technique is a "burr all" technique per the user's manual (Document ID: 500230 CORI Knee Arthroplasty for Australia, Hong Kong, South Korea, and New Zealand, as well as Investigator's Brochure for China). However, a hybrid approach using "distal precision burring" may be used per surgeon's discretion. This will be

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 134 of 167 |

| | | captured in the eCRF along with a |
|---|---|---|
| | | rationale of why this approach was |
| | | chosen. |
| | | Resurfacing of the patella will be left up |
| | | to the discretion of each investigator. |
| | | This will be captured in the eCRF. |
| | | Surgeons selected to participate in this |
| | | study will be familiar with CORI and |
| | | have written evidence of training and |
| | | expertise in the study procedure. The |
| | | surgeons will conduct pre-study CORI |
| | | cases, in order to establish the |
| | | expertise of the individual surgeons. |
| | | The exact number may be adjusted |
| | | depending on the level of the individual |
| | | experience of the surgeon, the subjects |
| | | will not be randomized. |
| | | CORI Case Report Forms of the non- |
| | | randomized cases will be collected as |
| | | proof of surgeons' experience and for |
| | | inclusion in the safety analysis set |
| | | (applicable only at sites in China). |
| | Original Text | Changed to |
| 7.1 "Subject | "A total of 140 subjects will | At least 145 subjects will be enrolled |
| Population" | be enrolled in the study in up | into the study. At least 5 of these |
| | to 8 sites in Australia, Hong | subjects will be treated with CORI |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 135 of 167 |

| | Kong, New Zealand, and China Mainland". | directly to fulfil the learning needs of the surgeons prior to enrolling, a further 140 subjects who will be enrolled in the randomized stage of the study in up to 8 sites in Australia, China (Hong Kong), New Zealand, South Korea, and China mainland. Seventy (70) subjects will be enrolled for UKA with the use of the CORI and 70 subjects will be enrolled for UKA with the use of conventional manual instrumentation. Vulnerable subjects will not be enrolled in this study. |
|---|---|---|
| Section 7.3 "Exclusion Criteria" | | "Subject currently enrolled in another orthopedic clinical trial study |
| Section 7.4<br>"Screening" | Original Text "Investigators should consecutively screen all subjects presenting with degenerative joint disease of the knee, requiring correction of functional deformity, or treatment of fractures that were unmanageable using other techniques to determine whether they meet | Changed To "Investigators should consecutively screen all subjects presenting with degenerative joint disease of the knee, requiring correction of functional deformity, or treatment of fractures that were unmanageable using other techniques to determine whether they |

# **Clinical Protocol**

A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure Study Number: CORI.2019.06

Version: 4.0-Master, 07 Sep

2022

document

**Page**: 136 of 167

all

all inclusion and none of the exclusion criteria.

Participating study sites are required to document all screened subjects considered for inclusion in this study. If a subject is excluded from the study, the reasons for exclusion will be documented the subject's source documents and noted on the Screening and Enrollment Log. All screening activities that occur prior to consent shall be referred to as prescreening".

meet all inclusion and none of the exclusion criteria.

Participating study sites are required to

screened

subjects

considered for inclusion in this study. If a subject is excluded from the study, the reasons for exclusion will be documented in the subject's source documents and noted on the Screening and Enrollment Log. All screening activities that occur prior to consent shall be referred to as pre-screening. In China sites, part of the screening process will include documentation of women's childbearing potential. If the woman is not of childbearing potential this should be documented in the medical history (e.g., surgically postmenopausal, postmenopausal [i.e., at least one year without menses]). For women of childbearing potential, their method of birth control should be documented in the source".

# Section 7.5 "Informed Consent"

"Before conducting any study procedures or examinations, the purpose and nature of the

study should be explained to

Original Text

#### Changed To

"Before conducting any study procedures or examinations, the purpose and nature of the study should be explained to the subject in their native language.

# **Clinical Protocol**

A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure

Study Number: CORI.2019.06

Version: 4.0-Master, 07 Sep

2022

**Page**: 137 of 167

the subject in their native language.

The subject, or their legally authorized representative (if applicable), will then read, sign, and personally date IRB/IEC-approved the informed consent document(s) (see below for difficulties with reading and writing). Additionally, the individual who obtains consent from the subject will sign and date the informed consent document. A copy of the signed informed consent document will be provided to the subject, a copy will be the subject's placed in medical record, with the original filed in the ISF.

If the subject is unable to read, the informed consent document and associated study information may be read aloud to the subject in the presence of an impartial witness. Ιf possible, the subject shall sign and

The subject, or their legally authorized representative (if applicable), will then read, sign, and personally date the IRB/IEC-approved informed consent document(s) (see below for difficulties with reading and writing). Additionally, the individual who obtains consent from the subject will sign and date the informed consent document. A copy of the signed informed consent document will be provided to the subject, a copy will be placed in the subject's medical record, with the original filed in the ISF. If the subject is unable to read, the informed consent document associated study information may be read aloud to the subject in the presence of an impartial witness. If possible, the subject shall sign and personally date the Informed Consent Form (ICF). Where this is not possible, due to difficulties in writing, the subject shall provide verbal consent to participate in the study. The witness shall then personally sign and date the informed consent form, attesting that the information was accurately explained and that the informed consent was freely given.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 138 of 167 |

ICFs will comply with applicable laws personally date the Informed and regulations in Australia (Privacy Consent Form (ICF). Where this is not possible, due to Act 1988), China, South Korea, and New Zealand (Privacy Act 1993). If new difficulties in writing, the subject shall provide verbal information becomes available during consent to participate in the the course of the study that can study. The witness shall then significantly affect a subject's future personally sign and date the health and medical care, Smith + informed consent form, Nephew will ensure that information attesting that the information shall be provided to the subject(s) was accurately explained and affected in written form and if relevant, that the informed consent all affected subjects shall be asked to confirm their continuing consent in was freely given. ICFs will comply with Health writing". Information Portability Accountability Act (HIPAA) regulations as well as and applicable laws and regulations in Australia (Privacy Act 1988), China, South Korea, and Zealand (Privacy Act 1993)" <u>Added</u> Section "Withdrawn subjects will not be 7.8.2 **Original Text** "Withdrawal replaced" from Study"

# **Clinical Protocol**

A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure

Study Number: CORI.2019.06

Version: 4.0-Master, 07 Sep

2022


# Original Text

"This study is a prospective, multi-center, randomized controlled, non-blinded follow-up study to evaluate the use of CORI in UKA procedure in achieving post-operative leg alignment. Up to 8 sites will participate within Australia, China (Hong Kong), New Zealand, and China Mainland.

# Section 8.1 "Study Design"

Subjects will be enrolled and randomized into one of two (2) groups, as shown in Table 8.1-8-1.

All groups are treated with knee arthroplasty with a S+N Knee Implant System. (The implant system will be selected according to the registration status in each country)"

# Changed To

"This study is a prospective, multicenter, randomized controlled, non-blinded follow-up study to evaluate the use of CORI in UKA procedure in achieving post-operative leg alignment. Up to 8 sites will participate within Australia, Hong Kong, New Zealand, South Korea, and China Mainland.

The pre-randomized stage of the study will comprise of at least 5 subjects enrolled and treated with CORI directly in order to fulfil the learning needs of the surgeons. Subjects who will comprise the randomized stage of the study will be enrolled and randomized into one of two (2) groups, as shown in Table 8.1-8-1.

All groups are treated with knee arthroplasty with a S+N Knee Implant System. (The implant system will be selected according to the registration status in each country)"

# **Clinical Protocol**

A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure

Study Number: CORI.2019.06

Version: 4.0-Master, 07 Sep

2022

**Page**: 140 of 167

| Figure 8.1-<br>8-3 Study<br>Recruitment<br>Timeline | August November March March May 2020 2021 2022 2023 UNA Market Training & Pre-Study Case Enrolment Follow-up | August March April March April 2020 2022 2022 2024 2025 USA Market Access Pre-study Enrolment Follow-L |
|---|---|---|
| Section 10.2 "Analysis Population" Dot point "Randomize d Population" and "Safety Population | Original Text "Randomized Population: This is defined as subjects randomized to either CORI or Conventional manual instrumentation groups. "Safety Population (SAF): This is defined as all subjects who completed a TKA with the use of the CORI or conventional manual instrumentation". | "Randomized population" changed to "Enrolled Population" "Enrolled Population: This is defined as subjects enrolled and/or randomized to either CORI or Conventional manual instrumentation groups. A total of 140 patients will be competitively enrolled and or/randomized in the study across all the sites including the sites in China". "Safety Population (SAF): This is defined as all subjects who completed a TKA (include non-randomized subjects in China as CORI is pre- market product in China) with the use of the CORI or conventional manual instrumentation" |
| Section 11 "Sample Size Justification" | Original Text | "To account for up to a 10% attrition rate in knees enrolled, 70 knees in each |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 141 of 167 |

| | | group (140 knees combined) will be enrolled into the randomized stage of the study. A minimum of an additional 5 subjects who will be treated with CORI directly to fulfil the learning needs of the surgeons will be enrolled at the pre-randomized study stage, thus leading to a minimum total study enrollment of 145 subjects". |
|---|---|---|
| Section 21.1<br>"Publication<br>of Study<br>Data" | Original Text | Deleted Reference to "Health Insurance Portability and Accountability Act of 1996" |
| Section<br>23.1.1<br>"General<br>Purpose" | Original Text | "The Purpose of 3rd amendment is to expand the pre-operative data collection period, to increase the enrolment at all the sites and restrict the enrolment of patient who are either enrolled in the other study or were enrolled in the other study at least 1 year prior to screening during the EC approval session. |
| Section<br>23.6.1 | | Updated to ISO 14155:2020 guidelines. |

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 142 of 167 |

| "Principal |
|--------------|
| Investigator |
| Obligation |
| according to |
| ISO14155:2 |
| 020" |

### 22.1.5 Approval/Notification

The version 2.0-master and 2.1-master of this protocol was not implemented as the study was still at design phase. The protocol v3.0-Master was implemented at all the sites following local EC approval. The protocol v4.0-Master will get implemented in each country following the local EC approval. China protocol v4.0-China, which incorporates the updates in the master, will be implemented at sites in China after local EC approval.

#### **22.2 Sponsor Details**

Smith & Nephew, Inc., 1450 E. Brooks Road, Memphis, TN 38116, United States

#### 22.3 Instructions For Use & User Manuals

- CORI user's manual (Document ID: 500230, REAL INTELLIGENCE™ CORI™ for Knee Arthroplasty)
- IFU REAL INTELLIGENCE™ CORI™ Burs (Document ID: 500172)
- IFU REAL INTELLIGENCE™ CORI™ Flat Markers (Document ID: 500198)
- IFU REAL INTELLIGENCE™ CORI™ Irrigation (Document ID: 500173)
- IFU REAL INTELLIGENCE™ CORI™ Instrumentation Tray (Document ID: 500229)

#### 22.4 EQUIPMENT AND SPECIAL INSTRUCTIONS

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 143 of 167 |

The following section provides a list of components of CORI (only UKA instruments will be used for this study):

Table 22.4-22-1 CORI Components

| Article | Description |
|----------|---------------------------------------|
| ROB10000 | CORI Starter Kit |
| ROB10024 | REAL INTELLIGENCE CORI |
| ROB10025 | REAL INTELLIGENCE Tracking Camera |
| ROB10026 | REAL INTELLIGENCE Foot Pedal |
| ROB10027 | REAL INTELLIGENCE Tablet |
| ROB10028 | REAL INTELLIGENCE Transportation Case |

#### Table 22.4-22-2 CORI Cart

| Article | Description |
|-----------|------------------------------------------|
| ROB10002 | REAL INTELLIGENCE Robotics Cart Column |
| ROB100021 | REAL INTELLIGENCE Robotics Cart Base 120 |
| ROB100022 | REAL INTELLIGENCE Robotics Cart Base 220 |

#### Table 22.4-22-3 CORI Monitor

| Article | Description |
|----------|---------------------------------------|
| ROB10003 | REAL INTELLIGENCE 24 in. Touch Screen |

# **Table 22.4-22-4 CORI Tray and Instrumentation**

| Article | Description |
|----------|--------------------------------------------|
| ROB10001 | REAL INTELLIGENCE Robotics Instruments |
| ROB10010 | REAL INTELLIGENCE Bone Pins 4 mm x 127 mm |
| ROB10011 | REAL INTELLIGENCE Bone Pins 4 mm x 152 mm |
| ROB10012 | REAL INTELLIGENCE Checkpoint Pins |
| ROB10013 | REAL INTELLIGENCE Robotic Drill |
| ROB10014 | REAL INTELLIGENCE Robotic Drill Tracker |
| ROB10015 | REAL INTELLIGENCE Robotic Drill Attachment |
| ROB10016 | REAL INTELLIGENCE Robotic Drill Guard |

#### 

This document contains information that is confidential and proprietary to Smith & Nephew PLC and Smith & Nephew, Inc. and is intended for use only by Smith+Nephew and its manufacturer. It shall not be reproduced or copied in whole or in part, nor shall the contents be disclosed by any means without prior written permission from Smith+Nephew, nor shall anyone make any use of it that is contrary to the expressed or implied wishes of Smith+Nephew.

TMP-CD-05-01 Clinical Protocol - Device - Revision D; SOP-CD-05 Clinical Protocol

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 144 of 167 |

| Article | Description |
|----------|---------------------------------------------|
| ROB10017 | REAL INTELLIGENCE Point Probe |
| ROB10018 | REAL INTELLIGENCE Femur Tracker |
| ROB10019 | REAL INTELLIGENCE Tibia Tracker |
| ROB10020 | REAL INTELLIGENCE Tracker Clamp |
| ROB10021 | REAL INTELLIGENCE Drill Guide |
| ROB10022 | REAL INTELLIGENCE Checkpoint Tool |
| ROB10050 | REAL INTELLIGENCE Robotics Instruments Tray |
| ROB10051 | REAL INTELLIGENCE Robotics Pin Caddy |
| ROB10052 | REAL INTELLIGENCE Robotics Pin Caddy Lid |
| 71441351 | Rasp |
| 74013489 | Speed Pin Driver |
| 71935186 | SCOTT CEMENT CURETTE |
| 71935187 | CEMENT CURETTE |
| ROB10086 | REAL INTELLIGENCE Plane Visualizer |

# **Table 22.4-22-5 CORI Shipping Inserts**

| Article | Description |
|----------|---------------------------------------|
| ROB10055 | REAL INTELLIGENCE Shipping Insert (A) |
| ROB10056 | REAL INTELLIGENCE Shipping Insert (B) |
| ROB10057 | REAL INTELLIGENCE Shipping Insert (C) |
| ROB10058 | REAL INTELLIGENCE Shipping Insert (F) |

#### **Table 22.4-22-6 CORI Lids**

| Article | Description |
|----------|--------------------------|
| ROB10087 | Universal Base Tray Lid |
| ROB10088 | Universal Insert Lid (A) |
| ROB10089 | Universal Insert Lid (B) |
| ROB10090 | Universal Insert Lid (C) |
| ROB10054 | Universal Insert Lid (F) |
| ROB10091 | Universal Insert Lid (G) |
| ROB10097 | Universal Insert Lid (H) |
| ROB10098 | Universal Insert Lid (I) |
| ROB10095 | Universal Insert Lid (J) |

#### 

This document contains information that is confidential and proprietary to Smith & Nephew PLC and Smith & Nephew, Inc. and is intended for use only by Smith+Nephew and its manufacturer. It shall not be reproduced or copied in whole or in part, nor shall the contents be disclosed by any means without prior written permission from Smith+Nephew, nor shall anyone make any use of it that is contrary to the expressed or implied wishes of Smith+Nephew.

TMP-CD-05-01 Clinical Protocol - Device - Revision D; SOP-CD-05 Clinical Protocol
| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 145 of 167 |

#### **Table 22.4-22-7 CORI Instrument Reduction Modules - Kits**

| Article | Description |
|----------|---------------------------|
| ROB10004 | JOURNEY II Uni Medial |
| ROB10085 | JOURNEY II Uni Lateral |
| ROB10005 | JOURNEY II TKA Essentials |
| ROB10006 | JOURNEY II Distal Burring |
| ROB10007 | JOURNEY II CR Module |
| ROB10008 | JOURNEY II BCS Module |
| ROB10009 | JOURNEY II XR Module |
| ROB10067 | JOURNEY II Options Module |

## Table 22.4-22-8 CORI JOURNEY II UKA Inserts

| Article | Description |
|----------|------------------------------------------|
| ROB10053 | ROBOTICS FINISHING INSERT (F) |
| 74036185 | LEFT MEDIAL BASEPLATE TRIALS |
| 74036127 | MEDIAL INSERT TRIALS |
| 74036174 | RESECTION FEMORAL FINISHING TRIALS LM/RL |
| 74036187 | RIGHT MEDIAL BASEPLATE TRIALS |
| 74036190 | RESECTION FEMORAL FINISHING TRIALS RM/LL |
| 74036196 | LATERAL BASEPLATE TRIALS |
| 74036198 | LATERAL INSERT TRIALS |
| 74036190 | RESECTION FEMORAL FINISHING TRIALS RM/LL |
| 74036196 | LATERAL BASEPLATE TRIALS |
| 74036174 | RESECTION FEMORAL FINISHING TRIALS LM/RL |

## **Table 22.4-22-9 CORI JOURNEY II Instrument Reduction Inserts**

| Article | Description |
|----------|------------------------------|
| ROB10060 | ROBOTICS FINISHING BASE |
| ROB10066 | TIBIA FINISIHING INSERT (F) |
| ROB10092 | LEFT TRIAL BASE |
| ROB10062 | FEMUR TRIAL INSERT LEFT (FF) |
| ROB10064 | TIBIA TRIAL INSERT LEFT (C) |

#### 

This document contains information that is confidential and proprietary to Smith & Nephew PLC and Smith & Nephew, Inc. and is intended for use only by Smith+Nephew and its manufacturer. It shall not be reproduced or copied in whole or in part, nor shall the contents be disclosed by any means without prior written permission from Smith+Nephew, nor shall anyone make any use of it that is contrary to the expressed or implied wishes of Smith+Nephew.

TMP-CD-05-01 Clinical Protocol - Device - Revision D; SOP-CD-05 Clinical Protocol

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 146 of 167 |

| Article | Description |
|----------|-----------------------------------------------------|
| ROB10093 | RIGHT TRIAL BASE |
| ROB10063 | FEMUR TRIAL INSERT RIGHT (FF) |
| ROB10065 | TIBIA TRIAL INSERT RIGHT (C) |
| ROB10061 | DISTAL BURRING INSERT (GG) |
| ROB10068 | CR POLY TRIAL INSERT LEFT (II) |
| ROB10069 | CR POLY TRIAL INSERT RIGHT (II) |
| ROB10070 | CAM TRIAL INSERT LEFT |
| ROB10072 | JOURNEY II BCS Finishing Insert (A) |
| ROB10071 | CAM TRIAL INSERT RIGHT |
| ROB10079 | JOURNEY II Robotics XR Poly Trial Insert Left (CC) |
| ROB10080 | JOURNEY II Robotics XR Poly Trial Insert Right (CC) |
| ROB10094 | JOURNEY II XR Tibia Finishing Insert (J) |
| ROB10096 | JOURNEY II XR TIBIA IMPACTOR INSERT (GG) |
| ROB10073 | JOURNEY II BCS Poly Trial Insert Left (HH) |
| ROB10074 | JOURNEY II BCS Poly Trial Insert Right (HH) |
| ROB10075 | JOURNEY II BCS Constrained Insert Left (HH) |
| ROB10076 | JOURNEY II BCS Constrained Insert Right (HH) |
| ROB10077 | JOURNEY II CR Deep Dish Insert Left (HH) |
| ROB10078 | JOURNEY II CR Deep Dish Insert Right (HH) |
| ROB10081 | JOURNEY II XR Poly Upslope Trial Insert Left (HH) |
| ROB10082 | JOURNEY II XR Poly Upslope Trial Insert Right (HH) |
| ROB10083 | J2 Robotics Universal Spacer Trial Insert (CC) |
| ROB10099 | REAL INTELLIGENCE Flex Base |

# **Table 22.4-22-10 Total Knee Instruments**

| Article | Description |
|----------|------------------------------------|
| ROB00003 | TKA Femur Cut Adapter |
| ROB00005 | TKA Femur Distal Cut Guide – Small |
| ROB00006 | TKA Femur Distal Cut Guide – Med |
| ROB00007 | TKA Femur Distal Cut Guide – Lg |
| ROB00014 | TKA Femur Stabilizer – Small |
| ROB00015 | TKA Femur Stabilizer – Med |
| ROB00016 | TKA Femur Stabilizer – Lg |
| ROB00018 | TKA Drill Guide – Journey II |

#### 

This document contains information that is confidential and proprietary to Smith & Nephew PLC and Smith & Nephew, Inc. and is intended for use only by Smith+Nephew and its manufacturer. It shall not be reproduced or copied in whole or in part, nor shall the contents be disclosed by any means without prior written permission from Smith+Nephew, nor shall anyone make any use of it that is contrary to the expressed or implied wishes of Smith+Nephew.

TMP-CD-05-01 Clinical Protocol - Device - Revision D; SOP-CD-05 Clinical Protocol

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 147 of 167 |

| Article | Description |
|----------|-------------------------------------|
| ROB00024 | TKA Drill Guide – Genesis II/Legion |
| ROB00025 | TKA Left Tibia Twin Peg Cut Guide |
| ROB00026 | TKA Right Tibia Twin Peg Cut Guide |
| ROB00060 | TKA Distal FMR Punches – 38mm |
| ROB00061 | TKA Distal FMR Punches – 45mm |

# Table 22.4-22-11 CORI Disposables

| Article | Description |
|-----------------------|------------------------------|
| 4951 | Tablet Drape |
| ROB10031 | Tubing Set |
| ROB10032<br>PFSDV0016 | Flat Markers |
| ROB10033 | 6 mm Bullet Bur |
| ROB10034 | 6 mm Chip Breaker Bullet Bur |
| ROB10035 | 5 mm Cylindrical Bur |
| ROB10036 | 6 mm Cylindrical Bur |
| 74013401 | Speed Pins (110 mm) |
| 74013490 | Speed Pins (80 mm) |

# Table 22.4-22-12 CORI Country Bundles

| Article | Description |
|----------|-----------------------------|
| ROB20000 | CORI Robotics USA |
| ROB20001 | CORI Robotics EMEA Bundle 1 |
| ROB20002 | CORI Robotics EMEA Bundle 2 |
| ROB20003 | CORI Robotics EMEA Bundle 3 |
| ROB20004 | CORI Robotics EMEA Bundle 4 |
| ROB20005 | CORI Robotics EMEA Bundle 5 |
| ROB20006 | CORI Robotics EMEA Bundle 6 |
| ROB20007 | CORI Robotics APAC Bundle 1 |
| ROB20008 | CORI Robotics APAC Bundle 2 |
| ROB20009 | CORI Robotics APAC Bundle 3 |
| ROB20010 | CORI Robotics APAC Bundle 4 |
| ROB20011 | CORI Robotics APAC Bundle 5 |
| ROB20012 | CORI Robotics ROW Bundle 1 |

#### 

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized | Version: 4.0-Master, 07 Sep<br>2022 |
| Controlled Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in | |
| unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 148 of 167 |

| Article | Description |
|----------|----------------------------|
| ROB20013 | CORI Robotics ROW Bundle 2 |
| ROB20014 | CORI Robotics ROW Bundle 3 |
| ROB20015 | CORI Robotics ROW Bundle 4 |
| ROB20016 | CORI Robotics ROW Bundle 5 |

## Table 22.4-22-13 CORI Welcome Box

| Article | Description |
|----------|--------------------|
| ROB10299 | Welcome Box USA |
| ROB10300 | Welcome Box ROW 1 |
| ROB10301 | Welcome Box ROW 2 |
| ROB10302 | Welcome Box ROW 3 |
| ROB10303 | Welcome Box ROW 4 |
| ROB10304 | Welcome Box ROW 5 |
| ROB10305 | Welcome Box EMEA 1 |
| ROB10306 | Welcome Box EMEA 2 |
| ROB10307 | Welcome Box EMEA 3 |
| ROB10308 | Welcome Box EMEA 4 |
| ROB10309 | Welcome Box EMEA 5 |
| ROB10310 | Welcome Box APAC 1 |
| ROB10311 | Welcome Box APAC 2 |
| ROB10312 | Welcome Box APAC 3 |
| ROB10313 | Welcome Box APAC 4 |
| ROB10314 | Welcome Box APAC 5 |
| ROB10315 | Welcome Box APAC 6 |

# Table 22.4-22-14 CORI Product Documents / Other

| Article | Description |
|----------|------------------------------------------|
| ROB10400 | REAL INTELLIGENCE Implant Database v2.85 |
| ROB10401 | REAL INTELLIGENCE Archiving USB |
| ROB10402 | REAL INTELLIGENCE Supporting Documents |
| ROB10403 | REAL INTELLIGENCE CORI Quick Start Guide |
| ROB10404 | REAL INTELLIGENCE CORI Tray Guide |
| ROB10400 | REAL INTELLIGENCE Implant Database v2.85 |

#### 

This document contains information that is confidential and proprietary to Smith & Nephew PLC and Smith & Nephew, Inc. and is intended for use only by Smith+Nephew and its manufacturer. It shall not be reproduced or copied in whole or in part, nor shall the contents be disclosed by any means without prior written permission from Smith+Nephew, nor shall anyone make any use of it that is contrary to the expressed or implied wishes of Smith+Nephew.

TMP-CD-05-01 Clinical Protocol - Device - Revision D; SOP-CD-05 Clinical Protocol

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 149 of 167 |

#### Table 22.4-22-15 CORI Power Cords

| Article | Description |
|----------|--------------------------|
| ROB10199 | Power Cord North America |
| ROB10200 | Power Cord ROW 1 |
| ROB10201 | Power Cord ROW 2 |
| ROB10202 | Power Cord ROW 3 |
| ROB10203 | Power Cord ROW 4 |
| ROB10204 | Power Cord ROW 5 |
| ROB10205 | Power Cord EMEA 1 |
| ROB10206 | Power Cord EMEA 2 |
| ROB10207 | Power Cord EMEA 3 |
| ROB10208 | Power Cord EMEA 4 |
| ROB10209 | Power Cord EMEA 5 |
| ROB10210 | Power Cord EMEA 6 |
| ROB10211 | Power Cord APAC 1 |
| ROB10212 | Power Cord APAC 2 |
| ROB10213 | Power Cord APAC 3 |
| ROB10214 | Power Cord APAC 4 |
| ROB10215 | Power Cord APAC 5 |

# 22.5 HEALTH ECONOMIC OUTCOME MEASURES/ QUALITY OF LIFE MEASURES

Refer to Section 9.2 & 9.3 for Quality of Life measures.

# 22.6 PRINCIPAL INVESTIGATOR OBLIGATIONS

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 150 of 167 |

## 22.6.1 Principal Investigator Obligation according to ISO14155:2020

- 1. General:
- 2. The role of the PI is to implement and manage the day-to-day conduct of the clinical investigation as well as ensure data integrity and the rights, safety, and well-being of the subjects involved in the clinical investigation.
- 3. The PI is responsible for ensuring adequate training and qualification of the investigation site team and for maintaining oversight of their activities. The principal investigator may delegate tasks to qualified members of the investigation site team but retains responsibility for the clinical investigation (see also 7.6). This also applies when activities are outsourced to an external organization by the principal investigator in which case he/she shall implement procedures to ensure the integrity of all tasks performed and any data generated by this external organization.
- 4. Qualification of the PI. The PI shall:
- be qualified by education, training, and experience to assume responsibility for the proper conduct of the clinical investigation in accordance with this International Standard; evidence of such qualifications of the PI and key

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 151 of 167 |

members of the investigation site team shall be provided to the Sponsor through up-to-date Curriculum Vitae (CV) or other relevant documentation,

- 6. be experienced in the field of application and trained in the use of the investigational device under consideration,
- 7. disclose potential conflicts of interest, including financial, that interfere with the conduct of the clinical investigation or interpretation of results, and
- 8. be knowledgeable with the method of obtaining informed consent.
- 9. Qualification of investigation site. The PI shall be able to demonstrate that the proposed investigation site:
- 10.has the required number of eligible subjects needed within the agreed recruitment period, and;
- 11.has an investigation site team that is: qualified by education, training, and experience to assume responsibility for the proper conduct of the clinical investigation in accordance with this document; evidence of such qualifications for members of the investigation site team shall be documented through up-to-date CVs or other relevant documentation,.
- 12.has adequate facilities.
- 13. Communication with the IEC. The PI shall:
- 14.provide the Sponsor with copies of any clinical-investigation-related communications between the PI and the IEC,
- 15.comply with the requirements described in 4.5 of ISO 14155.
- 16. Submit to the IEC the following information, any amendments and any additional documentation required by the IEC: The Protocol; IB or equivalent; informed consent form and any other written information provided to subjects; procedures

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 152 of 167 |

for recruiting subjects and advertising materials, if any; a copy of the CV of the PI(s) for with the IEC has oversight.

- 17.Provide documentation of the IECs approval/favorable opinion, identifying the documents and amendments on which the opinion was based, to the Sponsor, prior to commencing the clinical investigation.
- 18. Submit the following to the IEC if required by national regulations, the protocol or IEC, whichever is more stringent:

#### 19.SAEs

20.Requests for deviations, and reports of deviations, if the deviation affects subject's rights, safety, and well-being, or the scientific integrity of the clinical investigation. Document and report to the Sponsor and IEC a report of

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 153 of 167 |

deviations made to protect the rights, safety, and well-being of human subjects under emergency circumstances.

- 21. Progress reports, including safety summary and deviations
- 22. Amendments to any documents already approved by the IEC.
- 23.If applicable, notifications of suspension or premature termination
- 24.If applicable, justification and request for resuming the clinical investigation after suspension.
- 25. Clinical investigation report or summary.
- 26.As a minimum, during the clinical investigation, the following information shall be obtained in writing from the IEC prior to implementation:
- 27. Approval/favorable opinion of amendments
- 28.Approval of the request for deviations that can affect the subject's rights, safety, and well-being or scientific integrity of the clinical investigation
- 29. Approval for resumption of a suspended clinical investigation if applicable.
- 30.obtain the written and dated approval/favorable opinion of the IEC for the clinical investigation before recruiting subjects and implementing all subsequent amendments, if required,
- 31.promptly report any deviations from the protocol that affect the rights, safety or well-being of the subject or the scientific integrity of the clinical investigation, including those which occur under emergency circumstances, if required by the IEC, protocol or national regulations. In particular circumstances, the communication with the IEC can be performed by the Sponsor, partly or in full, in which case the Sponsor shall keep the Principal Investigator informed.
- 32.Informed consent process. The PI shall:
- 33.General:
- 34.Informed consent shall be obtained in writing from the subject and the process shall be documented before any procedure specific to the clinical investigation is

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 154 of 167 |

applied to the subject; except when special circumstances for emergency treatments apply (see below)

- 35.Process of obtaining informed consent. The general process for obtaining informed consent shall be documented in the protocol and shall comply with the following. These requirements also apply with respect to informed consent obtained from a subject's legally authorized representative:
- 36.Ensure that the PI or his/her authorized designee conducts the informed consent process
- 37.Include all aspects of the clinical investigation that are relevant to the subject's decision to participate throughout the clinical investigation
- 38.Avoid any coercion or undue improper influence on, or inducement of, the subject to participate
- 39. Not waive or appear to waive the subject's legal rights
- 40. Use native non-technical language that is understandable to the subject
- 41.Provide ample time for the subject to read and understand the informed consent form and to consider participation in the clinical investigation
- 42.Include personally dated signatures and the PI or an authorized designee responsible for conducting the informed consent process
- 43. Show how informed consent will be obtained in special circumstances (see below) where the subject is unable to provide him or herself, and
- 44.Ensure important new information is provided to new and existing subjects throughout the clinical investigation.
- 45. Special circumstances for informed consent (the following provisions are subject to national regulations):
- 46. Subject needing legally authorized representatives: informed consent may be given by the legally authorized representative only if a subject is unable to make the decision to participate in a clinical investigation (e.g., infant, child, or

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 155 of 167 |

juvenile, seriously ill or unconscious subject, mentally ill person, mentally handicapped person). In such cases, the subject shall also be informed about the clinical investigation within his/her ability to understand.

- 47. Subject unable to read or write: informed consent shall be obtained through a supervised oral process if a subject or legally authorized representative is unable to read or write. An independent witness shall be present throughout the process. The written informed consent form and any other information shall be read aloud and explained to the prospective subject or his/her legally authorized representative and, whenever possible, either shall sign and personally date the informed consent form. The witness also signs and personally dates the informed consent for attesting that the information was accurately explained and that the informed consent was freely given.
- 48. Emergency treatments:
- 49.For clinical investigations involving emergency treatments, when prior informed consent of the subject is not possible because of the subject's medical condition, the informed consent of the subject's legally authorized representative, if present, shall be requested.
- 50. When it is not possible to obtain prior informed consent from the subject, and the subject's legally authorized representative, is not available, the subject may still be enrolled if a specific process has been described in the protocol.
- 51.Arrangements shall be made to inform the subject or legally authorized representative, as soon as possible, about the subject's inclusion in the clinical investigation and about all aspects of the clinical investigation.
- 52. The subject shall be asked to provide informed consent for continued participation as soon as his/her medical condition allows.
- 53. The Principal Investigator may not enroll a subject without obtaining informed consent of the subject or his/her legally authorized representative only when the following conditions are fulfilled: the prospective subject fulfils the emergency

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 156 of 167 |

conditions and is obviously in a life-threatening situation; no sufficient clinical benefits are anticipated from the currently available treatment; there is a fair possibility that the life-threatening risk to the prospective subject can be avoided if the investigational device is used; anticipated risks are outweighed by the potential benefits of applying the investigational device; the legally authorized representative cannot be promptly reached and informed.

54.Information provided to the subject. All information pertinent to the clinical investigation, including at least the following, shall be provided in writing and in

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 157 of 167 |

native, non-technical language that is understandable to the subject (or the subject's legally authorized representative):

- 55.Description and purpose
- 56.Potential benefits
- 57.Risks and inconveniences or the subject and, when applicable, for any embryo, fetus or nursing infant
- 58. Alternative procedures
- 59. Confidentiality
- 60.Compensation
- 61.Anticipated expenses, if any, to be borne by the subject for participating in the clinical investigation
- 62. Information on the role of Sponsor's representative in the clinical investigation
- 63.Contact persons
- 64.Statement declaring that new findings or the reasons for any amendment to the protocol that affect the subject's continued participation shall be made available to the subject
- 65. Statement indicating that, upon the subject's approval, the subject's personal physician will be informed of the subject's participation in the clinical investigation
- 66.Statement indicating that a description of the clinical investigation has or shall be registered in a publicly accessible database
- 67.Termination procedures
- 68. Informed consent signature shall contain the following:
- 69. The voluntary agreement to participate in the clinical investigation and follow the investigator's instructions
- 70.A statement declaring that refusal of participation incurs no penalty for the subject and no loss of benefits to which the subject is otherwise entitled;

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 158 of 167 |

- 71.A statement declaring that discontinuation/withdrawal and thereby revoking the informed consent at any time incurs no penalty for the subject;
- 72.A statement with regard to the possible consequences of withdrawal
- 73.An acknowledgment of the information provided and confirmation that all the subject's questions were answered that the subject acknowledges the information provided during the informed consent process and that (s)he had ample time to consider participation
- 74.A statement confirming that the subject or his/her legally authorized representative agrees to the use of the subject's relevant personal data for the purpose of the clinical investigation
- 75.A statement confirming that the subject or his/her legally authorized representative agrees that Sponsor's representatives, regulatory authorities and IEC representatives will be granted direct access to the subject's medical records.
- 76. New information: if new information becomes available that can significantly affect a subject's future health and medical care, that information shall be provided to the subject(s) affected in written form. If relevant, all affected subjects shall be asked to confirm their continuing consent in writing.
- 77.ensure compliance with the applicable regulatory requirements and ethical principles for the process of obtaining informed consent, and ensure and

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | Version: 4.0-Master, 07 Sep<br>2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 159 of 167 |

document appropriate training if an authorized designee is appointed to conduct the informed consent process.

- 78. Compliance with the protocol. The Principal Investigator shall:
- 79.indicate his/her acceptance of the protocol in writing,
- 80.conduct the clinical investigation in compliance with the protocol,
- 81.create and maintain source documents throughout the clinical investigation and make them available as requested during monitoring visits or audits as well as maintain documentation of the type and location of these source documents,,
- 82.ensure that the investigational device is used solely by authorized users as specified in 7.2, and in accordance with the protocol and instructions for use,
- 83.propose to the Sponsor any appropriate modification(s) of the protocol or investigational device or of the use of the investigational device,
- 84.refrain from implementing any modifications to the protocol without agreement from the Sponsor, IEC and regulatory authorities, if required,
- 85.document and explain any deviation from the approved protocol that occurred during the course of the clinical investigation,
- 86.ensure that an adequate investigation site team and facilities exist and are maintained and documented during the clinical investigation,
- 87.ensure that maintenance and calibration of the equipment relevant for the assessment of the clinical investigation is appropriately performed and documented, where applicable,
- 88.ensure the accuracy, completeness, legibility, and timeliness of the data reported to the Sponsor in the CRF and in all required reports,
- 89.maintain the device accountability records,
- 90. Comply with the procedure for the safe return of investigational devices including potentially hazardous devices and, in the case of reported device deficiencies, collaborate with the sponsor to provide the necessary information allowing an

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized<br>Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 160 of 167 |

accurate analysis where appropriate. requirements and provide any information need to analyze device deficiencies, if applicable.

- 91.allow and support the Sponsor to perform monitoring and auditing activities,
- 92.be accessible to the monitor and respond to questions during monitoring visits,
- 93.determine the cause and implement appropriate corrective and preventative actions to address significant noncompliance,
- 94.allow and support regulatory authorities and the IEC when performing auditing activities,
- 95.ensure that all clinical-investigation-related records are retained as required taking measures to prevent accidental or premature destruction, and
- 96.review and sign the clinical investigation report, as applicable.
- 97. Medical care of subjects. The Principal Investigator shall
- 98.provide adequate medical care to a subject during and after a subject's participation in a clinical investigation in the case of adverse events,
- 99.inform the subject of the nature and possible cause of any adverse events experienced,
- 100. provide the subject with the necessary instructions on proper use, handling, storage, and return of the investigational device, when it is used or operated by the subject,
- 101. inform the subject of any new significant findings occurring during the clinical investigation, including the need for additional medical care that may be required,
- 102. provide the subject with well-defined procedures for possible emergency situations related to the clinical investigation, and make the necessary

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 161 of 167 |

arrangements for emergency treatment, including decoding procedures for blinded/masked clinical investigations, as needed,

- 103. ensure that clinical records are clearly marked to indicate that the subject is enrolled in a particular clinical investigation,
- 104. if appropriate, subjects enrolled in the clinical investigation shall be provided with some means of showing their participation in the clinical investigation, together with identification and compliance information for concomitant treatment measures (contact address and telephone numbers shall be provided),
- 105. inform, with the subject's approval or when required by national regulations, the subject's personal physician about the subject's participation in the clinical investigation, and
- 106. make all reasonable efforts to ascertain the reason(s) for a subject's premature withdrawal from the clinical investigation while fully respecting the subject's rights.
- 107. Safety reporting. The Principal Investigator shall:
- 108. record every adverse event and observed device deficiency, together with an assessment,
- 109. report to the Sponsor, without unjustified delay, all serious adverse events and device deficiencies that could have led to a serious adverse device effect; this

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 162 of 167 |

information shall be promptly followed by detailed written reports, as specified in the protocol,

- 110. report to the IEC serious adverse events and device deficiencies that could have led to a serious adverse device effect, if required by the national regulations or protocol or by the IEC,
- 111. report to regulatory authorities, serious adverse events and device deficiencies that could have led to a serious adverse device effect, as required by the national regulations, and
- 112. supply the Sponsor, upon Sponsor's request, with any additional information related to the safety reporting of a particular event.
- 113. Note, for studies conducted under 21 CFR Part 812 Investigational Device Exemption Regulations, an investigator shall prepare and submit the following complete, accurate, and timely reports:
- 114. Unanticipated Adverse Device Effects An investigator shall submit to the sponsor and to the reviewing IRB a report of any unanticipated adverse device effect occurring during an investigation as soon as possible, but in no event later than 10 working days after the investigator first learns of the effect.
- 115. Withdrawal of IRB approval. An investigator shall report to the sponsor, within 5 working days, a withdrawal of approval by the reviewing IRB of the investigator's part of an investigation.
- 116. Progress. An investigator shall submit progress reports on the investigation to the sponsor, the monitor, and the reviewing IRB at regular intervals, but in no event less often than yearly.
- 117. Deviations from the investigational plan. An investigator shall notify the sponsor and the reviewing IRB of any deviation from the investigational plan to protect the life or physical well-being of a subject in an emergency. Such notice shall be given as soon as possible, but in no event later than 5 working days after the emergency occurred. Except in such an emergency, prior approval by

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 163 of 167 |

the sponsor is required for changes in or deviations from a plan, and if these changes or deviations may affect the scientific soundness of the plan or the rights, safety, or welfare of human subjects, FDA and IRB also is required.

- 118. Informed consent. If an investigator uses a device without obtaining informed consent, the investigator shall report such use to the sponsor and the reviewing IRB within 5 working days after the use occurs.
- 119. Investigational device including clinical procedure risks and their disclosure.

  The PI shall:
- 120. Evaluate risks according to ISO 14971 before starting a trial,
- 121. Summarize benefit-risk analysis in trial documents,
- 122. Add residual risk and their nature, occurrence, severity, and outcome to the IB,
- 123. Include in CIP all anticipated adverse device effects and a rationale for the related benefit-risk ratio,
- 124. Include any anticipated adverse device effect in the consent form.

# 22.6.2 Principal Investigator Obligations according to GCP NMPA 2016

- Article 59 Before accepting clinical trial, clinical trial institutions shall evaluate relevant resources in accordance with the characteristics of investigational medical devices to decide whether to accept this clinical trial.
- Article 60 Clinical trial institutions shall properly keep clinical trial records and basic documents according to the agreement with the sponsor.
- Article 61 Investigators who are in charge of the clinical trial shall:
  - Have professional title and qualification above associate level, such as associate chief physician, associate professor and associate researcher in the clinical trial institutions;

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 164 of 167 |

- Have professional knowledge and experience required for investigational medical devices and pass relevant trainings if necessary;
- Be familiar with clinical trial requirements provided by sponsor, and the data and literatures related to clinical trial;
- ➤ Be able to coordinate, allocate and assign personnel and devices of this trial, and to handle the adverse events and other correlating events related to investigational medical devices;
- > Be familiar with relevant national laws, regulations and this Provision.
- Article 62 Prior to a clinical trial, the medical device clinical trial administrative department of clinical trial institutions shall coordinate sponsor to file applications to the ethics committee and submit relevant documents in accordance with relevant provisions.
- Article 63 Investigators shall ensure that the staff member participating in the trial are familiar with the principles, indications, product performance, operating methods, installation requirements and technical specifications of investigational medical devices, understand preclinical research data and safety data of investigational medical devices, and master precautions and emergency treatment for possible risks in clinical trial.
- Article 64 Investigators shall ensure all participants of clinical trial fully understand the clinical trial protocol, relevant provisions, characteristics of investigational medical devices and relevant responsibilities of clinical trial, make sure that enough subjects meeting inclusion criteria in clinical trial protocol can be enrolled into clinical trial, ensure enough time in the agreed trial period, to implement and complete clinical trial safely according relevant regulations.
- Article 65 The investigator shall ensure that the investigational medical devices are only used for subjects of the clinical trial, and used for free.
- Article 66 Investigators shall strictly comply with clinical trial protocol. Without consent of sponsor and ethics committee or approval of China Food and Drug

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 165 of 167 |

Administration in accordance with regulations, investigators shall not deviate the protocol or substantially change the protocol. However, in case of an emergency that subjects face direct danger that needs to be eliminated immediately, it can be reported in writing afterwards.

- Article 67 Investigators shall be responsible for recruiting subjects and talking
  with subjects or their guardians. Investigators are responsible to specify the
  details relating to investigational medical devices and clinical trial for subjects,
  inform subjects of possible benefits and known and foreseeable risks, and
  obtain the signed and dated informed consent form from subjects and their
  guardians.
- Article 68 Investigators and other personnel participated in the trial shall not force or induce subjects in improper way to take part in the trial.
- Article 69 In case of finding unanticipated adverse events of investigational medical devices during clinical trial, investigators shall revise relevant content of informed consent form together with the sponsor. After being reviewed and approved by ethics committee in accordance with relevant working procedure, the affected subjects and their guardians shall resign the revised informed consent form for confirmation.
- Article 70 Investigators shall be responsible for making decisions relating to clinical trial. In case of adverse events relating to clinical trial, clinical trial institutions and investigators shall provide sufficient and timely treatment and management to subjects. In case subjects have complications and need treatment and management, investigators shall timely notify subjects.
- Article 71 In case of serious adverse events during clinical trial, investigators shall take proper treatment measures for subjects immediately, then report to medical device clinical trial administrative departments of clinical trial institutions where they belong to, and notify sponsor in writing through them. Clinical trial administrative departments of medical devices shall report to corresponding ethics committee and Food and Drug Administration of province,

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 166 of 167 |

autonomous region or municipality and the Health and Family Planning Commission where the clinical trial institution is located in written form within 24 hours. For lethal events, clinical trial institutions and investigators shall provide all necessary data to ethics committee and sponsor.

- Article 72 Investigators shall record all adverse events and device deficiency
  that occur during the process of clinical trial, analyze event cases together with
  sponsor, draft written analysis report, put forward opinions of continuing,
  suspending or terminating the trial, and report to ethics committee for review
  through medical device clinical trial administrative departments of clinical trial
  institutions.
- Article 73 Investigators shall ensure that clinical trial data are filled in case report forms accurately, completely, clearly and timely. Case report forms shall be signed by investigators. Any change of data shall be signed and dated by investigator, original records should be kept, clear and recognizable.
- Article 74 Clinical trial institutions and investigators shall ensure authenticity, accuracy, clarity and safety of data and documents generated in clinical trial.
- Article 75 Clinical trial institutions and investigators shall accept the monitoring and audit of sponsor as well as supervision of ethics committee, and provide all required records relating to the trial. In case Food and Drug Administration and Health and Family Planning Commission send inspectors to implement inspection, clinical trial institutions and investigators shall cooperate with them.
- Article 76 In case clinical trial institutions and investigators identify risks
  overweighting possible benefits, or have obtained the results that is sufficient
  to judge the safety and effectiveness of investigational medical devices, thus
  need to suspend or terminate clinical trial, it is required to notify subjects and
  ensure subjects to obtain proper treatment and follow-up, report in accordance
  with regulations and provide detailed written explanation at the same time. If
  necessary, report to the Food and Drug Administration of province,
  autonomous region or municipality where it locates.

| Clinical Protocol | Study Number: CORI.2019.06 |
|---|---|
| A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and | <b>Version</b> : 4.0-Master, 07 Sep 2022 |
| Effectiveness of REAL INTELLIGENCE™ CORI™ in unicondylar knee arthroplasty (UKA) Procedure | <b>Page</b> : 167 of 167 |

- In case of receiving the notification of sponsor or ethics committee on the need
  of suspending or terminating clinical trial, investigators shall timely notify
  subjects and ensure subjects to obtain proper treatment and follow-up.
- Article 77 In case the sponsor violates relevant regulations or request to change
  the trial data and conclusion, clinical trial institutions and investigators shall
  report to Food and Drug Administration of province, autonomous region or
  municipality where the sponsor is located or report to the China Food and Drug
  Administration.
- Article 78 At the end of a clinical trial, the investigator shall ensure the
  completion of all records and reports. Meanwhile, the investigator shall ensure
  the quantity of received investigational medical devices is consistent with the
  used, discarded or returned devices, and ensure that the rest investigational
  medical devices are disposed properly and recorded for filing.
- Article 79 Investigators can authorize corresponding personnel to recruit subjects, continuously communicate with subjects, record the clinical trial data, and manage investigational medical devices in accordance with the needs of clinical trial. Investigators shall implement relevant training for the authorized personnel and document accordingly.